Official title: Study Protocol NCT number: NCT01745822 Document date: April 20, 2015

# Protocol

A phase III, placebo controlled, double blind, randomized clinical trial to assess the efficacy and safety of tenofovir disoproxil fumarate given from 28 weeks' gestation until 2 months postpartum to Hepatitis B (HB) virus chronically infected, HBsAg and HBeAg positive pregnant women to prevent perinatal transmission of HBV to their infants who receive passive-active HBV immunization

#### Short title:

Maternal antiviral prophylaxis to prevent perinatal transmission of HBV in Thailand (iTAP)

Version 3.0 April 20, 2015

#### Principal investigators:

- 1. Dr. Gonzague Jourdain
- 2. Dr. Nantasak Chotivanich

**Coordinating Center:** 

IRD PHPT - 187/10 Changklan Rd., Changklan, Muang, Chiang Mai, 50100 Thailand

Phone: 053819125-9 - Fax: 053252253, 053819130

Email: Gonzague.Jourdain@phpt.org, Nicole.Ngo-Giang-Huong@phpt.org

0 8 WH. 2558 คณะกรรมการจริยธรรมดารวิจัยในมนุษย์

สถาบันพัฒษาการโดยพระธาร**วิจัยในบนุพย์ (สกม** 

# **Table of Contents**

| 1. | Titl | e of the project | 3 |
|---|---|---|---|
| 2. | Pri | ncipal Investigator and Co-Investigators' names and contact information | 3 |
| 3. | Pro | pject Summary | 8 |
| 4. | Bad | ckground information | 9 |
| | 4.1. | Epidemiology | 9 |
| | 4.2. | Hepatitis B virus | 9 |
| | 4.3. | Natural history | 9 |
| | 4.4. | Antiviral treatment of HBV infection | 10 |
| | 4.5. | HBV infection during pregnancy and postpartum | 11 |
| | 4.6. | Perinatal transmission of HBV in the era of HBV immunization | 11 |
| | 4.7. | Additional interventions to potentially prevent perinatal transmission | 12 |
| | 4.7 | 7.1. Elective C-section | 12 |
| | 4.7 | 7.2. HBlg during pregnancy | 12 |
| | 4.7 | 7.3. Antivirals administered to the mother | 12 |
| | 4.7 | 7.4. Conclusion | 16 |
| | 4.8. | Sub-studies | 16 |
| 5. | Stu | udy objectives | 16 |
| 3. | Stu | udy sites and duration of the study | 18 |
| | 6.1. | Study sites | 18 |
| | 6.2. | Duration of the study | 20 |
| 7. | Wc | orkplan | 20 |
| | 7.1. | Selection of participants | 20 |
| | 7.1 | l.1. Eligibility criteria | 20 |
| | 7.1 | I.2. Inclusion and exclusion criteria | 21 |
| | 7.1 | l.3. Discontinuation criteria | 22 |
| | 7.2. | Implementation, data collection and monitoring procedures | 23 |
| | 7.2 | 2.1. Maternal follow up | 23 |
| | 7.2 | 2.2. Liver enzyme exacerbations | 25 |
| | 7.2 | 2.3. Assessment of Maternal Tenofovir Plasma Exposure | 26 |
| | 7.2 | 2.4. Bone Mineral Density Evaluations | 27 |
| | 7.2 | 2.5. Infant follow up and diagnosis of HBV infection | 27 |
| | 7.3. | Study drugs | 29 |
| | 7.4. | Statistical considerations | 29 |
| | 7.4 | 1.1. Endpoints | 29 |
| | 7.4 | 4.2. Randomization and Stratification | 29 |
| | 7.4 | 1.3. Sample size and Accrual | 30 |
| | | 4.4. Information of the co-investigators | |
| | 7.4 | 4.5. Monitoring by the program scientists | 30 |

| | 7.4.6. Data and Safety Monitoring Board (DSMB) | .31 |
|---|---|---|
| | 7.4.7. Analyses for the primary objective/endpoint | .31 |
| | 7.4.8. Analyses for secondary objectives/endpoints | .32 |
| | 7.4.9. Pharmacokinetic data to estimate individual maternal tenofovir exposure | .32 |
| | 7.4.10. Bone mineral density measurements | .32 |
| | 7.4.11. Exploratory analyses | .33 |
| 8. | Ethical considerations | .33 |
| 8 | 8.1. Possible risks including preventive or alleviative measures | .33 |
| | 8.1.1. Potential Risks to Participants | .33 |
| 8 | 3.2. Adequacy of protection against risks | .35 |
| | 8.2.1. Recruitment and informed consent (see Consent Form in Appendix 1) | .35 |
| 8 | 3.3. Protection against risk | .36 |
| | 8.3.1. Institutional Review Board | .36 |
| | 8.3.2. Expedited Adverse Experience Reporting | 36 |
| | 8.3.3. Confidentiality | 36 |
| | 8.3.4. Biohazard Containment | .36 |
| 9. | References | .38 |
| Арј | pendix 1: Informed Consent Form to Participate in iTAP Study (Thai Language) | .43 |
| Ap <sub>l</sub><br>Lar | pendix 1 (continued): Informed Consent Form to Participate in iTAP Study (Englishinguage) | 52 |
| App | pendix 2: Exempted Congenital Anomaly/Birth Defect (Listed by Body Site) | 59 |
| Ap | pendix 3: Screening program for symptoms possibly associated with mitochondrial sfunction in the EPF cohort (68) | |
| Apı | pendix 4: Cockcroft-Gault formula for women | 62 |
| Apı | pendix 5: How to Measure Head Circumference, Length and Weight | 63 |
| | pendix 6: Additional Informed Consent Form to Participate in Tenofovir Plasma Level asurements (Thai Language) | 64 |
| | pendix 6 (continued): Additional Informed Consent Form to Participate in Tenofovir Plasr<br>vel Measurements (English Language) | |
| | pendix 7: Additional Informed Consent Form to Participate in DXA Scan Assessments (T<br>nguage) | |
| | pendix 7 (continued): Additional Informed Consent Form to Participate in DXA Scan<br>sessments (English Language) | 75 |

# 1. Title of the project

A phase III, placebo controlled, double blind, randomized clinical trial to assess the efficacy and safety of tenofovir disoproxil fumarate given from 28 weeks' gestation until 2 months postpartum to Hepatitis B (HB) virus chronically infected, HBsAg and HBeAg positive pregnant women to prevent perinatal transmission of HBV to their infants who receive passive-active HBV immunization.

## **Short title:**

Maternal antiviral prophylaxis to prevent perinatal transmission of HBV in Thailand

## 2. Principal Investigator and Co-Investigators' names and contact information

| Principal Investigators: | |
|---|---|
| Gonzague Jourdain, MD, PhD<br>PHPT - IRD<br>187/10, Changklan Rd., Changklan, Muang<br>Chiang Mai 50100<br>Tel: +66 5381 9125<br>Fax: +66 5381 9130<br>Email: Gonzague.Jourdain@phpt.org | Nantasak Chotivanich, MD Obstetrics & Gynecology Department Chonburi Hospital, Chonburi 69 M. 2 Sukumvith Rd., T. Ban Suan, Muang, Chonburi 20000 Tel: +66 3893 1390, +66 3893 1000 Fax +66 3827 4911 Email: nantasak.cho@gmail.com |

| Co-investigators: | |
|---|---|
| Nicole Ngo-Giang-Huong, PharmD, PhD<br>PHPT - IRD<br>187/10, Changklan Rd., Changklan, Muang<br>Chiang Mai 50100<br>Tel: +66 5381 9125- Fax: +66 5381 9130<br>Email: Nicole.Ngo-Giang-Huong@phpt.org | Tim Roy Cressey, PhD<br>PHPT - IRD<br>187/10, Changklan Rd., Changklan, Muang<br>Chiang Mai 50100<br>Tel: +66 5381 9125 - Fax: +66 5381 9130<br>Email: tim.cressey@phpt.org |
| Satawat Thongsawat, MD Division of Gastroenterology Department of Internal Medicine, Faculty of Medicine, Chiang Mai University Muang, Chiang Mai 50200 Tel: +66 5394 5483-5 - Fax: +66 5394 5481 Email: satawat@yahoo.com | Thanyawee Puthanakit, MD Department of Pediatrics, Faculty of Medicine Chulalongkorn University 1873 Rama 4 Road, Pathumwan, Bangkok10330 Tel: +66 2256 4951- Fax: +66 2256 4911 Email: thanyawee.p@hivnat.org |
| Chureeratana Bowonwatanuwong, MD Medical Department Chonburi Hospital 69 M. 2 Sukumvith Rd., T. Ban Suan, Muang Chonburi 20000 Tel: +66 3827 4200 -7- Fax: +66 3893 1100 Email: c.bowon@gmail.com | Virat Klinbuayaem, MD Medical Department Sanpatong Hospital 149 M.9 T. yuwa Sanpatong, Sanpatong, Chiang Mai 50120 Tel: +66 5331 1404, 5331 1711 Fax: +66 5331 1712 Email: kggvirat@hotmail.com |



| Pornnapa Suriyachai, MD Obstetrics &Gynecology Department Phayao Hospital 269 Phaholyothin Rd., T. Tom, Muang, Phayao 56000 Tel: +66 5443 1209 - Fax: +66 5440 9330 Email: whan76_1@hotmail.com | Pannarai Srisuwan, MD Pediatrics Department Phayao Hospital 269 Phaholyothin Rd., T. Tom, Muang, Phayao 56000 Tel: +66 5443 1169 -Fax: +66 5448 1708 Email: pcaipyhos@gmail.com |
|---|---|
| Chaiwat Putiyanun, MD Obstetrics & Gynecology Department Chiang Kham Hospital 244 M.4 T. Yuan, Chiang Kham, Phayao 56110 Tel: +66 54451300-1 - Fax: +66 54416615 Email: putiyanun@hotmail.com | Sudanee Buranabanjasatean, MD Obstetrics & Gynecology Department Mae Chan Hospital 274 M.5 Phaholyothin Rd., Mae Chan, Chiang Rai 57110 Tel: +66 5377 1056 – Fax: +66 5366 0961 Email: sudanee2011@windowslive.com |
| Jullapong Achalapong, MD Obstetrics &Gynecology Department Chiangrai Prachanukroh Hospital 1039 Sathanpayaban Rd., Muang, Chiang Rai 57000 Tel: +66 5371 1300 ext 1217 - Fax: +66 5371 3044 Email: drjullapong@gmail.com | Chulapong Chanta, MD Pediatrics Department Chiangrai Prachanukroh Hospital 1039 Sathanpayaban Rd., Muang, Chiang Rai 57000 Tel: +66 5371 1300 ext 1274 - Fax: +66 5371 3044 Email: Chul_chan@yahoo.com |
| Aram Limtrakul, MD Obstetrics &Gynecology Department Nakornping Hospital 159 M.10 Chotana Rd., T. Don Keaw, Mae Rim, Chiang Mai 50180 Tel: +66 5399 9200 – Fax: +66 5322 2152 | Arunrat Suwannarat, MD Pediatrics Department Nakornping Hospital 159 M.10 Chotana Rd., T. Don Keaw, Mae Rim, Chiang Mai 50180 Tel: +66 5399 9200 – Fax: +66 5322 2152 Email: arunrat11@yahoo.com |
| Suraphan Sangsawang, MD Obstetrics &Gynecology Department Health Promotion Center Region 10 51 Prachasumphan Rd., T. Changklan, Muang, Chiang Mai 50100 Tel: +66 5327 2740 – Fax: +66 5327 4015 ext 119 Email: suraphan@anamai.moph.go.th | Kanokwan Jittayanun, MD Pediatrics Department Health Promotion Center Region 10 51 Prachasumphan Rd., T. Changklan, Muang, Chiang Mai 50100 Tel: +66 5327 2740 – Fax: +66 5327 4015 ext 119 Email: kkulsawad@yahoo.co.th |
| Wanmanee Matanasarawut,MD Obstetrics &Gynecology Department Lamphun Hospital 177 Sai Rim Ping Rd., T. Tonthong, Muang, Lamphun 51000 Tel: +66 5356 9100 ext 2150 – Fax: +66 5356 9123 Email: obgyn.lph@gmail.com | Rosalin Somsamai, MD Pediatrics Department Lamphun Hospital 177 Sai Rim Ping Rd., T. Tonthong, Muang, Lamphun 51000 Tel: +66 5356 9100 – Fax: +66 5356 9123 Email: sukannika_waan@hotmail.com |
| Prateung Liampongsabuddhi, MD Obstetrics &Gynecology Department Lampang Hospital 280 Paholyothin Rd., Huawieng, Muang, Lamphang 52000 Tel: +66 5422 3623-7 – Fax: +66 5422 6126 Email: prateung@yahoo.com | Kultida Pongdetudom, MD Pediatrics Department Lampang Hospital 280 Paholyothin Rd., Huawieng, Muang, Lamphang 52000 Tel: +66 5422 3623-7 – Fax: +66 5422 6126 Email: pongdetudom@yahoo.com |



| Thitiporn Siriwachirachai, MD Obstetrics &Gynecology Department Khon Kaen Hospital 56 Srichan Rd, Naimuang, Muang, | Ussanee Srirompotong, MD<br>Pediatrics Department<br>Khon Kaen Hospital<br>56 Srichan Rd, Naimuang, Muang, |
|---|---|
| Khon Kaen 40000<br>Tel: +66 4333 6789 – Fax: +66 4323 6974<br>Email: siriwachirachai@hotmail.com | Khon Kaen 40000<br>Tel: +66 4333 6789 – Fax: +66 4323 6974 |
| Prapap Yuthavisuthi, MD Obstetrics &Gynecology Department Prapokklao Hospital 38 Leibnern Rd., Muang Chantaburi 22000 Tel: +66 3932 4975 ext. 5253 - Fax: +66 3931 1511 Email: yuthavisuthi@gmail.com | Chaiwat Ngampiyasakul, MD Pediatrics Department Prapokklao Hospital 38 Leibnern Rd., Muang Chantaburi 22000 Tel: +66 3932 4975 ext. 5253 - Fax: +66 3931 1511 Email: chaiwat008@gmail.com |
| Prateep Kanjanavikai, MD Obstetrics &Gynecology Department Banglamung Hospital 669 M.5 Phattaya-Naklua T. Naklua, Banglamung, Chonburi 20150 Tel: +66 3841 1551-2 – Fax: +66 3842 8464 Email: prateep48@hotmail.com | Siriluk Phanomcheong, MD Pediatrics Department Banglamung Hospital 669 M.5 Phattaya-Naklua T. Naklua, Banglamung, Chonburi 20150 Tel: +66 3841 1551-2 – Fax: +66 3842 8464 Email: siriluk_lukk@yahoo.com |
| Sombat Thanprasertsuk, MD Senior Consultant Department of Disease Control Ministry of Public Health Tivanont Road, Muang Nonthaburi 11000 Tel: +66 2590 3201 - Fax: +66 25918413 | Suchat Hongsiriwon, MD Pediatrics Department Chonburi Hospital, Chonburi 69 M. 2 Sukumvith Rd., T. Ban Suan, Muang, Chonburi 20000 Tel: +66 3827 4000-7 Fax: +66 3827 4911 Email: suchat.hong@gmail.com |
| Supang Varadisai, MD Obstetrics &Gynecology Department Samutsakhon Hospital 1500 Akekachai Rd., T. Mahachai, Muang, Samutsakorn 74000 Tel: +66 34427099-104 – Fax: +66 34411488 | Sawitree Krikajornkitti, MD<br>Pediatrics Department<br>Samutsakhon Hospital<br>1500 Akekachai Rd., T. Mahachai, Muang,<br>Samutsakorn 74000<br>Tel: +66 3442 7099-104 – Fax: +66 3441 1488<br>Email: yuiwitree@gmail.com |
| Veeradate Chalermpolprapa, MD Obstetrics &Gynecology Department Nakhonpathom Hospital 196 Thesa Rd., T. Prapathomjadee, Muang, Nakhonpathom 73000 Tel: +66 34213606, +66 34213607-8 Fax: +66 34251553 Email: veeradate@hotmail.com | Suthunya Bunjongpak, MD Pediatrics Department Nakhonpathom Hospital 196 Thesa Rd., T. Prapathomjadee, Muang, Nakhonpathom 73000 Tel: +66 34213606, +66 34213607-8 Fax: +66 34251553 Email: suthunya12@thaimail.com |
| Prapan Sabsanong, MD Obstetrics & Gynecology Department Samutprakarn Hospital 71 Chakapak Rd., T. Pak Nam, Muang, Samutprakarn 10280 Tel: +66 27018 132-9, +66 2387 0053 Fax: +66 2173 8551 Email: prapandr@hotmail.com | Achara Puangsombat, MD Pediatrics Department Samutprakarn Hospital 71 Chakapak Rd., T. Pak Nam, Muang Samutprakarn 10280 Tel: +66 27018 132-9, +66 2387 0053 Fax: +66 2173 8551 |



| Orada Patamasingh Na Ayudhaya, MD Obstetrics & Gynecology Department Nopparat Rajathanee Hospital 679 Ram-Indra Rd., Kannayao, Bangkok 10230 Tel: +66 2517 4270-9 – Fax: +66 2917 8800 Email: oradaaom@hotmail.com | Anita Luvira, MD Pediatrics Department Nopparat Rajathanee Hospital 679 Ram-Indra Rd., Kannayao, Bangkok 10230 Tel: +66 2517 4270-9 – Fax: +66 2917 8800 Email: aluvira@yahoo.com |
|---|---|
| Sinart Prommas, MD Obstetrics &Gynecology Department Bhumibol Adulyadej Hospital Phaholyothin Rd., Saimai, Bangkok 10220 Tel: +66 2534 7317 - Fax: +66 2523 8873 Email: n_prommas@hotmail.com | Prapaisri Layangool, MD Pediatrics Department Bhumibol Adulyadej Hospital Phaholyothin Rd., Saimai, Bangkok 10220 Tel: +66 2534 7306 - Fax: +66 2534 7295 Email: p_layangool@yahoo.com |
| Rapee Chalermwutanont, <sup>1</sup> MD Obstetrics &Gynecology Department Ranong Provincial Hospital 11 Kamlangsupt Rd., Khao Niwet Muang Ranong, Thailand 85000 Tel: +66 7781 1574-5, +66 7781 2630-3 Fax: +66 7782 326-7 | Uraiwan Tuntrakul, MD Pediatrics Department Ranong Provincial Hospital 11 Kamlangsupt Rd., Khao Niwet Muang Ranong, Thailand 85000 Tel: +66 7781 1574-5, +66 7781 2630-3 Fax: +66 7782 326-7 |
| Pichit Puernngoluerm, MD Obstetrics &Gynecology Department Maharaj Nakornratchasrima Hospital 49 Changpuag Rd, Muang Nakornratchasrima 30000 Tel: +66 4423 5000 - Fax: +66 4424 6389 | Anucha Saeresjittima, MD Pediatrics Department Maharaj Nakornratchasrima Hospital 49 Changpuag Rd, Muang Nakornratchasrima 30000 Tel: +66 4423 5000 - Fax: +66 4424 6389 |
| Linda Harrison, MS Harvard School of Public Health Center for Biostatistics in AIDS Research FXB Building 514 651 Huntington Ave Boston, MA 02115, USA Tel: +1 6174320062 Email: lharriso@sdac.harvard.edu | Camlin Tierney, PhD Harvard School of Public Health Center for Biostatistics in AIDS Research FXB Building 514 651 Huntington Ave Boston, MA 02115, USA Tel: +1 6174320547 Email: tierney@sdac.harvard.edu |
| Wasna Sirirungsi, PhD Faculty of Associated Medical Sciences Chiang Mai University 110 Intawaroros Rd. T. Sripoom Muang, Chiang Mai 50200 Tel: +66 5394 5063 - Fax: +66 5394 6042 Email: wasna.s@cmu.ac.th | Stanislas Pol, MD, PhD Department of Hepato-Gastroenterology, Cochin University Hospital, 27 rue du Faubourg Saint-Jacques, 75679 Paris Cedex 14, France Tel: +33 1 58 41 19 55 Email: stanislas.pol@cch.aphp.fr |
| Raymond T. Chung, MD Massachusetts General Hospital Gastrointestinal Unit WRN 1007C, GI Unit 55 Fruit St Boston, MA 02114, USA Tel: +1 617/724-7562 - Fax: +1 617/643-0446 Email: rtchung@partners.org | George Siberry, MD, MPH Pediatric, Adolescent, and Maternal AIDS (PAMA) Branch Eunice Kennedy Shriver National Institutes of Child Health and Human Development National Institutes of Health 6100 Executive Boulevard, Room 4B11H Bethesda, MD 20892-7510, USA Tel: 301-496-7350 - Fax: 301-496-8678 Email: siberryg@mail.nih.gov |





| Trudy Murphy, MD Centers for Disease Control and Prevention DHHS/CDC//NCHHSTP/DVH/Vaccine Unit Bldg Corporate SQ 12, Room 3111 Atlanta GA 30329-1902, USA Tel: +1 404 639 8845 - Fax: +1 4047188595 Email: trudy.murphy@cdc.hhs.gov;tkm4@cdc.gov | Heather Watts, MD Pediatric, Adolescent, and Maternal AIDS Branch NIH, NICHD, CRMC 6100 Executive Blvd, Room 4B11, MSC 7510 Bethesda, MD 20892-7510, USA Tel:+1 301 435-6874 - Fax: +1 301 496-8678 Email: wattsh@exchange.nih.gov, hw59l@nih.gov |
|---|---|
| Woottichai Khamduang, PhD<br>PHPT - IRD<br>187/10, Changklan Rd., Changklan, Muang<br>Chiang Mai 50100<br>Tel: +66 5381 9125 - Fax: +66 5381 9130<br>Email: woottichai.khamduang@phpt.org | Noele P. Nelson, MD, PhD, MPH Centers for Disease Control and Prevention Division of Viral Hepatitis NCHHSTP/CDC Vaccine Research and Policy Unit, National Center for HIV/AIDS, Viral Hepatitis, STD, and TB Prevention 1600 Clifton Road, MS-G37, Atlanta, GA 30333, USA Tel:+1 404 718 8576 - Fax: 404-718-8595 Email: xdg9@cdc.gov, nnelson@cdc.gov |

#### 3. Project Summary

This is a phase III, placebo controlled, double blind, randomized clinical trial to assess the efficacy and safety of tenofovir disoproxil fumarate given from 28 weeks' gestation until 2 months postpartum to pregnant women with HBsAg/HBeAg-positive Hepatitis B virus (HBV) chronic infection in Thailand to prevent perinatal transmission of HBV to their infants who receive HBV passive-active immunization.

Chronic hepatitis B (CHB) infection is complicated by cirrhosis and hepatocellular carcinoma (HCC), which is the 10<sup>th</sup> leading cause of death worldwide. In 2011, about 7% of Thai adults were HBsAg carriers. Universal immunization programs have dramatically reduced the prevalence of infection wherever they have been implemented.

Infant hepatitis B (HB) immunization and HB immune globulin (HBIg) administered at birth effectively prevents most mother-to-child transmission (MTCT) of HBV. However, according to published studies often with limited sample sizes, using various methods for the diagnosis of infection in infants, it is thought that about 12% of HBV highly viremic mothers transmit the virus to their infants, despite active and passive immunization. It is likely that HBIg has no effect on infection already established in utero.

The presence in blood of a hepatitis B virus antigen, HBe (HBeAg), is a marker of high viral replication. Studies have suggested that antiviral treatment at the end of pregnancy and during early postpartum can reduce the risk of transmission to the child. A potential limitation to this approach is the risk of hepatic disease exacerbation (flare) following discontinuation of antiviral treatment postpartum, and this risk has not been properly evaluated. No randomized clinical trials have adequately demonstrated the efficacy and safety of maternal antiviral treatment for HBV MTCT prevention, and this approach is not currently recommended by the Associations for the Study of Liver Diseases.

We hypothesize that a potent antiviral, tenofovir, can decrease HBV viral load in HBV infected pregnant women and therefore reduce the risk of late *in utero*, intrapartum and postpartum transmission before infants are definitely protected by passive-active immunization. We also hypothesize that only moderate flares will be observed after discontinuation of a short antiviral course (5 months). While the primary objective of the study is to assess the efficacy of tenofovir versus placebo for the prevention of perinatal transmission, an important secondary objective is the assessment of the risk of postpartum hepatic disease exacerbation.

HBsAg positive pregnant women will be enrolled if they have a positive HBeAg test and ALT ≤30 U/L. They will be randomized to receive tenofovir or placebo from 28 weeks of pregnancy until 2 months postpartum. Within 2 years, 328 women and their infants will be enrolled from 19 public hospitals in Thailand where the health care teams have considerable experience in conducting trials for the prevention of mother to child transmission of HIV over the past 15 years. Mothers and infants will be followed until one year postpartum.

The primary endpoint will be the detection of HBsAg and HBV DNA in infants at six months of life. An interim analysis will be conducted when half of the outcomes are available.

The results of the study will help define policy to manage HBV infected pregnant women to prevent perinatal transmission.

สถาบันพัฒนาการคับกรองการวิจัยในบนุษย์ (สกม

#### 4. Background information

# 4.1. Epidemiology

An estimated 250 to 350 million people are chronically infected with the HBV worldwide [1], of whom over 100 million are in Asia [2]. The risk of adverse outcome from chronic HBV infection may approach 25% for cirrhosis and hepatocellular carcinoma (HCC). Chronic hepatitis B (CHB) is the 10<sup>th</sup> leading cause of death worldwide with 600,000 to 1.2 million deaths per year due to cirrhosis and HCC [3]. The prevalence of HBsAg, a marker of chronic infection, varies widely worldwide. Forty-five percent of the world's population lives in highly endemic countries, with prevalence of HBsAg ≥8%. In Thailand, an estimated 7%-8% of the adults born before 1992 (which includes most child-bearing women), when the national pediatric anti-HBV immunization program began, are chronic HBsAg carriers [4].

## 4.2. Hepatitis B virus

HBV is present in blood, saliva, semen, vaginal secretions, and to a lesser extent, perspiration, breast milk, tears, and urine. HBV is easily transmitted through contact with infected body fluids, and unprotected sexual activities. HBV, a prototype member of the Hepadnaviridae family, is a small (3.2 kb), partially double-stranded DNA virus. The hepatocytes represent the main target of HBV infection although the receptor for HBV is still unknown [5]. During active replication, viral particles are found in serum: the 42 nm complete virion and the empty viral envelopes made of HBsAg in the form of either the 22 nm sphere or filamentous forms [6, 7]. During highly replicative phases, a soluble antigen, HBeAg, is also found in serum, and is used as a marker of high replication.

Ten HBV genotypes (A to J) are known [8-12]: C and B predominate in Asia [13, 14] (Thailand 85% C and 15% B). Genotype C, compared to B, is associated with later and less sustained HBeAg seroconversion [15, 16], more hepatic necro-inflammation, more rapid progression to cirrhosis, and higher incidence of HCC [17-20].

#### 4.3. Natural history

The natural history of HBV infection differs according to the age of acquisition.

- In areas of low HBV endemicity, most infections are acquired in early adult life through sexual transmission or intravenous drug use [21]. The cytotoxic immune reaction is responsible for destruction of hepatocytes and increase in ALT, hyperbilirubinemia and jaundice and, in some cases, liver failure and death. In a minority of adults, HBV infection becomes chronic with HBsAg carriage [22, 23].
- In areas of high or intermediate endemicity, most transmissions occur in utero or during delivery when the newborn is exposed to maternal blood and contaminated secretions, or during the first years of life through contact with infected parents, siblings or other children. Without immunization, about 10% of infants born to HBsAg carrier mothers are found infected by one year, and 90% of these become HBsAg chronic carriers. Twenty-five to 30% of children infected between 1 and 5 years of age, develop chronic infection. The World Health Organization (WHO) recommends that HBsAg positive mothers breastfeed their infants based on studies finding similar rates of HBV infection in breastfed compared to bottle fed children [24].

There are 4 phases of chronic infection whose length depends on the age at HBV acquisition and HBV genotype: (1) "Immunotolerant" with minimal inflammation, (2) "Immune active" corresponding to chronic active disease and risk of progression to cirrhosis and liver cancer; (3) "Non-replicative" and (4) "HBeAg-negative chronic active" due to pre-core or core promoter mutants with progression to cirrhosis and liver cancer.

0913161 08 ปีค. 2558 คณะกรรมการจริยธรรมการวิจัยในมนุษฮ สภาบันพัฒนาการคับภรองการวิจัยในมนุษฮ์ (สคม.

While most carriers infected during adulthood eventually lose HBeAg and develop antibodies to HBeAg (anti-HBeAb), the vast majority of infected children enter in an immune tolerant phase with normal ALT levels and a rate of clearance of HBeAg much lower than in adults. The age at which HBeAg is lost varies with genotypes, and areas of the world: in Asia, about 40% of adult HBsAg carriers are HBeAg positive and about 10% outside Asia. In Asia, some HBV infected subjects test negative for HBeAg regardless of the level of HBV replication, due to a mutation in the pre-core region of HBV, which prevents the production of HBeAg [25], or a mutation in the basic core promoter (at nucleotides 1762 and 1764) [26-28]. However, among 52 HBsAg positive and HBeAg negative Thai pregnant women, we found only 2 with a HBV viral load > 6 log<sub>10</sub> IU/mL [29].

#### 4.4. Antiviral treatment of HBV infection

Since, in most cases, chronic HBV infection is not cleared, the goal of therapy is primarily to decrease the risk of cirrhosis and HCC. Current therapy uses interferon-alpha and nucleos(t)ide analogues. Interferon inhibits viral replication and acts as an immunomodulator. It is used as a short-term treatment that, when successful, may lead to long-term immune control without the need for further antiviral therapy. In contrast, it is considered that nucleos(t)ide analogs, which inhibit HBV replication, cannot usually be discontinued. While resistance mutations have been described in patients receiving long term treatment with lamivudine, emtricitabine, telbivudine, entecavir, and adefovir, they have not been reported for tenofovir [30, 31].

Studies have shown that interferon therapy or lamivudine therapy (with maintained virological response) reduce the risk of cirrhosis or HCC. Long term studies with other antiviral drugs are not available. However, the optimal time for starting therapy also depends on the risk of drug toxicity, development of resistance mutations and hepatic flares—liver inflammation indicated by ALT elevation—after discontinuation of therapy. The American Association for the Study of Liver Diseases (AASLD) [32] and Asian Pacific Association for the Study of the Liver (APASL) [33] recommend treatment for patients with an ALT level >2 ULN, and liver biopsy to guide treatment decisions if ALT is 1-2 x ULN, particularly if the age is >40 years. The recent European Association for the Study of Liver Diseases (EASL) [34] recommends therapy in patients with significant fibrosis, and ALT above the upper limit of normal or HBV DNA > 2000 IU/mL. Current guidelines recommend lifelong treatment except when HBeAg seroconversion and undetectable HBV-DNA have been documented. In HBeAg-negative patients, treatment discontinuation can be considered if undetectable HBV-DNA has been documented on three separate occasions 6 months apart [33].

The selection of tenofovir disoproxil fumarate (TDF) as the antiviral agent used in this study was based on safety, efficacy and cost considerations. Tenofovir is very potent anti HBV drug (median serum HBV DNA reduction after 1 year of treatment 6.2 log<sub>10</sub> copies/mL in HBV-infected HBeAg positive patients). It has been approved for HIV treatment and for HBV treatment for several years. Tenofovir has a high genetic barrier to resistance [31]. In previous studies, up to 192 weeks of tenofovir monotherapy, no mutations have been associated with resistance to tenofovir (genotypic and phenotypic analyses). [Viread Package insert, Gilead, Revised: January 2012]Previous studies have shown that the bioavailability and tolerance profile of tenofovir during pregnancy is favorable [35, 36]. No dose adjustment is currently recommended for TDF during pregnancy.

It is part of WHO recommended drug combinations to be started in HIV infected pregnant women after 14 weeks' gestation and continued through the breastfeeding period to prevent mother to child HIV transmission [37]. The US FDA classifies tenofovir in B. The risks for the fetus associated with the use of tenofovir during pregnancy are discussed below. Tenofovir crosses the placenta barrier with the potential added possible benefit of pre-exposure prophylaxis in the fetus and infant. Tenofovir crosses the placenta barrier with the potential added possible benefit of pre-exposure prophylaxis in the fetus and infant. The tenofovir form is excreted in the breast milk but a very low portion of it is absorbed by the infant. Indeed, a recent study estimated that the infant receives 0.03% of the proposed dose for neonates [38].


011171 08 ปีค. 2558 กณะกรรมการจริยธรรมดารวิจัยในมนุษย

#### 4.5. HBV infection during pregnancy and postpartum

HBV seems to have little effect on pregnancy but HBV viral load increases in pregnancy, probably in relation to immune-suppression and increased production of adrenal corticosteroids, estrogen and progesterone [39, 40]. Some women may experience increased in liver disease activity [41], with or without HBeAg seroconversion (HBeAg clearance occurred in 5 of 30 women in a study in Taiwan [42]), within the first months after delivery, presumably in relation with the rapid post-partum decrease in immunosuppression. See also "Antivirals administered to the mother" in Section 4.7.)

WHO [24] and Thai guidelines recommend HBV infected mothers to breastfeed as there is no evidence of additional transmission during breastfeeding.

#### 4.6. Perinatal transmission of HBV in the era of HBV immunization

WHO recommends universal perinatal HBV immunization, regardless of maternal HBV status. This strategy decreases perinatal transmission of HBV by 90-95% [43-46]. Since 1992, Thailand has integrated HBV vaccination in the national Expanded Program on Immunization (EPI). The recommended immunization schedule in Thailand is within 24 hours of birth (monovalent formulation), 2, 4 and 6 months (polyvalent formulations) [47], and an extra dose of monovalent HB vaccine is recommended at 1 month of age in infants born to HBsAg positive mothers (following the observation that infections occurred in infants whose 2-month dose was delayed [48]. As in Taiwan and Malaysia where this program has been implemented, a dramatic reduction in the prevalence of HBsAg carriers in children has been observed [49, 50]. However, a study in Thailand has shown that still 0.7% of children who have received immunization are HBV chronically infected [51].

HB Immune globulins (HBIg) at birth in infants born to HBsAg positive mothers. Administration of HBIg in addition to vaccine for infants born to HBsAg carriers, can halve the risk of transmission [52]. The injection of HBIg, in addition to vaccine, is thus recommended in newborns born to HBsAg+ mothers by the Royal College of Thai Pediatricians. Due to price (\$40 to \$130 depending on manufacturer) and short shelf life (up to one year), HBIg is actually not always available in Thai public hospitals. Moreover, although donors are tested for several known pathogens, concerns remain about the risk of transmission of unknown blood borne pathogens.

However, the combination of hepatitis B vaccine and HBlg does not protect all infants, in particular those born to mothers with high HBV replication (usually HBeAg positive). Such infants are at a significant risk of becoming HBV infected despite passive-active immunization, [53-55] mainly through in utero transmission, which may contribute to residual transmission of HBV.

In previous clinical studies, the rates of transmission in infants/children born to HBsAg and HBeAg positive mothers despite the use of HBlg at birth and HBV immunization have been variable, probably in relation with the various definitions and methods of diagnosis, as well as the quality of follow-up. In two studies evaluating the efficacy of antiviral prophylaxis the rates of transmission were:

- 7/88 (8%, 95% confidence interval [CI] 3% to 16%) HBsAg+ and HBV DNA + in infants at 7 months of age in China [56],
- 5/41 (12%, CI 4% to 26%) HBsAg+ in infants at 52 weeks of age in a randomized clinical trial in China and the Philippines [57] and 9/41 (22%, CI 11% to 38%) using HBV DNA.

In addition, the report of a meta-analysis [58], based on non-randomized studies mainly published in Chinese journals and the Xu's study [57], provides rates of HBsAg+ between 9 and 12 months in infants who received vaccine and HBlg at birth: 5/35 (14% CI 5% to 30%) (Han 2005), 7/44 (16%, CI 7% to 30%) (Li 2006), 16/42 (38%, CI 24% to 54%) (Feng 2007),



6/42 (14%, CI 5% to 29%) (Yang 2008), 2/19 (11%, CI 1% to 33%) (Yang 2008). However, this meta-analysis did not provide an overall single estimate of the transmission rate. Finally, in a recent cross sectional study conducted in Taiwan [59] in children of less than 2 years of age, 8 of 70 had HBsAg+ (11%, CI 5% to 21%). A reliable estimate of the transmission rate despite the use of HBlg at birth and HBV immunization cannot be drawn from these studies, owing the limited number of infants in each study and the methodological information provided.

#### 4.7. Additional interventions to potentially prevent perinatal transmission

#### 4.7.1. Elective C-section

A systematic review of 4 studies conducted in China involving 789 women showed a favorable effect of elective C-section performed before labor and rupture of membranes, consistent with the hypothesis that a significant part of transmission occurs at the time of delivery [60]. There is no published report on the efficacy of C-section in a setting where passive-active immune prophylaxis has been provided to infants.

Elective C-sections are not currently recommended for the prevention of HBV transmission.

#### 4.7.2. HBlg during pregnancy

According to a meta-analysis of 37 studies, the administration of HBIg during pregnancy in HBsAg carrier women may decrease intrauterine transmission and the rate of infection at one year of age [61]. However, this intervention is not recommended by WHO or other organizations, owing to the cost and limited production of HBIg and limited efficacy data.

#### 4.7.3. Antivirals administered to the mother

In HBsAg positive women, the reduction of HBV DNA load by nucleos(t)ide analogue therapy at the end of pregnancy may be effective and safe in reducing the risk of child vaccination breakthrough. Three studies, summarized below, have provided preliminary data.

# 4.7.3.1. Efficacy

- a) Study by van Zonneveld et al, 2003 [62]. In an open label study conducted in the Netherlands, 8 children born to 8 pregnant women (6 Caucasians and 2 Blacks, no Asians) who received 150 mg of lamivudine daily from 34 weeks' gestation until delivery were compared to 25 historical controls born to 24 mothers (4 Asians). All mothers had high HBV-DNA loads (>150 pg/mL using a hybridization technique no longer used, i.e. around 10<sup>8</sup> copies/mL). All infants received passive-active immunization. HBV DNA, HBsAg, anti-HBs and anti-HBc were measured in infants at birth and at 3, 6 and 12 months. At 12 months, 1 of the 8 infants (12.5%) was still HBsAg and HBV-DNA positive in the lamivudine group, versus 7 of the 25 controls (28%).
- b) Study by Xu et al, 2009 [57]. This multicenter study conducted in China and the Philippines was originally designed as a randomized, double-blind, 3arm, placebo-controlled trial, with an expected sample size of 410 highly HBV viremic pregnant women. Subjects were to be randomized in a 2:2:1 ratio to one of the three arms: (A) maternal lamivudine 100 mg once daily from 32 weeks of gestation until one month postpartum + infant passiveactive immunization; (B) maternal placebo + passive-active immunization; or (C) maternal lamivudine + vaccine but without HBIg. However, arm C was removed early during the study due to ethical concerns and the study faced a number of challenges. Firstly only 155 women were enrolled. Only 56 infants in the lamivudine group and 59 in the placebo group received passive active immunization. A large and unbalanced number of infants were lost to follow up: 13% in the lamivudine arm and 31% in the placebo arm. More than 50% of the women had serum HBV DNA >1000 MEq/mL (using bDNA assay, about 108 IU/mL) at baseline. At week 52, 3 of the 49 infants evaluable (6%) in the lamivudine group versus 5 of 41 infants in the placebo


group (12%) had evidence of HBV transmission at one year of age (P=0.368). However, from the intent to treat analyses where missing outcomes were considered as failures, the authors concluded that there was a significant decrease in HBsAg infection in infants born in the lamivudine group (10/56 versus 23/59, P=0.014). There were no safety concerns although some women experienced flares.

c) Study by Han G et al, 2011 [56]. This was a prospective, non-randomized, open-label study of telbivudine during pregnancy for the prevention of perinatal HBV transmission. HBeAg+ women with HBV DNA load >10<sup>7</sup> copies/mL were invited to choose either to receive 600 mg/day telbivudine from 20-32 weeks' gestation through week 4 after delivery or no treatment, and all infants received passive-active immunization. 187 women were enrolled: 94 chose to take telbivudine and 92 no treatment. The two groups had similar characteristics but 11% in the telbivudine group had received previous antiviral treatment versus 0% in the control group. At baseline, the mean HBV DNA load was 8.07 log<sub>10</sub> copies/mL versus 7.94 log<sub>10</sub>; at delivery, HBV DNA was below 1,000 copies/mL in 30% versus 0%, respectively. At week 28, in an intent-to-treat analysis where missing outcomes were considered as failures, 2% of infants were considered HBsAg positive in the telbivudine group, compared with 13% in the control group (p=0.004). The actual percentages were 0% and 9%, respectively.

Recently, a retrospective study in the US reported that 11 infants born to 11 mothers who received tenofovir disoproxil fumarate starting at 29 weeks' gestation were all HBsAg negative at age 28-36 weeks of age [63]. In addition, a prospective open label study in Nanjing, China, reported that, of 88 HBeAg+ pregnant women receiving telbivudine, with levels of HBV DNA 6 log<sub>10</sub> copies/mL, and increased levels of ALT, none transmitted HBV to their infants [64].

In summary, it is not possible to draw solid efficacy conclusions from the first two lamivudine studies [57, 62] described above due to obvious methodological flaws. The third study by Han et al [56], although not randomized, suggests that an antiviral administered during pregnancy, in addition to passive-active immunization, may decrease HBV transmission.

## 4.7.3.2. Safety

a) Safety of a 5 month tenofovir course in pregnant / lactating women

The short- and long-term effects of TDF on pregnant and breastfeeding women, fetuses and children is a key research gap identified in the WHO Guidelines. These include bone effects on both the woman and HIV-exposed infant [65].

## a.1) TDF renal toxicity in pregnant women

The main safety concern related to TDF treatment is its long-term renal toxicity, which has been described in HIV-HBV co-infected patients on multidrug combination therapy. However, it is not expected that such toxicity will be observed in HBV mono-infected women receiving this drug for 5 months. In 152 HBV mono-infected Asian patients, no increase of serum creatinine >0.5 mg/dl or of eGFR<50 ml/min was found in up to 3 years of TDF treatment [66].

The effect of tenofovir on bone metabolism seems related to its renal toxicity, which may lead to a syndrome similar to the Fanconi syndrome that involves the proximal tubules of the kidneys, with hyperphosphaturia and hypophosphatemia affecting bone metabolism. During pregnancy, the mother provides phosphate and calcium to the fetus. As the toxicity may be dose dependent, there is a need to quantify maternal tenofovir exposure and renal disturbances during pregnancy in perinatal studies.

Tenofovir exposure may cause maternal proximal renal tubular dysfunction and modification of calcium-phosphorus metabolism, resulting in lower maternal and/or infant BMD persisting until one year after delivery/birth. The relationship between maternal tenofovir exposure and infant/maternal low bone mineral density has never been studied in exposed HIV-uninfected

**0 143.161** 0 8 MA 2558 naznssuntsosustsuarsõõuluuuse pregnant women and their infants. Within this study, there is a unique opportunity to clarify the relationship between tenofovir exposures and maternal and infant bone mineral density.

#### a.2) TDF Bone toxicity

Maternal bone metabolism during pregnancy and the lactating period is regulated through complex mechanisms that ensure the infant bone growth, involving the supply of large amounts of calcium by the mother, and minimize maternal consequences for the maternal bones.

Few clinical trials have compared the effect of tenofovir versus placebo on bone mineral density as tenofovir is mostly prescribed to HIV-infected individuals. A study, conducted in the US, randomly assigned adolescents chronically infected with HBV to either TDF or placebo for 72 weeks and showed that no patients met the safety endpoint of a 6% decrease in spine bone mineral density at week 72 [67]. A pre-exposure prophylaxis study in HIV uninfected men in San Francisco also compared TDF versus placebo. The study found a small but statistically significant decrease in mean BMD in the TDF vs. the pre-treatment/placebo group at some bone sites (femoral neck, hip, L2–L4 spine) [68]. Of note, a pooled analysis of two studies comparing TDF versus adefovir found no differences in loss of bone mineral density between Asian and non-Asian patients infected with HBV on TDF [69].

Maternal bone resorption seems necessary to provide significant amounts of calcium to the baby but this may result in a decrease in maternal bone mineral density in some bones. As TDF may cause hyperphosphaturia and hypophosphatemia, and secondary changes in bone resorption, the composition of the breast milk may be altered, which may in turn impact the bone mineral density of the infant.

## b) Safety of antiviral discontinuation given to HBV infected pregnant women

During the course of HBV infection, acute exacerbations of liver inflammation or hepatic flares can occur spontaneously, be induced by IFN-a therapy or the discontinuation of treatment with nucleos(t)ide analogues. The AASLD defines "flares" as intermittent elevations of aminotransferase activity to more than 10 times the upper limit of normal and more than twice the baseline value (for this study, flares will be defined as ALT elevations above 300 IU/L, regardless of baseline values). Flares are also observed during induced immune suppression, which favors viral replication. They are most often preceded by high levels of HBV replication and by progressive accumulation of HBV antigens.

In 2000, Honkoop et al [70] reported that seven of 41 (17%) patients monitored for at least 6 months after discontinuation of lamivudine therapy experienced hepatitis flares. ALT peak occurred at a median 16 weeks (range 7-44 weeks) after withdrawal of therapy. Two of these cases (5%) were associated with jaundice and liver failure. Among the 9 patients with cirrhosis at start of therapy, one developed a severe hepatic flare. High HBV-DNA levels were seen at the time of the ALT peak. Hepatitis after withdrawal of lamivudine resembled acute hepatitis B with a predominance of an icteric flares within a time frame of 6 months.

Flares have been also observed within the first 4–8 weeks of tenofovir treatment, accompanied by decreases in HBV DNA levels but there have been no reports of hepatic decompensation in this setting. ALT flares typically resolved within 4 to 8 weeks without changes in therapy [Tenofovir Package Insert, Gilead, 2010].

In the first perinatal study described above, van Zonneveld et al [62] reported that SGPT/ALT levels increased in seven of eight women receiving lamivudine, but remained below 5 times the upper limit of normal (ULN) in all women and below 2 ULN in five of eight women after a follow-up of 1 to 7 months.

In the second study by Xu et al [57], two subjects in the placebo group experienced an increase in ALT: in one case, ALT reached 21 ULN, with no bilirubin increase, at six weeks postpartum, then decreased to 2 ULN at 12 weeks postpartum; in the second case, ALT increased to 16–18 ULN with bilirubin >2.5 ULN at the end of study treatment (placebo) and persisted until 6 weeks after delivery, then ALT decreased to baseline levels with bilirubin


0 8 ปีเค. 2558

คณะกรรมการจริยธรรมการวิจัยในมนุษย์

สถาบันพัฒนาการวังเกษตาการวิจัยในหนุษย์ (สคน

remaining elevated (1.8 ULN). During treatment and follow-up, Grade III/IV ALT elevations occurred in 22/89 (25%) of the mothers in the lamivudine group and 30/61 (49%) in the placebo group. After treatment discontinuation (week 4 postpartum) up to 12 weeks postpartum (end of maternal follow-up), one or more Grade III/IV ALT elevations first occurred in 16/83 (19%) mothers in the lamivudine group (3–5 ULN for 14 of the 16) and 15/46 (33%) mothers in the placebo group (3–5 ULN for 11 of the 15). One subject in each group had ALT levels increased to >10 ULN following treatment cessation. This is difficult to interpret because the rate of loss to follow up was higher in women on placebo, and the follow up after discontinuation of lamivudine was limited to 12 weeks post-partum, probably too short to adequately evaluate the risk of flare.

As for the third study reported by Han et al [56], only 36 of 94 women discontinued telbivudine at 4 weeks postpartum as per protocol. ALT elevations, 2-5 ULN occurred in 13% of women who discontinued therapy in the treated arm and 18% in the control arm. No cases of severe hepatitis flares (ALT >10 x ULN) were reported. Also, the follow up after treatment discontinuation was too short to fully assess the risk of flare and the reasons for treatment continuation in the majority of women were not reported. We did not find any other study adequately designed for a rigorous assessment of flares after discontinuation of antiviral treatment used for the prevention of HBV perinatal transmission in young pregnant women with a positive HBeAg test.

#### c) Safety in infants

Tenofovir is classified B in the FDA Pregnancy Category. Reproductive studies performed in rabbits and rats at doses up to 19 and 14 times the human dose, respectively, have shown no evidence of harm to the fetus. Of 1370 HIV infected women with first trimester use registered in the Pregnancy ARV registry [71], there have been no evidence of an association between major teratogenic effects and the use of tenofovir during pregnancy.

Tenofovir crosses the placental barrier [36]. Since the end of the 1990's, studies have raised concerns about possible mitochondrial dysfunction associated with in utero exposure to nucleoside reverse transcriptase inhibitors to prevent HIV perinatal transmission [72-74]. However, these disorders have been described in infants exposed in utero to nucleoside analogues (such as zidovudine or lamivudine) and born to HIV infected mothers. To our knowledge, such disorders have never been reported with the use of the nucleotide reverse transcriptase inhibitor, tenofovir.

Based on animal studies where high doses of TDF were administered, other safety concerns for TDF during pregnancy were raised about fetal/infant growth, bone mineralization and renal function. A study in Africa concluded that there was no evidence that *in utero* tenofovir affected growth after 2 years [75]. Another study in the US found that TDF use during pregnancy was not associated with increased risk for LBW or SGA but a slightly lower mean length-for-age z-scores and head circumference-for-age at one year age in TDF-exposed infants, of uncertain significance [76]. Recent data on bone mineralization and renal function in utero exposed infants found no impairment of growth and bone health [77]. A study conducted in the US in the context of the IMPAACT network recently reported the lack of effect of tenofovir in utero exposure and weight at birth and at 6 months of age (82).

DXA scans in newborns have been found accurate [78]. The ionizing radiation exposure from a scan is extremely low, indeed within the range of "negligible" annual individual dose as recommended by the National Council of Radiation Protection and Measurements (NCRP). There are no DXA measure norms for infants but measurements obtained using Hologic scanners have been shown reliable enough to compare groups of infants [79, 80], which will be the case for the proposed investigations.

<sup>&</sup>lt;sup>2</sup>Category B: Animal reproduction studies have failed to demonstrate a risk to the fetus and there are no adequate and well-controlled studies in pregnant women OR Animal studies have shown an adverse effect, but adequate and well-controlled studies in pregnant women have failed to demonstrate a risk to the fetus in any trimester.



TDF is currently recommended by WHO HIV treatment guidelines as part of one of the preferred drug combinations in pregnant women after 14 weeks' gestation and continued throughout breastfeeding. In the US Recommendations for Use of Antiretroviral Drugs in Pregnant HIV-1-Infected Women [81]. TDF is recommended and is the preferred NRTI choice for women who are co-infected with hepatitis B virus.

Finally, the recent 2012 Asia Pacific Association for the Study of the Liver (APASL) guidelines states that telbivudine or tenofovir can be used in mono HBV infected pregnant women [82].

#### 4.7.4. Conclusion

In summary, no interventions in addition to active-passive HBV immunization of the newborn are recommended to fully prevent perinatal transmission of HBV from mothers with high HBV viral loads. This remains an obstacle to HBV eradication.

Elective C-section and use of HBIg during pregnancy may be efficacious but they are associated with logistic complications and risks.

Previous studies of antivirals have failed to provide clear efficacy and safety data: two of the published studies were not randomized, and the other was randomized but not completed as planned; and none offers adequate information on the risk of hepatic flare in women after discontinuation of therapy. This placebo-controlled study is designed to formally test the concept in a rigorous manner and to provide data on the efficacy of a short maternal course of antiviral prophylaxis and the safety of antiviral discontinuation in mothers. Tenofovir disoproxil fumarate is approved by the Thai FDA in Thailand for HBV chronic infection treatment but not for the prevention of perinatal transmission. Due to the lack of such data, there are currently no or only weak recommendations for this approach by the Associations for the Study of Liver Diseases, the WHO or national health authorities in America, Europe and Asia, Moreover, the recent 2012 APASL Guidelines stated that previous studies "have shown that antiviral therapy administered in late pregnancy may further reduce the risk of perinatal HBV infection from highly viremic mothers, as compared with passive-active immunization alone. However, the extent of benefit, the threshold of serum HBV DNA level for initiating therapy, the optimal time to start therapy, the appropriate choice of antiviral agent, and the optimal duration of therapy have not been determined." [82]

The study results could change clinical practice for pregnant women living with HBV in Thailand and throughout the world.

#### 4.8. Sub-studies

The data and samples collected in this study may be a source for sub-studies regarding immune response during and after discontinuation of antiviral treatment (in particular analyzing immunologic and gene expression changes taking place before the occurrence of flares, using viable PBMC and total RNA from whole blood collected in the study), HBV resistance and other aspects, including HBV and host genetics. None of these sub-studies are included in this protocol. Specific protocols will be developed and submitted to ethics committees, and funding sought separately.

## 5. Study objectives

## Primary objective

1. To assess the efficacy of tenofovir disoproxil fumarate, versus placebo, in HBV infected HBsAg and HBeAg positive pregnant women, from 28 weeks' gestation until 2 months postpartum (5- month course) to prevent perinatal transmission of HBV to their infants who receive HBV passive-active immunization.

 0 8 ปี.A. 2558

**Hypothesis**: an anti-HBV agent, tenofovir disoproxil fumarate (TDF) administered from the beginning of the last trimester of pregnancy to two months postpartum to HBV infected, HBeAg-positive, pregnant women with ALT ≤30 U/L will reduce the risk of *in utero*, *intrapartum* and early *postpartum* transmission to their infants from 12% to 3% or less.

## Secondary objectives

- To assess the safety of tenofovir disoproxil fumarate administered for 5 months perinatally in HBsAg and HBeAg positive women with ALT ≤30 U/L, and their in utero exposed infants.
- 2. To compare the risk of acute exacerbation or flare (ALT >300 U/L) up to 12 months postpartum, following planned discontinuation of study treatment, in HBeAg positive women randomized to tenofovir disoproxil fumarate or placebo.

The following secondary objectives have been added in Protocol Version 3.0.

**Hypothesis**: Tenofovir exposure causes maternal proximal renal tubular dysfunction and modification of calcium-phosphorus metabolism, resulting in lower maternal and/or infant BMD persisting until one year after delivery/birth.

- 3. To compare the bone mineral density (BMD) at 12 months postpartum in HBV chronically infected, breastfeeding mothers, randomized to receive TDF or matching placebo from 28 weeks gestational age to 2 months postpartum.
- To compare the bone mineral density (BMD) in infants at 12 months of age whose mothers were randomized to receive TDF or matching placebo within the iTAP clinical trial.

#### Design

The design of the study is a multicenter, controlled, double blind, randomized clinical trial to assess the efficacy to prevent hepatitis B virus (HBV) perinatal transmission, safety and tolerance of tenofovir disoproxil fumarate versus placebo, given from 28 weeks' gestation until 2 months post-partum to hepatitis B sAg and eAg positive mothers.



Figure 1. Overview of the randomized trial design with 12 month follow-up

U F6 30 V 8 0 8 19 ค. 2558 คณะกรรมการจริยธรรมการวิจัยในหนุษย์ สถาบันพัฒนาการ (และการาชวิจัยในหนุษย์ (สคม. We opted for a design where antiviral drug will be discontinued because it is not currently recommended to start chronic antiviral treatment in case of ALT level < ULN, even with high replication. We considered that a two month postpartum treatment would ensure that the infant is protected from a maternal transmission until three vaccine injections have been administered.

The study will involve a population of subjects easy to identify using tests widely available in Thailand (with HBsAg+, HBeAg+, ALT ≤ 30 U/L), at high risk of transmission but in the immune tolerant phase and, therefore, at lower risk of liver enzyme elevation after discontinuation of treatment.

# 6. Study sites and duration of the study

## 6.1. Study sites

PHPT affiliated Obstetrics, Internal Medicine and Pediatrics Departments in Thai public hospitals have been highly trained in conducting clinical research on prevention of perinatal transmission of HIV, and have been participating in NICHD and NIAID/DAIDS sponsored studies for the last 15 years. Each site is regularly monitored by a PHPT clinical research assistant to ensure that study procedures are implemented according to the protocol and regulations.

| Site | FWA |
|-----------------------------------------------|-------------|
| Phayao Provincial Hospital | FWA00001646 |
| Chiangrai Prachanukroh Hospital | FWA00001607 |
| Prapokklao Hospital | FWA00001643 |
| Chonburi Hospital | FWA00001604 |
| Bhumibol Adulyadej Hospital | FWA00001651 |
| Health Promotion Center Region 10, Chiang Mai | FWA00001608 |
| Lamphun Hospital | FWA00002135 |
| Chiang Kham Hospital | FWA00001609 |
| Mae Chan Hospital | FWA00001619 |
| Banglamung Hospital | FWA00001610 |
| Nakornping Hospital | FWA00001605 |
| Nopparat Rajathanee Hospital | FWA00002134 |
| Khon Kaen Hospital | FWA00001612 |
| Samutsakhon Hospital | FWA00001644 |
| Nakhonpathom Hospital | FWA00001606 |
| Samutprakarn Hospital | FWA00002128 |
| Lampang Hospital | FWA00007260 |
| Maharaj Nakornratchasrima Hospital | FWA00007370 |
| Ranong Hospital* | On process |

<sup>\*</sup> Ranong Hospital after formal approval by the sponsor (NICHD and US CDC, USA).

04119 0 8 W.A. 2558 site, the approximate number of patients to be enrolled per site is as follows:

Considering the data currently available regarding prevalence of HBV chronic infection in each

Site Estimate number of patients to be enrolled Phayao Provincial Hospital 8 Chiangrai Prachanukroh Hospital 56 25 Prapokklao Hospital 8 Chonburi Hospital Bhumibol Adulyadej Hospital 8 Health Promotion Center Region 10, Chiang Mai 30 8 Lamphun Hospital 8 Chiang Kham Hospital 8 Mae Chan Hospital Banglamung Hospital 36 8 Nakornping Hospital 30 Nopparat Rajathanee Hospital Khon Kaen Hospital 24 Samutsakhon Hospital 20 Nakhonpathom Hospital 5 16 Samutprakarn Hospital 10 Lampang Hospital Maharaj Nakornratchasrima Hospital 10

Ranong Hospital\*

Total

Study co-investigators and study nurses will be trained before the beginning of and during the study to the specific aspects of Hepatitis B management and treatment. The pediatric nurses will receive refresher training at the outset to ensure that length, weight, head circumference are recorded in a standardized way.

10

328

The PHPT Clinical Trial Unit (CTU) team is responsible for the overall organization and monitoring of the study, as well as data entry, data management and statistical analysis in compliance with Good Clinical Practices and reporting to the sponsors. The technical team in charge of the study at the CTU will be composed of 1 junior physician, 1 coordinator, 1 nurse in charge of the safety monitoring, at least 4 full-time-equivalent clinical research assistants, 1 data manager, 3 data entry technicians, 1 laboratory technician, 1 logistician, 1 translator and


0 9 9 19 19

0 8 19 A. 2558

กณะกรรมการจริย์ธรรมการวิจัยในบนุษย์

สถาบันพัฒนาการกับอรกงการวิจัยในบนุษย์ (สก)

<sup>\*</sup> Ranong Hospital after formal approval by the sponsor (NICHD and US CDC, USA).

1 secretary. In addition, the PHPT CTU pharmacist will oversee the management of study drugs.

Site co-investigators are responsible for the medical management of the patients, the implementation of the study interventions according to the protocol and the completion of the Case Report Forms (CRFs). At each site, the study teams consist of obstetricians, pediatricians, nurses, laboratory technicians, pharmacists and counselors.

The completed CRFs are reviewed and signed by the site co-investigator and forwarded to the CTU. Upon arrival at the CTU, they are immediately recorded in a tracking database and filed. The tracking database provides updated information on each patient every week, as well as the total number of patients at each stage of follow-up.

Data will be keyed using a double data entry system, and programs check the datasets for range checks on each field within a form, consistency checks between fields on the same form, and between fields on different forms. The data managers generate queries as necessary until final validation of the CRFs. Validated CRFs serve as evidence that the history and clinical data has been recorded, and that all lab tests and procedures have been completed. All serious adverse events will be reported according to GCP. As required by GCP, any change made to the original CRFs/data set is fully documented. The databases are stored in My-SQL format in central computers with restricted access and regular backups are made and stored in another place to prevent accidental loss of data. All important operations are described in procedures within our IRD UMI 174 quality management system, accredited according to the standards of ISO 9001:2008.

As for previous studies conducted by our group, investigators and co-investigators will facilitate any audit of the data, procedures at study sites and at the laboratory by independent external monitors sent by sponsors.

The PHPT laboratory has received ISO accreditation 15189: 2007. It is responsible for the centralized laboratory exams, virological testing, and samples repository. The blood samples will be stored at the central laboratory for retrospective assessments as needed.

The PHPT laboratory staff will also monitor the quality control of the site laboratories.

#### 6.2. Duration of the study

First enrollment: December 1, 2012
Planned enrollment duration: 24 months

Approximate duration of maternal follow up from enrollment to delivery: 3 months

Postpartum and infant follow up: 12 months

Planned date of last visit completed: March 31, 2016

Final analysis and submission of a manuscript: last quarter 2016.

# 7. Workplan

#### 7.1. Selection of participants

#### 7.1.1. Eligibility criteria

The population enrolled in the study will be composed of pregnant women meeting all eligibility and inclusion criteria, and none of the exclusion criteria, and their infants.

Women who meet the eligibility criteria (see Table1, below) will be systematically approached, informed about HBV perinatal transmission and about the study, and proposed participation in the study. If they agree, they will be asked to sign the Study Informed Consent Form before any study procedures (see Appendix 1).


คณะกรรมการจริยธรรมการวิจัยในมนุษย์ สถาทันพัฒนาการกับกรดสถารวิจัยในมนุษย์ (สคน



Figure 2: Selection of participants

Table 1: Eligibility Criteria

| 1 | Pregnancy |
|---|---|
| 2 | Age: at least 18 years |
| 3 | Negative Human Immunodeficiency Virus (HIV) serology test performed less than 3 months prior to enrollment. |
| 4 | HBsAg test positive performed less than 6 months prior to enrollment. |

# 7.1.2. Inclusion and exclusion criteria

Women who meet all inclusion criteria (see Table 2) and none of the exclusion criteria (see Table 3) will be offered enrollment in the study.

Table 2: Inclusion Criteria

| 1 | Gestational age of 28 weeks (+ or – 10 days) as determined by obstetrician. |
|---|---|
| 2 | Positive HBeAg test performed less than 6 months prior to enrollment. |
| 3 | ALT/SGPT ≤30 U/L performed less than 3 months prior to enrollment and confirmed ≤60 U/L at the Pre-Entry visit. |


**01/1/17**0 8 ปี.ค. 2558
คณะกรรมการจริย์ธรรมการวิจัยในมนุษย์

Written informed consent for participation in this study.

Agreeing to bring their infants at the planned study visits at one study site until one year after delivery and to inform the site investigators if they plan to move to another place and not be able to return to the clinic.

Understanding the need for adequate infant immunization and agreeing to the blood

Understanding the need for adequate infant immunization and agreeing to the blood draws from their infants and the need for close follow up to manage possible exacerbation of hepatitis.

#### Table 3: Exclusion criteria

| 1 | History of tenofovir at any time, or any other anti-HBV treatment during the current pregnancy. |
|---|---|
| 2 | Creatinine clearance <50 ml/min, calculated using the Cockcroft-Gault formula (Appendix 4). |
| 3 | Dipstick proteinuria>1+ (>30 mg/dL) or normoglycemic glucosuria confirmed on two separate occasions. |
| 4 | Positive serology for Hepatitis C infection less than 12 months prior to enrollmen |
| 5 | Evidence of pre-existing fetal anomalies incompatible with life. |
| 6 | Any concomitant condition or treatment that, in the view of the clinical site investigator, would contraindicate participation or satisfactory follow up in the study. |
| 7 | Concurrent participation in any other clinical trial without written agreement of the two study teams. |

As part of the consent process, participants will be asked for their authorization to record laboratory test results performed as part of their clinical care before their formal consent to participate in this study.

#### Infant inclusion criteria

• All live born infants, born to mothers participating in this study.

#### Infant exclusion criteria

· Stillbirth.

## 7.1.3. Discontinuation criteria

## Maternal and infant discontinuation criteria

Women enrolled in the study are free to withdraw their or their infants' participation in the study at any time without jeopardizing their access to standard medical care or possible participation in future research studies.

Pregnant women and their infants will continue to be followed in the study, regardless of maternal adherence to study treatment.

A study site co-investigator may decide to end a subject's participation in the study if, in his/her own judgment, such a participation would be detrimental to a subject's health or well-being. However, all efforts should be made to inform the study team and discuss options prior such a decision.

0 9 13 16. 2558 คณะกรรมการจริยธรรายการวิจัยในมนุษย์ สถาบันพัฒนาการกุ้มสารคาร "ผู้เกินมนุษย์ (สคม Study **treatment** discontinuation: a site co-investigator in charge of the patient's care may consider, if possible after discussion with the study team, discontinuing double blind study treatment if he/she considers that a patient is experiencing toxicity that could be caused by tenofovir. In such a case, the patient should continue follow up in the study.

The study could be discontinued if required by Thailand health authorities or the sponsors.

## 7.2. Implementation, data collection and monitoring procedures

#### 7.2.1. Maternal follow up

Eligibility and pre-enrolment tests should be performed within the previous 3 months prior to enrollment. After enrollment, maternal visits will be performed at 28, 32, 36 weeks' gestation, delivery, and at 1, 2, 3, 4, 6 and 12 months postpartum (see scheduled assessments in Table 4).

Study treatment will be provided every month from 28 weeks' gestation through 2 months postpartum. All effort should be made to strictly follow the maternal and infant visit schedule but occasional departures of no more than one week will be considered acceptable.

For future sub-studies, in participants enrolled in sites with PBMC isolation capacity, PBMC will be isolated at the enrollment visit, prior to starting study treatment, and at 32, 36 weeks gestation, and at 1, 2, 3 and 4months postpartum and kept stored in liquid nitrogen until use for laboratory analyses. Total RNA from whole blood will be collected at the same visits.

#### Urine sample collection

Tenofovir has been associated with renal function impairment in HIV infected patients. In this study, participants are not HIV infected. In addition to the routine serum creatinine and phosphorus measurements already planned in the protocol, a maternal urine sample will be collected at study entry, at the 32 weeks' gestation visit, at time of study treatment discontinuation (visit scheduled at 2 months postpartum) and at the last maternal visit. Some urinary biomarkers, for example Kidney injury molecule-1, Neutrophil gelatinase associated lipocalin, have been found earlier indicators of proximal tubular injury, compared to traditional markers. After centrifugation, aliquots will be stored frozen. The samples could be used for individual investigation in case of serum creatinine elevation. If deemed necessary, a systematic analysis of the samples will be described in a separate protocol, which will be submitted for ethical approval and for funding.



Table 4: Maternal assessments

| Maternal assessments | Antepartum | | | | | Delivery | | Postpartum (months) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Scr<br>een<br>ing | Pre-<br>entry | Enroll<br>ment<br>28 wks | 32<br>wks | 36<br>wks | | Before<br>discharge | 1 | 21 | 3 | 4 | 6 | 12 <sup>2</sup> |
| | | | | | Study | treat | tment | | | | | | |
| Counseling and Questionnaire | Х | Х | Х | Х | X | Х | | Х | Х | Х | Х | Х | Х |
| Physical/Obstetric exam | Х | Х | | Х | Х | Х | | Х | Χ | Х | Χ | Χ | Х |
| Study treatment dispensation, return of used study treatment bottles/adherence assessment | | | Х | Х | Х | Х | | Х | Х | | | | |
| Record results of HBsAg, HIV serology and Ultra sound | Х | | | | | | | | | | | | |
| SGPT/ALT | Х | Х | | Х | Х | X | | Х | Х | Х | Х | Х | Х |
| HBeAg test | | | | | | | | | | | - | | |
| (if negative during postpartum period, anti-HBeAb will be tested) | Х | | | | | | | | Х | | | | Х |
| Complete Blood Count <sup>3</sup> | | Х | | | | Х | | | X | | | | |
| Serum SGOT/AST, bilirubin<br>(direct& conjugated), alkaline<br>phosphatases, albumin | | X | | | | | | | | | | | Х |
| Hepatitis C serology | | Х | | | | | | | | | | | |
| Serum creatinine <sup>4</sup> | | Х | | Х | Х | Х | X | Х | Х | | X <sup>5</sup> | | |
| Serum phosphorus | | Х | | X | Х | Х | | Х | Х | | Х | | |
| Dipstick glycosuria and proteinuria | | Х | | Х | | Х | | | Х | | | | |
| Urine sample collection <sup>8</sup> | | | Х | Х | | | | | Χ | | , | | X |
| DXA assessment | | <u> </u> | | | | | | | | | | | X <sup>10</sup> |
| HBV DNA load (retrospective) | | | Х | | | X <sup>6</sup> | | X <sup>6</sup> | | | | | |
| Tenofovir plasma level | | | | X <sup>9</sup> | X <sub>9</sub> | X | | | | | | | |
| Plasma/serum storage | X | Х | X | Х | Х | X | X | Х | X | Х | X | X | X |
| RNA storage | | | Х | Х | Х | | | Х | X | Х | X | | |
| PBMC isolation <sup>7</sup> | | | Х | Х | Х | | | Х | Х | Х | Х | | |
| Total blood volume (mL) | 5 | 16 | 3 | 10 | 10 | 10 | 4 | 8 | 13 | 8 | 8 | 8 | 10 |
| Total blood volume for PBMC(mL) <sup>7</sup> | | | 30 | 30 | 30 | | | 30 | 30 | 30 | 30 | | |
| Cord blood volume (mL) | | | | | | 15 | | | | | | | |

In case of liver enzyme exacerbation (see section 7.2.2 liver enzyme exacerbations below), additional immediate, prospective, and retrospective evaluations on stored samples will be performed: AST/SGOT, ALT/SGPT, gamma-glutamyl-transferase, alkaline phosphatase, total bilirubin and albumin and HBV DNA load.

Laboratory procedures for serum HBV quantitation, HBsAg test in infants for diagnosis purpose, Anti-HBs Ab, and determination of tenofovir plasma concentrations will be described in the Manual of operations.

With patient's authorization, study teams will record contact information including mobile phone number and address (this information will not be entered in the study databases) to be used if she does not show up at a visit for contact and possible home visit by the hospital social workers. All patients starting study treatment will be introduced to a gastroenterologist or internist experienced in management of Hepatitis B, for future long term care. Women will be asked to report any concomitant treatments at all follow up visits. Women wishing to withdraw from the study will be referred to a specialist in Hepatitis B management in a public hospital as close as possible to her dwelling. In case of early discontinuation, the investigator will ask the mother the authorization to perform a last mother and infant blood draw for safety evaluations and for documentation of the infant's HBV status (see Tables 4 and 5).

Grade 3 and 4 abnormalities as defined by the NIAID Division of AIDS in the Table for Grading the Severity of Adult and Pediatric Adverse Events (Version 1.0, December, 2004) will be reported immediately to the PHPT Clinical Trial Unit (CTU). Any serious adverse event, as defined by ICH Good Clinical Practice (GCP) [83], whether or not considered to be related to the study treatment, will be also reported within 3 business days to the Thai Ministry of Public Health and the drug manufacturer (following requirements).

Management of toxicities will be discussed and reviewed with the site study teams during on-site trainings organized prior to starting the study, and described in detail in the Manual of onsite Operations. The PHPT CTU staff can be reached 24 hours a day through phone, and by fax and e-mail. At each visit, the study nurse in charge will record the history and the results of the physical exam, record and grade adverse experiences. Concomitant treatments and medical interventions, including details about mode of delivery, will be recorded in CRFs.

#### 7.2.2. Liver enzyme exacerbations

After delivery, women will be closely followed up until one year postpartum and any confirmed elevations of SGPT/ALT will warrant consideration for prompt re-introduction of study treatment. There is no evidence that HBV exacerbation depends on the level of replication at the time of discontinuation; thus women in the post-treatment phase will be primarily monitored based on SGPT/ALT levels.

0 9 19 10 1 2558 กละกรรมการกริยธรรมการวิจัยในบนุษย์ สถาบันพัฒนาการจัดการ (พ. โมมนุษย์ (สกม

<sup>&</sup>lt;sup>1</sup>Or early study treatment discontinuation

<sup>&</sup>lt;sup>2</sup>Or early study discontinuation (if subject consents)

<sup>&</sup>lt;sup>3</sup>Including platelet count;

<sup>&</sup>lt;sup>4</sup>Calculatecreatinine clearance using the Cockcroft-Gault formula (see Appendix 4) or online calculation at http://nephron.com/cgi-bin/CGSl.cgi).

<sup>&</sup>lt;sup>5</sup> In case of Grade 1 or higher creatinine at 2 months postpartum

<sup>&</sup>lt;sup>6</sup>Funding will be sought to retrospectively measure HBV DNA load in women who transmitted HBV and a control sample of women who did not, at time of delivery and 1 month postpartum.

<sup>&</sup>lt;sup>7</sup>For women enrolled in sites with PBMC isolation capacity (flares sub-studies)

<sup>&</sup>lt;sup>8</sup>If possible, a urine sample of 10 ml will be collected at study entry, at the 32 weeks' gestation visit, at time of study treatment discontinuation (visit scheduled at 2 months postpartum) and at the last maternal visit to evaluate the potential renal toxicity of tenofovir. After centrifugation, 10 aliquots will be stored frozen.

<sup>&</sup>lt;sup>9</sup> For women who consent for the pharmacokinetic sub-study

<sup>&</sup>lt;sup>10</sup> For women who consent for the DXA assessment sub-study

Women will be informed of possible adverse effects following discontinuation of antiviral treatment without medical supervision or imperfect adherence. In case of liver enzyme elevation, additional visits and tests will be performed for case management and documentation.

In case of SGPT/ALT >60 U/L, with or without associated symptoms, a clinical assessment of the subject will be performed and SGPT/ALT will be repeated on another blood draw as soon as possible and within 3 days, along with the following laboratory examinations: bilirubin, prothrombin/INR, and albumin. Plasma will be stored for further evaluations: HBV DNA load, HBeAg and antibodies and other viruses as appropriate. The site investigator will immediately inform a PHPT CTU physician by phone, at any time (24/24 hours, 7/7 days).

- If SGPT/ALT is confirmed between 60 and 150 U/L, a new SGPT/ALT test will be scheduled 2
  weeks later. The patient's contact information will be checked before the patient leaves the clinic and
  the patient informed that she should return to the clinic if she has any clinical symptoms.
- If SGPT/ALT >150 U/L is confirmed immediately, or if SGPT/ALT is confirmed between 60 and 150 U/L two weeks after the first test, the site investigator will contact a PHPT CTU physician and reintroduction of double blind study treatment will be considered by the reference site internist.



Figure 3: Flow diagram of postpartum flare management

Patients restarting antiviral treatment will be followed within the study until one year after delivery. After the end of the patient's participation in the study, her treatment will be replaced with the commercial form of the drug originally assigned (except if it was placebo), and followed off study by the reference internist according to current guidelines within the Thai Universal Health Coverage system. Patients will not discontinue antiviral treatment during their participation in the study but discontinuation may later be considered according to current APASL recommendations [33].

# 7.2.3. Assessment of Maternal Tenofovir Plasma Exposure

Two extra blood samples will be drawn in a subset of women to measure study drug concentrations at the 32 week and 36 week maternal visits. Women will be asked to sign an additional consent form to


**อายุมร์**0 8 ปี.ค. 2558
คณะกรรมการจริยธรรมการวิจัยในบนุษย
สถาบันพัฒนาการกุ้มครองการวิจัยในบนุษย์ (สคม.

join the sub-study (see Appendix 6. Additional consent form for plasma drug level measurements). These samples will be collected between 0.5 to 3 hours post-dose and between 3 to 6 hours post-dose (at least 1 hour after the previous sample). A population pharmacokinetic model will be used to estimate tenofovir exposure in all women.

## 7.2.4. Bone Mineral Density Evaluations

In sites with access to DXA scan equipment, the option for DXA scan evaluations in mothers and infants will be explained to women at their 6-month maternal visit, and/or at the 9 month infant visit. The examinations will be explained in detail, including their practical aspects (need for specific appointments, transfer to the DXA scan facility). Women who consent will be asked to sign an additional consent form.

Consenting women will have DXA scans of their hip and lumbar spine at 12 months postpartum.

For this study, a <u>Hologic Discovery A</u> DXA scan (Software Version: 4.0.2) is currently available at 3 locations:

- Maharaja Nakorn Chiang Mai Hospital, Chiang Mai University;
- Bhumibol Adulyadej Hospital, Bangkok;
- Maharaja Nakhonratchasima Hospital, Nakhonratchasima.

Each woman/infant pair will be accompanied by a study staff.

We have estimated that a total of 98 women <u>could</u> have DXA scan measurements one year after delivery/birth, over a 1 year period.

## 7.2.5. Infant follow up and diagnosis of HBV infection

All infants will receive anti HBV passive immunization (HBIg) within 12 hours of birth (at a site different from the HBV vaccine), and intensive active immunization following Thai national guidelines for infants born to HBsAg positive mothers, i.e. within 12 hours of birth and at 1, 2, 4 and 6 months of age. Infant visits will be performed at birth, 1, 2, 4, 6 and 12 months for clinical safety evaluation and determination of HBV status.

A check list of signs and conditions suggesting possible mitochondrial dysfunction that may trigger other investigations will be completed at the 6 and 12 month visit (see list in Appendix 3)



Table 5: Infant assessments

| Infant assessments | Birth | 1<br>month | 2<br>months | 4<br>months | 6<br>months | 9<br>months | 12<br>months <sup>1</sup> |
|---|---|---|---|---|---|---|---|
| Physical examination including length, weight and head circumference <sup>2</sup> | Х | Х | Х | Х | Х | Х | Х |
| Mitochondrial dysfunction check list <sup>3</sup> | | | | | Х | | Х |
| Counseling and Questionnaire | Х | X | Χ | Χ | Х | Х | Х |
| Record date and time of HB Immune globulin (HBIg) injection <sup>4</sup> | Х | | | | | | |
| Record date and time of HB immunization | Х | Х | Х | Х | Х | | |
| Complete Blood Count | Х | | | | | | Х |
| Serum creatinine | Х | | | | | | |
| Serum phosphorus/calcium | Х | | | | | | |
| HBsAg <sup>1,5</sup> | X <sup>5</sup> | X <sup>5</sup> | $X^5$ | X <sup>5</sup> | X <sup>5</sup> | Χ | Х |
| HBV DNA <sup>1</sup> | Х | | | | X <sup>6</sup> | Х | X <sup>6</sup> |
| SGPT/ALT | Х | | | | | | X <sup>6</sup> |
| Anti-HBsAb | | | Х | Х | Х | Х | X <sup>7</sup> |
| HBeAg and anti-HBeAb if positive HBsAg | • | | | | | | Х |
| DXA assessment | | | | | | | X <sup>8</sup> |
| Plasma storage | X <sup>5</sup> | X <sup>5</sup> | X <sup>5</sup> | X <sup>5</sup> | X <sup>5</sup> | X <sup>5</sup> | Х |
| Total blood volume (mL) | 3 | 3 | 2 | 2 | 3 | 3 | 4 |

Additional investigations if HBsAg+ (except at birth): retrospective HBV DNA loads, HBeAg ¹Or early discontinuation, with mother's/guardian's/parents' consent.

<sup>8</sup> For infants who consent for the DXA assessment sub-study

# Diagnosis of HBV infection in infants

The significance of a positive HBsAg or HBV DNA test within the first days of life is unclear as some infants may test negative a few weeks or months later [84, 85]. Blood will be systematically drawn before vaccine administration.

In this study, for the interim and final analyses, HBV transmission will be defined by a positive HBsAg and positive HBV DNA at 6 months of age. All infants will be tested for HBV DNA at birth and at 9 months of age, regardless of HBsAg test results.

Appropriate laboratory analyses (HBV DNA and HBeAg) will be conducted retrospectively to determine the timing or clearance of infection in HBV DNA negative cases at 6 months with a positive HBsAg test at any time. Secondary analyses will include HBV transmission as defined by a positive HBsAg and positive HBV DNA through 12 months of age.

## Bone Mineral Density Evaluations in Infants

In infants from sites where DXA scan evaluations are accessible, these evaluations will be explained to mothers at the occasion of the 6-month maternal visit, and/or at the 9 month infant visit, including their




<sup>&</sup>lt;sup>2</sup>Including Ballard Score at birth. See also Appendix 5: How to Measure Head Circumference, Length and Weight.

<sup>3</sup> Assessment for possible mitochondrial dysfunction: see list of major and minor neurological and other organ signs in Appendix 3.

<sup>&</sup>lt;sup>4</sup>InjectHBIg at a site different from HBV vaccine.

<sup>&</sup>lt;sup>5</sup>Draw blood before injection of HBIg and vaccine.

<sup>&</sup>lt;sup>6</sup> If HBsAg positive at this time point

<sup>7</sup> If anti-HBs < 10 IU/L (and HBsAg/HBV DNA negative), the pediatrician in charge will be encourage to consider revaccination.

practical aspects (See above BMD in Mothers). <u>Infants</u> will have a DXA scan of their lumbar spine at 12 months of age.

# 7.3. Study drugs

Patients will receive study drugs (tenofovir disoproxil fumarate 300mg tablet or indistinguishable matching placebo) in the form of tablets manufactured by Gilead for clinical trials.

For information, tenofovir disoproxil fumarate is commercialized in Thailand:

Trade name: Viread®

Generic name: tenofovir disoproxil fumarate tablets

Manufacturer's: Gilead Sciences, Inc.

Distributor's: IDS Marketing (Thailand) Limited

Registration number of drug license: 1C 144/2549(NC)

Study drugs (TDF and placebo) will be provided by Gilead Sciences, Inc, in the form of bottles of 30 tablets. The PHPT CTU pharmacist will organize the labeling ("secondary packaging") of the study drugs in collaboration with the study statistician, in accordance to regulations. Each individual study treatment bottle will be uniquely identified and dispensation of study drugs will be documented. The details will be provided in the Manual of Operations.

#### 7.4. Statistical considerations

## 7.4.1. Endpoints

## 7.4.1.1 Primary Endpoint

 Infant's HBV infection status, defined as HBsAg positive confirmed by HBV DNA, at 6 months of age.

Note: transmission to one or more offspring of a multiple pregnancy will be considered as only one transmission.

## 7.4.1.2 Secondary Endpoints

- Occurrence of maternal and infant adverse events (AE), including ICH SAEs and DAIDS grade 3/4 signs and symptoms, regardless of their relatedness to the study treatment.
- Occurrence of acute exacerbation or flare of hepatitis B, following planned discontinuation of study treatment up to 12 months postpartum. The acute exacerbation or flare of hepatitis B is defined as ALT >300 IU/L regardless of baseline values.
- Infant's HBV infection status, defined as HBsAg positive confirmed by HBV DNA, at or after 6
  months through 12 months of age.
- Infant growth related outcomes, including weight, height and HC Z-scores at 6 months and 12 months of age.

# 7.4.2. Randomization and Stratification

Participants will be randomized 1:1 to receive TDF or placebo stratified by site using permuted blocks of size determined by the study team. Subjects' baseline HBV viral load, which might affect transmission rate, is unavailable in real time and cannot be stratified. The imbalance of baseline HBV viral load will be evaluated. If an imbalance exists, an exact logistic regression accounting for baseline HBV viral load will be conducted as a sensitivity analysis.

0 8 ปี A. 2558 คณะกรรมการจริยธรรมการวิจัยในมนุษย สถาบันพัฒนาการวันครจงการวิจัยในมนุษย์ (สณ.

#### 7.4.3. Sample size and Accrual

The sample size is calculated accounting for one interim efficacy monitoring between the TDF arm and the placebo arm. It is hypothesized that TDF will lower the transmission rate. To target 90% of power at a one-sided

0.049 significance level in Fisher's exact test, 312 evaluable neonates, 156/arm, are needed to detect an infection rate of 3% in the TDF arm, assuming 12% infection rate in the placebo arm. This is equivalent to a relative reduction of 75% in infection rate in the TDF arm. The table below summarizes the power of the study

if the infection rate in the placebo arm is lower than 12%, e.g., if the infection rate in the placebo arm is only 10%, the study has 83.2% of power to detect a 75% reduction in the infection rate, i.e., an infection rate at 2.5%, in the TDF arm. However, if the infection rate is only 8%, the power of detecting 75% reduction in the infection rate, i.e. 2% infection rate in the placebo arm, reduces to only 72.6%. Therefore the infection rate in the placebo arm needs to be considered carefully during the interim efficacy monitoring as outlined in the next section.

Table: Power of the study assuming different infection rate in the placebo arm (based on one-sided Fisher's exact test at 0.049 significance level)

| Power (156/arm) | Infection rate in the active treatment arms | | | |
|---|---|---|---|---|
| Infection rate in the placebo arm | 1% | 2% | 2.5% | 3% |
| 8% | 90.1% | 72.6% | 62.5% | 52.4% |
| 10% | 97.5% | 89.5% | 83.2% | 75.8% |
| 12% | 99.5% | 96.7% | 94.0% | 90.1% |

To further account for a maximum of 5% lost to follow-up, 328 pregnant women will be enrolled.

#### 7.4.4. Information of the co-investigators

To inform the co-investigators about the study and its progress, a meeting will be held before the beginning of the study, then every year. In addition, a monthly progress report, prepared by the data management team at the PHPT CTU, will be provided to all co-investigators, including the Program Scientists during the trial.

#### 7.4.5. Monitoring by the program scientists

Program scientists should be notified, within one week of protocol team awareness, of selected serious adverse events (maternal and fetal/infant), including:

- deaths:
- all Grade 4 adverse events (including hospitalizations; congenital anomalies (with the exception of those listed in Appendix 2); persistent or significant disability/incapacity.

Sites will be asked to include a description of the event, an assessment of potential relatedness to study drug (TDF), description of how the subject was managed, and final outcome. To discuss the progress of the study, a <u>quarterly</u> teleconference will be held including program scientists and the study coordination team (including at least the study principal investigator, virologist, pharmacologist, study nurse coordinator).

## 7.4.6. Data and Safety Monitoring Board (DSMB)

The Data and Safety Monitoring Board (DSMB) will be composed of at least 1 gastroenterologist/ hepatologist, 1 pediatrician, 1 obstetrician, 1 infectious diseases specialist, and 1 statistician/ epidemiologist, at least 3 of them Thais. The program scientists will participate as observers on open sessions of DSMB calls/meetings.

The study will be presented in detail to the DSMB during a protocol initiation review before study open. At this meeting, a detailed study monitoring plan, outlining open reports on study conduct and safety profiles pooled across study arms and closed reports on by-arm information and efficacy, will be presented.

The study will be monitored by the DSMB at least annually. First DSMB data review will be held when 100 pregnant women have been enrolled, or one year after the first enrollment. This meeting will allow for the review of the conduct of the study and Adverse Events (regardless of randomization). No efficacy analysis will be presented at this meeting. Additional DSMB reviews could be triggered if deemed necessary by the principal investigator, in particular in case of issues related to the occurrence of flares. DSMB could help program scientists with monitoring as a closed DSMB report would include by-arm information.

The first interim efficacy monitoring will be performed when 50% of information on the primary endpoint is available, i.e. when 164 infants either have their 6 month HBV status available or are off study before the 6 month visit. A Haybittle-Peto use function will be employed for the group sequential design. At the interim efficacy monitoring, the comparison of the primary endpoint will be considered significant only if p < 0.001. In addition, sensitivity analysis considering any positive HBsAg, confirmed by HBV DNA, at or after month 6 up to 12 months of age as having a neonate HBV infection will be provided. Futilities will also be considered based on conditional powers, safety profiles of the treatment arm and possible low transmission rate in the placebo arm. Details will be provided in the study monitoring plan. Additional interim efficacy monitoring could be considered in conjunction with the DSMB, and the final analysis for the comparison between TDF and the placebo arm will employ an alpha level of 0.05 - N \* 0.001, where N represent the number of interim efficacy monitoring throughout the entire statistical consideration section.

In case of premature discontinuation of the clinical trial for any reasons, further management of patients will be organized with the advice of the DSMB and health authorities.

## 7.4.7. Analyses for the primary objective/endpoint

Proportions of neonates, who have HBV infection at 6 months of age, along with their 95% confidence intervals, will be provided by arm based on exact Binomial distribution and compared between the TDF arm and the placebo arm based on Fisher's exact test. The tests will be adjusted for the interim efficacy monitoring by considering p < 0.05 – N \* 0.001as significant. The imbalance of mother's baseline HBV viral load between treatment arms will be evaluated based on Wilcoxon rank sum test. If imbalance exists, an exact logistic regression will be conducted as a sensitivity analysis. The primary analysis will be conducted as a complete case analysis including infants whose 6 month endpoint is available in their original randomized group, regardless of the duration of study treatment the mothers actually received if at least one dose was taken. A secondary analysis will be conducted in a modified intent to treat (mITT) population, where all randomized pregnant women who received at least one dose of study treatment, will be included and infants who are lost to follow-up before their 6 months HBV status is available will be considered as having an event. Further sensitivity analysis may be performed, including imputing infants' last available HBV infection status as their 6 months status for those who are lost to follow-up prior to 6 months or multiple imputations accounting for possible reasons of loss to follow-up, to explore the effect of loss to follow up. A secondary supporting analysis, considering any

014 11/21 08 ปี ค.ศ. 2558 คณะกรรมการจริชธรรมดารวิจัยในมนุษย เเถาบันพัฒนาการศ์มลงองการวิจัยในมนุษย์ (สคม. positive HBsAg, confirmed by HBV DNA, at or after 6 months up to 12 months of age as having a neonate HBV infection, will be conducted in the complete case population. Logistic regressions, accounting for factors that are known to be associated with mother-to-child HBV transmission could also be conducted to provide an adjusted odds ratio between treatment arms.

As indicated in literature, the significance of a positive HBsAg or HBV DNA test within the first days of life is unclear as some infants can test negative a few weeks or months later. Time to first HBsAg positive will not be considered in the primary analyses.

## 7.4.8. Analyses for secondary objectives/endpoints

7.4.8.1 Proportions of women with severe hepatic disease exacerbation or flare from study treatment discontinuation up to 12 months postpartum, along with their 95% confidence interval, will be provided by

treatment arm and compared between treatment arms based on exact binomial distribution and Fisher's exact test. Flares will be defined as ALT elevations above 300 IU/L, regardless of baseline values.

- 7.4.8.2 Proportions of women with any adverse event (AE) from randomization until study exit will be analyzed similarly as those specified in section 7.4.8.1. Poisson regressions, with an offset of follow-up time will be further conducted to model repeated occurrence of AE.
- AEs in infants will be analyzed in a similar manner.
- 7.4.8.3. Infants' mean weight, height and HC z-scores at 6 and 12 months, along with their 95% confidence intervals, will be provided by treatment arm and compared between arms based on normal approximation and two-sample t-test.

## 7.4.9. Pharmacokinetic data to estimate individual maternal tenofovir exposure

For each participant mother, a plasma sample will be available for PK analysis during pregnancy at Week 32 and 36 GA study visits (328 samples). It is expected that half of those women (164) will receive TDF. To ensure samples are available within the early part of the dosing interval an additional two timed samples will be collected in approximately 44 women at week 32 and 36 GA study visits (88 samples). Overall, we expect a total of 208 samples from 164 women will be available to develop a population pharmacokinetic model.

The tenofovir plasma concentration data available will be pooled to generate the population pharmacokinetic model. Non-linear mixed effects regression (NONMEM) will be used to estimate the population means and variances of tenofovir pharmacokinetic parameters. Individual patient characteristics will be evaluated for their inclusion in the model using a stepwise forward inclusion and backward elimination model building procedure. Post-hoc subject specific PK parameters will be estimated (i.e. AUC,  $C_{12}$  and  $C_{24}$ ). The approach will be similar to that we used to develop a population pharmacokinetic model in HIV-infected adults receiving TDF containing antiretroviral therapy [86].

## 7.4.10. Bone mineral density measurements

Sample size estimate for BMD measurement: additional investigations will start after approval by ethical review committees and training of radiologists. All women who deliver after May 15, 2014 will have their 12-month postpartum visit (window of 1.5 months) after July 1, 2015 and are therefore eligible to participate. Taking into account that enrollment and delivery are about 3 months apart, a maximum of 231 women can be eligible for DXA evaluation.

A recent study provides data on the expected lumbar spine bone mineral density (BMD) in infant of 1 year of age (mean  $\pm$  SD): 0.312  $\pm$  0.070 g/cm<sup>2</sup> [87]. An older paper provided a similar estimation: 0.446

**อาโมงา** กละกรรมการจรับสรรรมการวิจัยในมนุษย์ สถาบันพัฒนาการกุ้มครองการวิจัยในมนุษย์ (สคม ± 0.048 g/cm<sup>2</sup> [88], but we will prefer the newer one which derived from measurements with more recent DXA technology.

Assuming a lumbar spine BMD mean (standard deviation) of 0.312 g/cm<sup>2</sup> (0.070 g/cm<sup>2</sup>) in the control group, a sample size of 45 infants per arm would ensure a power of 80% to detect a 13.5% mean difference, i.e. 0.042 g/cm<sup>2</sup> between the tenofovir and placebo groups (two-sided test with  $\alpha$ =0.05). Assuming 5% un-evaluable cases, 47 infants and their mothers in each arm should undergo DXA scan assessments, i.e. a total of 94 mothers.

The relationship between maternal tenofovir exposure and one-year postpartum/age BMD measures will be studied using analysis of variance models, taking into account characteristics such as the duration of lactation.

## 7.4.11. Exploratory analyses

Proportions of infants with seroprotection, i.e., proportions of infants with anti-HBs > 10 IU/L, along with their 95% confidence intervals will be provided by treatment arm and compared between arms based on either normal approximation or the nonparametric method as appropriate for the data.

Proportions of premature labors (birth before 37 weeks of gestational age assessed by Ballard Score), associated or not with flares, along with their 95% confidence intervals, will be provided by treatment arm and compared between arms based on either exact method or normal approximation as appropriate for the data.

Additional analyses include, but not are limited to, analysis on time to treatment discontinuation and/or study discontinuation and analysis on adherence.

Details on these analyses will be further provided in the statistical analysis plan before their initiation.

#### f) Special considerations

The number, quality and frequency of blood collection, as well the tests to be performed on these samples, are specified in Tables 4 and 5.

## 8. Ethical considerations

#### 8.1. Possible risks including preventive or alleviative measures

## 8.1.1. Potential Risks to Participants

We hypothesize that there will be a significant reduction in the risk of HBV transmission to the fetus/infant born to women who receive tenofovir disoproxil fumarate during the last trimester of pregnancy and for two months following delivery, and this outweighs the risk of administering tenofovir to pregnant women and their fetuses in a carefully monitored trial.

Maternal risks associated with the use of tenofovir disoproxil fumarate (TDF) during pregnancy;

TDF is a nucleotide analogue which inhibits both HIV and HBV viral replication through inhibition of the virus reverse transcriptase. TDF is indicated for HIV treatment and HBV treatment, and is part of a WHO recommended drug combination to be started in HIV infected pregnant women after 14 weeks' gestation and continued through the breastfeeding period to prevent mother to child HIV transmission.

In subjects with chronic hepatitis B who participated in controlled clinical trials Gilead 0102 and 0103, more subjects treated with tenofovir during the 48-week double-blind period experienced nausea (9% versus 3% with adefovir) [89]. Other treatment-emergent adverse reactions reported in >5% of subjects treated with tenofovir included: abdominal pain, diarrhea, headache, dizziness, fatigue, nasopharyngitis, back pain and skin rash. No significant change in the tolerability\_profile (nature or


**อาเมรา** 0 8 ฟิฟิ 2558 คณะกรรมการจริยธรรมดารวิจัยในมพุษช severity of adverse reactions) was observed in subjects continuing treatment with tenofovir for up to 144 weeks in these studies.

Flares have been also observed within the first 4–8 weeks of treatment, accompanied by decreases in HBV DNA levels. No subject had evidence of decompensation. ALT flares typically resolved within 4 to 8 weeks without changes in therapy [Viread Package insert, Gilead, October 2010].

# · Maternal risks associated with discontinuation of antiviral treatment after delivery

During the course of HBV infection, acute exacerbations of liver damage or hepatic flares can occur spontaneously, be induced by IFN- $\alpha$  therapy or the discontinuation of treatment with nucleos(t)ide analogues. Flares are also observed during induced immune suppression, favoring viral replication. They are most often preceded by high levels of HBV replication and by progressive accumulation of HBV antigens.

The three perinatal studies presented above have provided more information on the risk of exacerbation after discontinuation of antiviral treatment for the prevention of HBV perinatal transmission:

In the study by van Zonneveld et al [62], ALT levels increased in seven of eight women who received lamivudine from 36 weeks' gestation to delivery, but remained below 5 times the upper limit of normal (ULN) in all women and below 2 ULN in five of eight women after a follow-up of 1 to 7 months.

In the second study by Xu et al [57], two subjects in the placebo group experienced an increase in ALT: in one case, ALT reached 21 ULN, with no bilirubin increase, at six weeks postpartum, then decreased to 2 ULN at 12 weeks postpartum; in the second case, ALT increased to 16–18 ULN with bilirubin >2.5 ULN at the end of study treatment and persisted until 6 weeks after delivery, then ALT decreased to baseline levels with bilirubin remaining elevated (1.8 ULN). During treatment and follow-up, Grade III/IV ALT elevations occurred in 22/89 (25%) and 30/61 (49%) of the mothers in the lamivudine and placebo groups, respectively. After treatment was discontinuation (week 4 postpartum) up to 12 weeks postpartum (end of maternal follow-up), one or more Grade III/IV ALT elevations first occurred in 16/83 (19%) mothers in the lamivudine group (3–5 ULN for 14 of the 16) and 15/46 (33%) mothers in the placebo group (3–5 ULN for 11 of the 15). One subject in each group had ALT levels increased to >10 ULN following treatment cessation. This is difficult to interpret because the rate of loss to follow up was higher in women on placebo, and the follow up after discontinuation of lamivudine was limited to 12 weeks post-partum, probably too short to adequately evaluate the risk of flare.

In the third study by Han et al [56], 36 of 94 women discontinued telbivudine at 4 weeks postpartum as per protocol. ALT flares 2-5 times the upper limit of normal occurred in 13% of women who discontinued therapy in the treated arm and 18% in the control arm. No cases of severe hepatitis flares (ALT > 10 x ULN) were reported. In this study, the duration of follow up was probably too short to fully evaluate the risk of flare after treatment discontinuation and the reasons for treatment continuation in the majority of women were not reported.

In the proposed study, we will follow the protocol used for registrational clinical trials for TDF (for the management of flares following discontinuation of antiviral treatment. Women will be informed of possible adverse effects following discontinuation of antiviral treatment without medical supervision or imperfect adherence. In case of liver enzyme elevation, additional visits and tests will be performed for case management and documentation. After delivery, women will be closely followed up until one year postpartum and any confirmed significant elevations of ALT will warrant consideration for prompt reintroduction of antiviral therapy (see Section 7.2.2. Liver enzyme exacerbations)

**อามาร** 0 8 ปีค. 2558 คณะกรรมการจริยธรรมการวิจัยในมนุษช
Infant risks associated with in utero exposure to tenofovir

Tenofovir is classified in category B of the US FDA. The data collected in the Antiretroviral in Pregnancy Registry show that there have been no increase in birth defects in 981 women exposed during the first trimester and 584 women during the second and third trimester (105). However, the Pediatric HIV/AIDS Cohort Study "Surveillance Monitoring of Antiretroviral Toxicity" (SMARTT), which enrolls HIV-exposed uninfected children in the US, recently reported a marginal increase in the risk of low length and weight z-scores at one year of age. However confounders may explain this finding. In the proposed study, the growth of the infants will be evaluated and compared between treatment arms. Prior to study commencement, a literature review will be performed to consider with the DSMB whether there is a need for additional evaluations.

Possible mitochondrial toxicity following exposure to nucleoside analogues in utero

Tenofovir is phosphorylated intracellularly to compounds which compete not only with the natural substrates for HBV reverse transcriptase but also with those for DNA polymerase gamma, the enzyme necessary for the replication of mitochondrial DNA.

Possible mitochondrial toxicity in children exposed to nucleoside analogues has been reported. Researchers observed an increase in febrile seizures in children in utero exposed to nucleoside [90]. The nucleoside safety review of perinatally-exposed children in US studies has revealed no excess deaths before the age of 5 that might represent toxic effects on the mitochondria among more than 20,000 infants assessed [91]. European and U.S. investigators have found small transient reductions in hemoglobin, and more persistent but clinically insignificant reductions in granulocytes, and lymphocytes associated with perinatal exposure to nucleoside reverse transcriptase inhibitors (NRTI). In 2007, Brogly and colleagues [74] conducted a retrospective review of the 1,037 HIV-uninfected children born in 1991–2002 and enrolled in Pediatric AIDS Clinical Trials Group protocols 219/219C and found 20 cases of possible cases with unexplained signs of mitochondrial dysfunction. Their analysis suggested that first exposure to lamivudine or lamivudine/zidovudine in the third trimester may be associated with the occurrence of possible mitochondrial dysfunction. However, to our knowledge, no cases of mitochondrial toxicity in children exposed to tenofovir in utero have been reported to date.

## 8.2. Adequacy of protection against risks

## 8.2.1. Recruitment and informed consent (see Consent Form in Appendix 1)

Nineteen clinical sites will participate in this study. All co-investigators have passed a training curriculum course on Human Subjects Protection. As for our previous studies, a specific training for the co-investigators, nurses and counselors will be conducted prior to the implementation of the study. Training will address the specific aspects of the study, the Good Clinical Practice (GCP) requirements, and procedures for protection of human subjects in clinical research, emphasizing issues related to vulnerable populations (pregnant women, fetus, newborns and children.

All pregnant women are screened for HBV infection in Thailand. In this study, if HBsAg positive, they will receive counseling and comprehensive information about HBV infection, the risk of transmission to their infants and the details of the proposed study and, following consent, further testing (HBeAg) to assess their individual risk of transmission. They will be enrolled in the study if they meet the selection criteria.

The consent form has been discussed, and reviewed with the PHPT CTU Community Advisory Board. At each site, a member of the study team will thoroughly discuss with each woman the information included in the consent. The consent form describes the purpose of the study, the procedures to be followed and the potential risks and benefits of participation. The consent document specifies the woman's freedom to withdraw her participation or the participation of her baby, at any time without

**014319** 0 8 U.A. 2558 narnssumssäusssumsääiluuyva

สถาบันพัฒนาการกับครองการได้ อนนุษย์ (สอน

compromising access to future medical care. Written informed consent from the father will also be obtained if possible, for the participation of the infant.

The consent form includes the names and contact details of the site co-investigator, whom the study participant may contact with any questions. A copy of the consent document will be given to the patient. In addition, study participants may contact personnel from the PHPT Clinical Trial Unit, 24 hours a day by phone. The original consent forms will be kept in a locked cabinet at the site. If new information relevant to the patient's consent or her willingness to continue participation in the trial becomes available, the participants and potential participants will be informed. Any changes to the consent document will be submitted to the relevant Ethics Committees.

## 8.3. Protection against risk

## 8.3.1. Institutional Review Board

Prior to the initiation of the study, the protocol and patient consent documents will be reviewed and approved by a national ethics committee at the Thai Ministry of Public Health, the Ethics Committee at the Faculty of Associated Medical Sciences, Chiang Mai University, and at each local hospital site. Subsequent modifications will be submitted for approval before implementation.

## 8.3.2. Expedited Adverse Experience Reporting

All clinical adverse events and abnormal laboratory values will be recorded and graded. For severe toxicity and serious adverse events, as defined by ICH GCP [83], possibly related to study drugs, an Expedited Adverse Experience Report (EAE) will be sent to the Thai Ministry of Public Health, Ethics Committees, and program scientists, within three business days of awareness. If a subject dies, events prior to and at the time of death will be transcribed from hospital records, and possible cause(s) of death will be investigated. Management of toxicities and dose modifications for patients will be managed with experts' advice.

#### 8.3.3. Confidentiality

Every effort will be made to maintain the confidentiality of the study participants. All site staff receive initial and ongoing training on Human Subjects Protection and confidentiality. To minimize this risk, study participants will not be identified by name on any study documents but will be identified by the provided patient identification number. All evaluation forms, laboratory specimens, reports and other records will be identified only by the patient identification number to maintain subject confidentiality. All records will be kept in a locked file cabinet in the clinical research unit. All computer entry and networking programs will be processed with patient identification number only. Clinical information will not be released without the written permission of the patient except when necessary for monitoring by the PHPT Clinical Trial Unit (CTU) or the sponsors.

#### 8.3.4. Biohazard Containment

As the transmission of HBV and other blood-borne pathogens can occur through contact with contaminated needles, blood, and blood products, appropriate precautions will be used by all personnel in the drawing of blood and shipping and handling of all specimens for this study, as currently recommended by the US Centers for Disease Control. All infectious specimens will be transported using requirements for shipping infectious substances.

Compensation, medical care and other services to be provided to the subjects who may be affected by any complication


O No Me Subjects who may be affected to the subjects who may be affected to the subject who subjects who s

When appropriate, mothers are reimbursed for transportation costs.

Policy Regarding Research Related Injuries:

Immediate necessary care is available free of charge to mothers and her infant in the case of medical problems related to participation in this study. However, the study is not responsible for treatments unrelated to the study and no financial compensation will be provided (see consent form Appendix 1).

Other related ethical aspects

The subject information sheet is written in Thai language, and physician or hospital's names, contact address and telephone number have been included.




กณะกรรมการจริยธรรมดารวิจัยในมนุษย์ สถาบันพัฒนาการคุ้มกรองการวิจัยในมนุษย์ (สคน 9. References

- 1. World Health Organization. Hepatitis B. Fact sheet N204. Revised August 2008. Available at:http://www.who.int/mediacentre/factsheets/fs204/en/. In: WHO; 2008.
- 2. Heathcote EJ. Demography and presentation of chronic hepatitis B virus infection. *Am J Med* 2008,121:S3-11.
- 3. Lavanchy D. Hepatitis B virus epidemiology, disease burden, treatment, and current and emerging prevention and control measures. *J Viral Hepat* 2004,11:97-107.
- 4. Tanprasert S, Somjitta S. Trend study on HBsAg prevalence in Thai voluntary blood donors. Southeast Asian J Trop Med Public Health 1993,24 Suppl 1:43-45.
- 5. Glebe D, Urban S. Viral and cellular determinants involved in hepadnaviral entry. *World J Gastroenterol* 2007,13:22-38.
- 6. Lee WM. Hepatitis B virus infection. N Engl J Med 1997,337:1733-1745.
- 7. Seeger C, Mason WS. Hepatitis B virus biology. *Microbiol Mol Biol Rev* 2000,64:51-68.
- 8. Kramvis A, Kew M, Francois G. Hepatitis B virus genotypes. *Vaccine* 2005,23:2409-2423.
- 9. Mahtab MA, Rahman S, Khan M, Karim F. Hepatitis B virus genotypes: an overview. Hepatobiliary Pancreat Dis Int 2008,**7**:457-464.
- 10. Olinger CM, Jutavijittum P, Hubschen JM, Yousukh A, Samountry B, Thammavong T, et al. Possible new hepatitis B virus genotype, southeast Asia. *Emerg Infect Dis* 2008,14:1777-1780.
- 11. Tatematsu K, Tanaka Y, Kurbanov F, Sugauchi F, Mano S, Maeshiro T, et al. A genetic variant of hepatitis B virus divergent from known human and ape genotypes isolated from a Japanese patient and provisionally assigned to new genotype J. *J Virol* 2009,83:10538-10547.
- 12. Tran TT, Trinh TN, Abe K. New complex recombinant genotype of hepatitis B virus identified in Vietnam. *J Virol* 2008,82:5657-5663.
- 13. Sa-Nguanmoo P, Tangkijvanich P, Thawornsuk N, Vichaiwattana P, Prianantathavorn K, Theamboonlers A, et al. Molecular epidemiological study of hepatitis B virus among migrant workers from Cambodia, Laos, and Myanmar to Thailand. *J Med Virol* 2010,82:1341-1349.
- 14. Zeng G, Wang Z, Wen S, Jiang J, Wang L, Cheng J, et al. Geographic distribution, virologic and clinical characteristics of hepatitis B virus genotypes in China. *J Viral Hepat* 2005,12:609-617.
- 15. Chu CJ, Hussain M, Lok AS. Hepatitis B virus genotype B is associated with earlier HBeAg seroconversion compared with hepatitis B virus genotype C. *Gastroenterology* 2002,122:1756-1762.
- 16. Livingston SE, Simonetti JP, Bulkow LR, Homan CE, Snowball MM, Cagle HH, et al. Clearance of hepatitis B e antigen in patients with chronic hepatitis B and genotypes A, B, C, D, and F. Gastroenterology 2007,133:1452-1457.
- 17. Lin CL, Kao JH. The clinical implications of hepatitis B virus genotype: Recent advances. *J Gastroenterol Hepatol* 2011,26 Suppl 1:123-130.
- 18. McMahon BJ. The influence of hepatitis B virus genotype and subgenotype on the natural history of chronic hepatitis B. *Hepatol Int* 2009,**3**:334-342.
- 19. Sumi H, Yokosuka O, Seki N, Arai M, Imazeki F, Kurihara T, et al. Influence of hepatitis B virus genotypes on the progression of chronic type B liver disease. *Hepatology* 2003,37:19-26.
- 20. Yang HI, Yeh SH, Chen PJ, Iloeje UH, Jen CL, Su J, et al. Associations between hepatitis B virus genotype and mutants and the risk of hepatocellular carcinoma. *J Natl Cancer Inst* 2008,100:1134-1143.
- 21. Lavanchy D. Chronic viral hepatitis as a public health issue in the world. Best Pract Res Clin Gastroenterol 2008,22:991-1008.


- 22. Dienstag JL, Hepatitis B virus infection. N Engl J Med 2008,359:1486-1500.
- 23. Liang TJ. Hepatitis B: the virus and disease. *Hepatology* 2009,49:S13-21.



- 24. World Health Organization. Hepatitis B and breastfeeding. A statement prepared jointly by the Global Programme for Vaccines and Immunization (GPV) and the Divisions of Child Health and Development (CHD), and Reproductive Health (Technical Support) (RHT) World Health Organization. No. 22, November 1996. In; 1996.
- 25. Carman WF, Jacyna MR, Hadziyannis S, Karayiannis P, McGarvey MJ, Makris A, et al. Mutation preventing formation of hepatitis B e antigen in patients with chronic hepatitis B infection. Lancet 1989,2:588-591.
- 26. Funk ML, Rosenberg DM, Lok AS. World-wide epidemiology of HBeAg-negative chronic hepatitis B and associated precore and core promoter variants. *J Viral Hepat* 2002,9:52-61.
- 27. Okamoto H, Tsuda F, Akahane Y, Sugai Y, Yoshiba M, Moriyama K, et al. Hepatitis B virus with mutations in the core promoter for an e antigen-negative phenotype in carriers with antibody to e antigen. *J Virol* 1994,68:8102-8110.
- 28. Tangkijvanich P, Theamboonlers A, Jantaradsamee P, Hirsch P, Mahachai V, Suwangool P, et al. Core promoter and precore mutants of hepatitis B virus: prevalence and clinical relevance in chronic hepatitis patients. Southeast Asian J Trop Med Public Health 2000,31:627-635.
- 29. Ngo-Giang-Huong N, Sirirungsi W, Boonprasit W, Khamduang W, Suwannachat B, Achalapong J, et al. Transmission of Hepatitis B Virus from HIV Co-infected Mothers to their Infants in Thailand. In: *The XV International AIDS Conference*. Bangkok, Thailand: MedGenMed, 2004 Jul 11;6(3):MoPeB3331 [eJIAS. 2004 Jul 11;1(1):MoPeB3331]; 2004.
- 30. Heathcote EJ, Marcellin P, Buti M, Gane E, De Man RA, Krastev Z, et al. Three-year efficacy and safety of tenofovir disoproxil fumarate treatment for chronic hepatitis B. Gastroenterology 2011,140:132-143.
- 31. Kwon H, Lok AS. Hepatitis B therapy. Nat. Rev. Gastroenterol. Hepatol. 2011, 8:275–284.
- 32. Lok AS, McMahon BJ. Chronic hepatitis B: update 2009. http://www.aasld.org/practiceguidelines/Documents/Bookmarked%20Practice%20Guidelines/Chronic\_Hep\_B\_Update\_2009%208\_24\_2009.pdf. Access 19-May 2011. *Hepatology* 2009.50:661-662.
- 33. Liaw YF, Leung N, Kao JH, Piratvisuth T, Gane E, Han KH, et al. Asian-Pacific consensus statement on the management of chronic hepatitis B: a 2008 update. *Hepatol Int* 2008,**2**:263-283.
- 34. European Association For The Study Of The L. EASL Clinical Practice Guidelines: Management of chronic hepatitis B virus infection. *J Hepatol* 2012,57:167-185.
- 35. Burchett S, Best B, Mirochnick M, Hu C, Capparelli E, Holland D, et al. Tenofovir Pharmacokinetics during Pregnancy, at Delivery and Postpartum. Abstract 738b. In: 14th Conference on Retroviruses and Opportunistic Infections. Los Angeles, CA, USA; 2007.
- 36. Hirt D, Urien S, Ekouevi DK, Rey E, Arrive E, Blanche S, *et al.* Population pharmacokinetics of tenofovir in HIV-1-infected pregnant women and their neonates (ANRS 12109). *Clin Pharmacol Ther* 2009.**85**:182-189.
- 37. World Health Organization. Antiretroviral therapy for HIV infection in adults and adolescents: recommendations for a public health approach.— 2010 rev. Accessed on 22 September 2010. In; 2010. pp. 44.
- 38. Benaboud S, Pruvost A, Coffie PA, Ekouevi DK, Urien S, Arrive E, et al. Concentrations of tenofovir and emtricitabine in breast milk of HIV-1-infected women in Abidjan, Cote d'Ivoire, in the ANRS 12109 TEmAA Study, Step 2. Antimicrob Agents Chemother 2011,55:1315-1317.
- 39. Ip HM, Lelie PN, Wong VC, Kuhns MC, Reesink HW. Prevention of hepatitis B virus carrier state in infants according to maternal serum levels of HBV DNA. *Lancet* 1989,**1**:406-410.
- 40. Soderstrom A, Norkrans G, Lindh M. Hepatitis B virus DNA during pregnancy and post partum: aspects on vertical transmission. *Scand J Infect Dis* 2003,**35**:814-819.


**อามา**ชีวิ 0 8 ปีเค. 2558 คณะกรรมการจริยธรรมการวิจัยในมนุษย์ สถาบันพัฒนาควรศัยยรครการวิจัยโรยสมุษย์ (สคม

41. ter Borg MJ, Leemans WF, de Man RA, Janssen HL. Exacerbation of chronic hepatitis B infection after delivery. *J Viral Hepat* 2008,**15**:37-41.

- 42. Lin HH, Chen PJ, Chen DS, Sung JL, Yang KH, Young YC, et al. Postpartum subsidence of hepatitis B viral replication in HBeAg-positive carrier mothers. *J Med Virol* 1989,29:1-6.
- 43. Coursaget P, Kane M. Overview of clinical studies in developping countries. In: *Hepatitis B vaccines in clinical practice*. Edited by Ellis RW. New York: Marcel Dekker; 1993. pp. 209-238.
- 44. Da Villa G, Pelliccia MG, Peluso F, Ricciardi E, Sepe A. Anti-HBs responses in children vaccinated with different schedules of either plasma-derived or HBV DNA recombinant vaccine. *Res Virol* 1997,148:109-114.
- 45. Goldfarb J, Baley J, Medendorp SV, Seto D, Garcia H, Toy P, et al. Comparative study of the immunogenicity and safety of two dosing schedules of Engerix-B hepatitis B vaccine in neonates. *Pediatr Infect Dis J* 1994,13:18-22.
- 46. Greenberg DP, Vadheim CM, Wong VK, Marcy SM, Partridge S, Greene T, et al. Comparative safety and immunogenicity of two recombinant hepatitis B vaccines given to infants at two, four and six months of age. *Pediatr Infect Dis J* 1996,**15**:590-596.
- 47. Poovorawan Y, Theamboonlers A, Vimolket T, Sinlaparatsamee S, Chaiear K, Siraprapasiri T, et al. Impact of hepatitis B immunisation as part of the EPI. *Vaccine* 2000, **19**:943-949.
- 48. Tharmaphornpilas P, Rasdjarmrearnsook AO, Plianpanich S, Sa-nguanmoo P, Poovorawan Y. Increased risk of developing chronic HBV infection in infants born to chronically HBV infected mothers as a result of delayed second dose of hepatitis B vaccination. *Vaccine* 2009,**27**:6110-6115.
- 49. Chang MH. Hepatitis B vaccination: disease and cancer prevention-a Taiwanese experience. *Clin Liver Dis* 2010,14:521-530.
- 50. Ng KP, Saw TL, Baki A, Rozainah K, Pang KW, Ramanathan M. Impact of the Expanded Program of Immunization against hepatitis B infection in school children in Malaysia. *Med Microbiol Immunol* 2005,194:163-168.
- 51. Chongsrisawat V, Yoocharoen P, Theamboonlers A, Tharmaphornpilas P, Warinsathien P, Sinlaparatsamee S, et al. Hepatitis B seroprevalence in Thailand: 12 years after hepatitis B vaccine integration into the national expanded programme on immunization. *Trop Med Int Health* 2006,11:1496-1502.
- 52. Lee C, Gong Y, Brok J, Boxall EH, Gluud C. Effect of hepatitis B immunisation in newborn infants of mothers positive for hepatitis B surface antigen: systematic review and meta-analysis. *BMJ* 2006,332:328-336.
- 53. Boot HJ, Hahne S, Cremer J, Wong A, Boland G, van Loon AM. Persistent and transient hepatitis B virus (HBV) infections in children born to HBV-infected mothers despite active and passive vaccination. *J Viral Hepat* 2010.
- 54. del Canho R, Grosheide PM, Schalm SW, de Vries RR, Heijtink RA. Failure of neonatal hepatitis B vaccination: the role of HBV-DNA levels in hepatitis B carrier mothers and HLA antigens in neonates. *J Hepatol* 1994,20:483-486.
- 55. Xu DZ, Yan YP, Choi BC, Xu JQ, Men K, Zhang JX, *et al.* Risk factors and mechanism of transplacental transmission of hepatitis B virus: a case-control study. *J Med Virol* 2002,**67**:20-26.
- 56. Han GR, Cao MK, Zhao W, Jiang HX, Wang CM, Bai SF, et al. A prospective and open-label study for the efficacy and safety of telbivudine in pregnancy for the prevention of perinatal transmission of hepatitis B virus infection. *J Hepatol* 2011,55:1215-1221.
- 57. Xu WM, Cui YT, Wang L, Yang H, Liang ZQ, Li XM, *et al.* Lamivudine in late pregnancy to prevent perinatal transmission of hepatitis B virus infection: a multicentre, randomized, double-blind, placebo-controlled study. *J Viral Hepat* 2009,16:94-103.



- 58. Shi Z, Yang Y, Ma L, Li X, Schreiber A. Lamivudine in late pregnancy to interrupt in utero transmission of hepatitis B virus: a systematic review and meta-analysis. *Obstet Gynecol* 2010,**116**:147-159.
- 59. Chen HL, Lin LH, Hu FC, Lee JT, Lin WT, Yang YJ, et al. Effects of maternal screening and universal immunization to prevent mother-to-infant transmission of HBV. Gastroenterology 2012,**142**:773-781 e772.
- 60. Yang J, Zeng XM, Men YL, Zhao LS. Elective caesarean section versus vaginal delivery for preventing mother to child transmission of hepatitis B virus--a systematic review. *Virol J* 2008,**5**:100.
- 61. Shi Z, Li X, Ma L, Yang Y. Hepatitis B immunoglobulin injection in pregnancy to interrupt hepatitis B virus mother-to-child transmission-a meta-analysis. *Int J Infect Dis* 2010,**14**:e622-634.
- 62. van Zonneveld M, van Nunen AB, Niesters HG, de Man RA, Schalm SW, Janssen HL. Lamivudine treatment during pregnancy to prevent perinatal transmission of hepatitis B virus infection. *J Viral Hepat* 2003,**10**:294-297.
- 63. Pan CQ, Mi LJ, Bunchorntavakul C, Karsdon J, Huang WM, Singhvi G, et al. Tenofovir Disoproxil Fumarate for Prevention of Vertical Transmission of Hepatitis B Virus Infection by Highly Viremic Pregnant Women: A Case Series. *Dig Dis Sci* 2012.
- 64. Pan CQ, Han GR, Jiang HX, Zhao W, Cao MK, Wang CM, et al. Telbivudine prevents vertical transmission from HBeAg-positive women with chronic hepatitis B. *Clin Gastroenterol Hepatol* 2012, **10**:520-526.
- 65. WHO. In: Consolidated Guidelines on the Use of Antiretroviral Drugs for Treating and Preventing HIV Infection: Recommendations for a Public Health Approach. Geneva; 2013.
- 66. Van Bommel F, Wiegand J, Berg T. Hepatitis B treatment. In: *Hepatoloy 2012 A clinical textbook*. Edited by Mauss B, Rockstroh, Sarrazin, Wedemeyer. Third ed: Flying Publisher; 2012. pp. 128-159.
- 67. Murray KF, Szenborn L, Wysocki J, Rossi S, Corsa AC, Dinh P, et al. Randomized, placebo-controlled trial of tenofovir disoproxil fumarate in adolescents with chronic hepatitis B. *Hepatology* 2012,**56**:2018-2026.
- 68. Liu AY, Vittinghoff E, Sellmeyer DE, Irvin R, Mulligan K, Mayer K, et al. Bone mineral density in HIV-negative men participating in a tenofovir pre-exposure prophylaxis randomized clinical trial in San Francisco. *PLoS One* 2011,**6**:e23688.
- 69. Tsai NC, Marcellin P, Buti M, Washington MK, Lee SS, Chan S, et al. Viral suppression and cirrhosis regression with tenofovir disoproxil fumarate in Asians with chronic hepatitis B. *Dig Dis Sci* 2015,**60**:260-268.
- 70. Honkoop P, de Man RA, Niesters HG, Zondervan PE, Schalm SW. Acute exacerbation of chronic hepatitis B virus infection after withdrawal of lamivudine therapy. *Hepatology* 2000, **32**:635-639.
- 71. Antiretroviral Pregnancy Registry. Antiretroviral Pregnancy Registry International Interim Report for 1 January 1989 31 January 2012. In; 2012.
- 72. Barret B, Tardieu M, Rustin P, Lacroix C, Chabrol B, Desguerre I, et al. Persistent mitochondrial dysfunction in HIV-1-exposed but uninfected infants: clinical screening in a large prospective cohort. AIDS 2003,17:1769-1785.
- 73. Blanche S, Tardieu M, Rustin P, Slama A, Barret B, Firtion G, et al. Persistent mitochondrial dysfunction and perinatal exposure to antiretroviral nucleoside analogues. *Lancet* 1999, **354**:1084-1089.
- 74. Brogly SB, Ylitalo N, Mofenson LM, Oleske J, Van Dyke R, Crain MJ, et al. In utero nucleoside reverse transcriptase inhibitor exposure and signs of possible mitochondrial dysfunction in HIV-uninfected children. *AIDS* 2007,**21**:929-938.


คณะกรรมการจรียธรรมการวิจัยในมนุษธ

- 75. Gibb DM, Kizito H, Russell EC, Chidziva E, Zalwango E, Nalumenya R, et al. Pregnancy and infant outcomes among HIV-infected women taking long-term ART with and without tenofovir in the DART trial. *PLoS Med* 2012,**9**:e1001217.
- 76. Siberry GK, Williams PL, Mendez H, Seage GR, 3rd, Jacobson DL, Hazra R, *et al.* Safety of tenofovir use during pregnancy: early growth outcomes in HIV-exposed uninfected infants. *AIDS* 2012,**26**:1151-1159.
- 77. Vigano A, Mora S, Giacomet V, Stucchi S, Manfredini V, Gabiano C, et al. In utero exposure to tenofovir disoproxil fumarate does not impair growth and bone health in HIV-uninfected children born to HIV-infected mothers. *Antivir Ther* 2011,**16**:1259-1266.
- 78. Binkovitz LA, Henwood MJ, Sparke P. Pediatric dual-energy X-ray absorptiometry: technique, interpretation, and clinical applications. *Semin Nucl Med* 2007,**37**:303-313.
- 79. Akcakus M, Koklu E, Kurtoglu S, Kula M, Koklu SS. The relationship among intrauterine growth, insulinlike growth factor I (IGF-I), IGF-binding protein-3, and bone mineral status in newborn infants. *Am J Perinatol* 2006,**23**:473-480.
- 80. Binkovitz LA, Henwood MJ, Sparke P. Pediatric DXA: technique, interpretation and clinical applications. *Pediatr Radiol* 2008,**38 Suppl 2**:S227-239.
- 81. Panel on Treatment of HIV-Infected Pregnant Women and Prevention of Perinatal Transmission. Recommendations for Use of Antiretroviral Drugs in Pregnant HIV-1-Infected Women for Maternal Health and Interventions to Reduce Perinatal HIV Transmission in the United States. September 14, 2011. In; 2011. pp. 1-207.
- 82. Liaw Y-F, Kao J-H, Piratvisuth T, Chan HLY, Chien R-N, Liu C-J, et al. Asian-Pacific consensus statement on the management of chronic hepatitis B: a 2012 update. *Hepatol Int* 2012:531–561.
- 83. International conference on harmonisation of technical requirements for registration of pharmaceuticals for human use. Good clinical practice: consolidated guideline: availability. *Fed regist* 1997,**62**:25691-25709.
- 84. Roingeard P, Diouf A, Sankale JL, Boye C, Mboup S, Diadhiou F, et al. Perinatal transmission of hepatitis B virus in Senegal, west Africa. *Viral Immunol* 1993,**6**:65-73.
- 85. Papaevangelou V, Paraskevis D, Anastassiadou V, Stratiki E, Machaira M, Pitsouli I, et al. HBV viremia in newborns of HBsAg(+) predominantly Caucasian HBeAg(-) mothers. *J Clin Virol* 2011,**50**:249-252.
- 86. Sirirungsi W, Urien S, Harrison L, Kamkon J, Tawon Y, Luekamlung N, et al. No relationship between drug transporter genetic variants and tenofovir plasma concentrations or changes in glomerular filtration rate in HIV-infected adults. *J Acquir Immune Defic Syndr* 2015, **68**:e56-59.
- 87. Kalkwarf HJ, Zemel BS, Yolton K, Heubi JE. Bone mineral content and density of the lumbar spine of infants and toddlers: influence of age, sex, race, growth, and human milk feeding. *J Bone Miner Res* 2013,**28**:206-212.
- 88. Glastre C, Braillon P, David L, Cochat P, Meunier PJ, Delmas PD. Measurement of bone mineral content of the lumbar spine by dual energy x-ray absorptiometry in normal children: correlations with growth parameters. *J Clin Endocrinol Metab* 1990,**70**:1330-1333.
- 89. Marcellin P, Heathcote EJ, Buti M, Gane E, de Man RA, Krastev Z, et al. Tenofovir disoproxil fumarate versus adefovir dipivoxil for chronic hepatitis B. *N Engl J Med* 2008,**359**:2442-2455.
- 90. Landreau-Mascaro A, Barret B, Mayaux MJ, Tardieu M, Blanche S. Risk of early febrile seizure with perinatal exposure to nucleoside analogues. *Lancet* 2002, **359**:583-584.
- 91. Lindegren ML, Rhodes P, Gordon L, Fleming P. Drug safety during pregnancy and in infants. Lack of mortality related to mitochondrial dysfunction among perinatally HIV-exposed children in pediatric HIV surveillance. *Ann N Y Acad Sci* 2000,**918**:222-235.



## **Appendices**

## Appendix 1: Informed Consent Form to Participate in iTAP Study (Thai Language)

แบบแสดงความยินยอมเข้าร่วมการวิจัย

ชื่อโครงการวิจัย:การวิจัยทางคลินิค ระยะที่ 3 แบบสุ่มตัวอย่าง ปกปิดทั้ง 2 ฝ่าย เปรียบเทียบกับสารไร้ฤทธิ์ เพื่อ ประเมินประสิทธิผลและความปลอดภัยของยาทีโนโฟเวียร์ ไดโซพรอกซิล ฟูมาเรต (tenofovir disoproxil fumarate) ที่ให้แก่หญิงตั้งครรภ์ตั้งแต่อายุครรภ์ 28 สัปดาห์ จนถึง 2 เดือนหลังคลอดที่ติดเชื้อไวรัสตับอักเสบบีเรื้อรัง และตรวจพบแอนติเจนเปลือกนอก (HBsAg) และแอนติเจนอี (HBeAg) ของไวรัสตับอักเสบบีเพื่อป้องกันการถ่ายทอด เชื้อไวรัสตับอักเสบบีจากมารดาสู่ทารกที่ได้รับวัคซีนและอิมมิวโนโกลบูลิน (immunoglobulin) ต่อไวรัสตับอักเสบบี

ชื่อย่อ: ยาต้านไวรัสสำหรับมารดาเพื่อป้องกันการถ่ายทอดเชื้อไวรัสตับอักเสบบีจากมารดาสู่ทารกในประเทศไทย

## <u>วัตถุประสงค์</u>

ท่าน<u>และทารกของท่าน</u>กำลังได้รับการเชิญให้เข้าร่วมการศึกษาวิจัยของยาทีโนโฟเวียร์ซึ่งอาจจะช่วยป้องกันการ ถ่ายทอดเชื้อไวรัสตับอักเสบบี (ซึ่งเรียกว่าเอช บี วี) จากหญิงตั้งครรภ์ที่ติดเชื้อไวรัสตับอักเสบบีไปสู่ทารก วัตถุประสงค์ของ การวิจัยนี้คือเพื่อแสดงให้เห็นว่า การรับประทานยาทีโนโฟเวียร์ในช่วงไตรมาสสุดท้ายของการตั้งครรภ์จนถึง 2 เดือนหลัง คลอดสามารถลดความเสี่ยงของการถ่ายทอดเชื้อไวรัสตับอักเสบบีไปสู่ทารกของท่านได้แบบแสดงความยินยอมเข้าร่วมการ วิจัยนี้ มีรายละเอียดเกี่ยวกับการวิจัย ซึ่งแพทย์ผู้ดูแลท่านจะร่วมพูดคุยให้ข้อมูลกับท่าน เพื่อท่านจะได้ทราบรายละเอียด ของการวิจัย และตัดสินใจว่าจะสมัครเข้าร่วมการวิจัยนี้หรือไม่

การเข้าร่วมในการศึกษาวิจัยนี้ของท่านจะเป็นไปโดยสมัครใจอย่างเต็มที่ ท่านมีอิสระที่จะปฏิเสธการเข้าร่วมการ วิจัยในวันนี้หรือขอถอนตัวจากการวิจัยในอนาคตได้ทุกเมื่อที่ท่านต้องการโดยไม่สูญเสียโอกาสการได้รับบริการทาง การแพทย์ที่ได้มาตรฐาน หรือโอกาสในการเข้าร่วมการศึกษาวิจัยอื่นๆ ในอนาคต

การศึกษาวิจัยนี้เป็นความร่วมมือระหว่างคณะนักวิจัยและแพทย์โดยได้รับการสนับสนุนจากกระทรวงสาธารณสุข ไทย สถาบันสุขภาพแห่งชาติสหรัฐอเมริกา (เอ็น ไอ เอช) และศูนย์ควบคุมและป้องกันโรค (ซีดีซี) แห่งสหรัฐอเมริกา

## เหตุผลและความจำเป็นที่ต้องทำการวิจัย

ประชากรที่ติดเชื้อไวรัสตับอักเสบบีเรื้อรังจะมีชิ้นส่วนเล็กๆของเชื้อไวรัส ที่เรียกว่าแอนติเจนอยู่บนเปลือกนอกของ เชื้อไวรัส (เอชบีเอสเอจี) ในเลือดซึ่งสามารถตรวจพบได้จากการตรวจเลือด ด้วยวิธีง่ายๆ ซึ่งเป็นวิธีที่ใช้อย่างแพร่หลายใน ประเทศไทย มีผู้ใหญ่จำนวนประมาณ 2-3 ล้านคนในประเทศไทยที่ติดเชื้อไวรัสตับอักเสบบี (เอช บี วี) เรื้อรัง การอักเสบที่ เกิดจากไวรัสตับอักเสบบีเป็นเวลานานสามารถทำลายเซลล์ตับและเป็นสาเหตุให้เกิดตับแข็งและโรคมะเร็ง ซึ่งโดยปกติ เกิดขึ้นในวัยผู้ใหญ่

ท่านกำลังตั้งครรภ์และติดเชื้อไวรัสตับอักเสบบี และท่านไม่ติดเชื้อเอช ไอ วี (เอช ไอ วีและเอช บี วีเป็นไวรัส 2 ชนิดที่แตกต่างกัน) ปัจจุบันทารกทุกรายที่คลอดจากมารดาที่ติดเชื้อไวรัสตับอักเสบบีต้องได้รับการฉีดวัคซีนไวรัสตับอักเสบ บีเมื่อแรกเกิด และเมื่ออายุ 1, 2, 4และ 6 เดือนเพื่อป้องกันการติดเชื้อนี้ นอกจากนี้ราชวิทยาลัยกุมารแพทย์แห่งประเทศ ไทยแนะนำว่าทารกควรได้รับอิมมิวโนโกลบูลิน (สารภูมิต้านทานต่อต้านไวรัสตับอักเสบบี) ภายในชั่วโมงแรกหลังจากคลอด



อย่างไรก็ตาม หญิงตั้งครรภ์ที่มีระดับไวรัสตับอักเสบบีสูงในเลือดมีความเสี่ยงประมาณร้อยละ 10 - 12 ในการ ถ่ายทอดเชื้อไวรัสไปสู่ทารก ทั้งๆ ที่มีการฉีดวัคชีนไวรัสตับอักเสบบีและสารภูมิต้านทานต่อต้านไวรัสตับอักเสบบีเพื่อการ ป้องกันการติดเชื้อ ผู้ใหญ่ส่วนมากที่มีระดับไวรัสตับอักเสบบีสูงในเลือดสามารถตรวจพบแอนติเจนอีกชนิดหนึ่งด้วยที่ เรียกว่าแอนติเจนอีของไวรัสตับอักเสบบี (เอชบีอีเอจี) ในประชากรที่อายุน้อยที่มีแอนติเจนเปลือกนอกของไวรัสตับอักเสบบี และมีแอนติเจนอีของไวรัสตับอักเสบบี หากว่ามีการ ตอบสนองต่อการติดเชื้อ ระดับเอนไซม์ของตับ (ที่เรียกว่าค่าเอแอลที หรือโดยปกติในประเทศไทยเรียกค่านี้ว่าค่าเอสจีพีที) ในเลือดจะมีค่าสูงกว่าปกติ ปริมาณเอสจีพีทีในเลือดสามารถวัดได้โดยใช้วิธีการตรวจเลือดอย่างง่ายๆ ซึ่งเป็นวิธีที่ใช้อย่าง แพร่หลายในประเทศไทย หากระดับค่าเอสจีพีทีปกติ หมายความว่าระบบภูมิคุ้มกันไม่มีปฏิกิริยาในการต่อต้านไวรัสตับ อักเสบบี ในการวิจัยนี้ หญิงตั้งครรภ์ที่ตรวจพบแอนติเจนอีของไวรัสตับอักเสบบีในเลือดและมีระดับค่าเอสจีพีทีปกติเท่านั้น (น้อยกว่า 30 ยูนิต/ลิตร) จึงจะได้รับการร้องขอให้เข้าร่วมการวิจัย

ยาที่โนโฟเวียร์เป็นยาต้านไวรัสตับอักเสบบีที่ได้รับการรับรองโดยสำนักงานคณะกรรมการอาหารและยาประเทศ ไทยสำหรับการรักษาไวรัสตับอักเสบบี แต่ยังไม่ทราบว่าการรับประทานยาที่โนโฟเวียร์ในช่วงไตรมาสสุดท้ายของการ ตั้งครรภ์จนถึง 2 เดือนหลังคลอดจะช่วยลดความเสี่ยงของการถ่ายทอดเชื้อไวรัสตับอักเสบบีไปสู่ทารกได้หรือไม่

หญิงตั้งครรภ์มากกว่า 1370 รายได้รับประทานยาทีโนโฟเวียร์และไม่มีหลักฐานที่แสดงว่ายาทีโนโฟเวียร์ก่อให้เกิด อันตรายแก่ทารกในครรภ์ ยาทีโนโฟเวียร์ไปรบกวนต่อกระบวนการเปลี่ยนแปลง (เมตาบอลิซึม) ของกระดูก อย่างไรก็ตาม ในกลุ่มทารกที่มารดาได้รับยาทีโนโฟเวียร์เป็นองค์ประกอบในสูตรยาในระหว่างตั้งครรภ์ไม่ได้มีผลต่อน้ำหนักแรกคลอดของ ทารกที่ได้สัมผัสยาทีโนโฟเวียร์ หรือมีผลต่อการเจริญเติบโตของทารก

ในการวิจัยนี้ หญิงตั้งครรภ์ที่ติดเชื้อไวรัสตับอักเสบบีจำนวน 328 ราย และมีอายุอย่างน้อย 18 ปีจะได้เข้าร่วมการ วิจัย ตลอดระยะเวลา 2 ปีในโรงพยาบาลรัฐ 19 แห่งทั่วประเทศไทย ทั้งในโรงพยาบาลประจำจังหวัดลและภูมิภาค ได้แก่ โรงพยาบาลพะเยา โรงพยาบาลเชียงรายประชานุเคราะห์ โรงพยาบาลพระปกเกล้าจังหวัดจันทบุรี โรงพยาบาลชลบุรี โรงพยาบาลภูมิพลอดุลยเดช กรมแพทย์ทหารอากาศ กรุงเทพฯ ศูนย์อนามัยที่ 10 โรงพยาบาลส่งเสริมสุขภาพ จังหวัด เชียงใหม่ โรงพยาบาลลำพูน โรงพยาบาลเชียงคำ จังหวัดพะเยา โรงพยาบาลแม่จัน จังหวัดเชียงราย โรงพยาบาลบางละมุง จังหวัดชลบุรี โรงพยาบาลนครพิงค์ จังหวัดเชียงใหม่ โรงพยาบาลนพรัตนราชธานีกรุงเทพฯ โรงพยาบาลขอนแก่น โรงพยาบาลสมุทรสาคร โรงพยาบาลนคปฐม โรงพยาบาลสมุทรปราการ โรงพยาบาลลำปาง โรงพยาบาลมหาราช นครราชสีมา และ โรงพยาบาลระนอง

มารดาแต่ละรายจะถูกจัดเข้ากลุ่มโดยการสุ่มให้เข้าร่วมใน 1 กลุ่มการวิจัยจากจำนวน 2 กลุ่มการวิจัยในจำนวน เท่ากันได้แก่:

- กลุ่มที่ 1 (ยาทีโนโฟเวียร์):อาสาสมัครหญิงจะได้รับประทานยาทีโนโฟเวียร์จำนวน 1 เม็ด ขนาด 300 มก. วันละครั้ง ตั้งแต่อายุครรภ์ 28 สัปดาห์ จนถึง 2 เดือนหลังคลอด
- กลุ่มที่ 2 (สารไร้ฤทธิ์):อาสาสมัครหญิงจะได้รับประทานสารไร้ฤทธิ์จำนวน 1 เม็ด วันละครั้งตั้งแต่อายุครรภ์ 28 สัปดาห์ จนถึง 2 เดือนหลังคลอด

ทารกทุกรายจะได้รับอิมมิวโนโกลบูลินและวัคซีนตับอักเสบบีตามที่ราชวิทยาลัยกุมารแพทย์แห่งประเทศไทยได้ แนะนำให้ฉีดสำหรับทารกที่คลอดจากมารดาติดเชื้อไวรัสตับอักเสบบี ท่านและแพทย์ผู้ดูแลท่านจะไม่สามารถเลือกหรือ ทราบได้ว่าท่านจะอยู่ในกลุ่มการวิจัยกลุ่มไหน

> **อาเมโต** 0 8 ปีค. 2558 คณะกรรมการจริยธรรมดารวิจัยในมนุษย


สถาบันพัฒนาการคุ้มกรองการวิจัยในบนุษย์ (สคม

## วิธีการดำเนินการวิจัยสำหรับท่าน

ก่อนอื่นทางโครงการจะเสนอให้มีการเจาะเลือดท่าน (5 ซีซีหรือน้อยกว่าครึ่งช้อนโต๊ะ) สำหรับการตรวจเพื่อให้ ทราบว่าท่านมีแอนติเจนอีของไวรัสตับอักเสบบี (เอชบีอีเอจี) ในเลือดของท่านหรือไม่และเพื่อวัดระดับของค่าเอสจีพีที ต้อง ดำเนินการตรวจสิ่งเหล่านี้ในระหว่างตั้งครรภ์ เพื่อให้ทราบผลโดยเร็วก่อนอายุครรภ์ 28 สัปดาห์

ทางโครงการจะขออนุญาตท่านให้ทางโครงการได้ทำการบันทึกผลการตรวจทางห้องปฏิบัติการต่างๆ ซึ่งเป็นส่วน หนึ่งของการตรวจประเมินเพื่อการดูแลรักษาทางคลินิกตามปกติของท่าน ก่อนที่ท่านจะลงชื่อแสดงความยินยอมเข้าร่วม โครงการวิจัยนี้

เฉพาะหญิงที่มีค่าแอนติเจนอีของไวรัสตับอักเสบบีอาจจะมีปริมาณไวรัสในร่างกายสูงและมีความเสี่ยงของการ ถ่ายทอดเชื้อไวรัสตับอักเสบบีสูงจะได้รับการร้องขอให้เข้าร่วมในการวิจัยต่อไป อย่างไรก็ตามหากระดับเอสจีพีทีสูงเกินไป (มากกว่า 30 ยูนิต/ลิตร) ท่านจะไม่ได้รับการร้องขอให้เข้าร่วมในการวิจัยต่อไปและทางโครงการจะแนะนำให้พบแพทย์ ผู้เชี่ยวชาญด้านไวรัสตับอักเสบบีเพื่อแนะนำท่านในการตรวจเพิ่มเติมหรือรับการรักษาหากจำเป็น

หากท่านตรวจพบแอนติเจนอีของไวรัสตับอักเสบบี (เอชบีอีเอจี) และระดับของค่าเอสจีพีที่เท่ากับหรือน้อยกว่า 30 ยูนิต/ลิตร ท่านจะได้รับการเสนอให้เข้าร่วมในการวิจัยต่อไป เมื่ออายุครรภ์ 26 สัปดาห์ จะพิจารณาประวัติทางการแพทย์ ของท่านและท่านจะได้รับการตรวจร่างกายและเจาะเลือดเพื่อการตรวจเพิ่มเติม (ประมาณ 16 ซีซีหรือประมาณหนึ่งช้อน โต๊ะ) เพื่อดูว่าท่านมีคุณสมบัติให้เข้าร่วมในการวิจัยต่อไป ท่านจะถูกจัดเข้ากลุ่มโดยการสุ่มให้เข้าร่วมใน 1 กลุ่มการวิจัยจากจำนวน 2 กลุ่มเมื่ออายุครรภ์ 28 สัปดาห์ และท่านจะได้รับยาที่ใช้ในการวิจัยจำนวน 1 ขวด ท่านต้องรับประทานยาจำนวน 1 เม็ดวันละครั้ง โดยรับประทานยาในเวลาเดียวกัน ทุกวันจนถึง 2 เดือนหลังคลอด ท่านจะไม่ทราบว่าท่านกำลังรับประทานยาเม็ดที่โนโฟเวียร์หรือสารไร้ฤทธิ์ หลังจากการเข้า ร่วมโครงการ ท่านจะได้รับการตรวจสุขภาพทางการแพทย์เป็นประจำที่คลินิคฝากครรภ์เช่นเดียวกับหญิงตั้งครรภ์รายอื่น และทางโครงการจะประเมินสุขภาพของท่านเพื่อดูผลข้างเคียงต่างๆของการรักษาที่เกิดขึ้น ด้วยการเจาะเลือด (33-38 ซีซี หรือประมาณสองข้อนโต๊ะครึ่ง) ในแต่ละนัดหมายที่แตกต่างกันจะมีการเจาะเลือดเพิ่มเติม (30ซีซี หรือประมาณ 2 ซ้อนโต๊ะ) สำหรับเก็บ peripheral blood mononuclear cells (PBMC) ซึ่ง PBMC จะถูกเก็บไว้สำหรับการศึกษาวิจัยเพิ่มเติมที่ เกี่ยวข้องกับการตอบสนองของภูมิค้มกันต่อเชื้อไวรัสตับอักเสบบีก่อนที่จะเกิดการมีตับอักเสบรนแรง

เมื่อท่านเจ็บครรภ์คลอด ท่านจะต้องไปที่แผนกคลอดทันที เมื่อท่านมาถึงแผนกคลอด จะมีการเจาะเลือดท่านเพื่อ การตรวจต่างๆ (ประมาณ 10 ซีซีหรือประมาณหนึ่งข้อนโต๊ะ) การตรวจต่างๆ ได้แก่ การตรวจนับเม็ดเลือดอย่างสมบูรณ์ (ซี บีซี) เอสจีพีที ระดับครีเอตินิน (เพื่อวัดการทำงานของไต) ซีรัมฟอสฟอรัส (เพื่อวัดการเปลี่ยนแปลงของเนื้อเยื่อกระดูก) ปริมาณไวรัสตับอักเสบบีในกระแสเลือด และระดับยาทีโนโฟเวียร์เพื่อติดตามผลของการรักษา

หลังคลอดท่านจะถูกขอให้มาตามนัดหมายการวิจัยที่ 1, 2, 3, 4, 6 และ 12 เดือนเพื่อติดตามผลของการรักษา ท่านจะได้รับการตรวจร่างกายและเจาะเลือด (38-43 ซีซี หรือประมาณสามข้อนโต๊ะ) เพื่อติดตามการเปลี่ยนแปลงของค่า เอสจีพีที ซีรัมฟอสฟอรัสและ ครีเอตินิน ปริมาณไวรัสตับอักเสบบีในกระแสเลือด แอนติเจนอีของไวรัสตับอักเสบบีและการ ตรวจนับเม็ดเลือดอย่างสมบูรณ์

ในระหว่างหรือช่วงหลังการรักษา ท่านควรจะติดต่อแพทย์ผู้ดูแลของท่านหรือพยาบาลผู้รับผิดชอบในการวิจัยทันที (ดูหมายเลขโทรศัพท์ในส่วนท้ายของแบบแสดงความยินยอมนี้) หากท่านมีอาการเจ็บปวดจากสภาวะต่างๆ โดยเฉพาะหาก ท่านมีอาการแสดงหรืออาการซึ่งเกิดจากปัญหาของตับดังต่อไปนี้:

- ผิวหนังของท่านหรือส่วนตาขาวของท่านได้เปลี่ยนเป็นสีเหลือง (ดีซ่าน)
- ปัสสาวะของท่านมีสีเข้ม




คณะกรรมการจริยธรรมการวิจัยในมนุษช

- อุจจาระสีจางลง
- ท่านไม่รู้สึกอยากรับประทานอาหารเป็นเวลาหลายวันหรือเป็นเวลานานกว่านั้น
- ท่านรู้สึกไม่สบายท้อง (มีอาการคลื่นไส้)
- ท่านปวดบริเวณท้องน้อย

หากระดับของค่าเอสจีพีทีเพิ่มขึ้นเป็น 60 ยูนิต/ลิตร หรือมากกว่านั้น ท่านจะได้รับการติดต่อและถูกขอให้กลับมายัง โรงพยาบาลโดยเร็วที่สุดภายใน 3 วัน เพื่อการเจาะเลือดอีกครั้งหนึ่งเพื่อยืนยันระดับค่าเอสจีพีทีที่สูงนี้ หากท่านสังเกตพบ อาการแสดงหรืออาการตามรายการที่ได้กล่าวมาด้านบน ท่านควรจะกลับไปที่โรงพยาบาลโดยทันที หากการเจาะเลือดครั้ง ที่สองยังยืนยันว่ามีค่าเพิ่มขึ้น ท่านจะถูกขอให้กลับมาตรวจเลือดใหม่อีกครั้งในเวลาสองสัปดาห์ต่อมา หากเมื่อใดก็ตามที่ ระดับค่าเอสจีพีทีของท่านเกิน 150 ยูนิต/ลิตร แพทย์ผู้ดูแลท่านจะพิจารณาให้เริ่มยาที่ใช้ในการวิจัยอีกครั้ง ท่านจะได้รับการติดตามในโครงการวิจัยจนถึง 1 ปีหลังคลอด หลังจากสิ้นสุดการเข้าร่วมการวิจัยของท่าน การรักษาที่ท่านได้รับจะถูก ปรับเปลี่ยนเป็นยาที่โนโฟเวียร์ที่มีจัดจำหน่ายหากว่าท่านได้เริ่มการรักษา หรือท่านจะได้รับการบอกกล่าวหากท่านได้รับ สารไร้ฤทธิ์ และได้รับการติดตามโดยอายุรแพทย์ตามแนวทางปฏิบัติปัจจุบัน โดยที่ยังไม่ทราบว่าท่านจะได้รับการรักษานี้ ต่อเนื่องไปนานเท่าไร

## วิธีการดำเนินการวิจัยสำหรับทารกของท่าน

ทารกของท่านจะได้รับอิมมิวโนโกลบูลินของไวรัสตับอักเสบบีภายใน 12 ชั่วโมงหลังคลอด และได้รับวัคซีนไวรัสตับ อักเสบบีภายใน 12 ชั่วโมงหลังคลอดและเมื่อทารกอายุ 1, 2, 4 และ 6 เดือน โครงการจะขอให้ท่านนำทารกไปโรงพยาบาล ในนัดหมายสำหรับทารกหลังคลอดที่ 1, 2, 4, 6, 9 และ 12 เดือนเพื่อประเมินความปลอดภัยทางคลินิคและการพิจารณา สรุปผลสถานะการติดเชื้อไวรัสตับอักเสบบี

จะมีการเก็บตัวอย่างเลือดจากทารกของท่าน (2-4 ซีซี หรือไม่เกิน 1 ช้อนชา) ในแต่ละนัดหมายเพื่อตรวจ ผลข้างเคียงของการรักษาและเพื่อค้นหาหลักฐานของการติดเชื้อไวรัสตับอักเสบบี

การเลี้ยงลูกด้วยนมมารดา ท่านสามารถเลี้ยงทารกของท่านด้วยนมมารดาเนื่องจากความเสี่ยงในการถ่ายทอดเชื้อไวรัสตับ อักเสบบีไปสู่ทารกของท่านไม่ได้เพิ่มขึ้นเนื่องด้วยการเลี้ยงลูกด้วยนมมารดา

วิธีป้องกันสุขภาพของท่าน ท่านและทารกของท่านจะได้รับการตรวจร่างกายโดยละเอียดตลอดการวิจัย สิ่งสำคัญก็คือท่าน จะต้องมาตามนัดหมายทุกครั้งรับประทานยาตามคำสั่งของแพทย์ ในแต่ละนัดหมายทางโครงการจะสอบถามท่านว่าท่าน และทารกของท่านมีปัญหาสุขภาพใดๆหรือไม่ กำลังรับประทานยาชนิดอื่น หรือมีเหตุการณ์ไม่พึงประสงค์ใดๆ หากจำเป็น ท่านสามารถติดต่อหรือไปคลินิคได้ทุกเมื่อ แม้จะไม่ใช่เวลาตามตารางนัดหมายก็ตาม

ค่าใช้จ่ายในการเข้าร่วมโครงการ ไม่มีค่าใช้จ่ายสำหรับท่านหรือทารกของท่านไม่ว่าจะเป็นค่ายา นัดหมายพิเศษทางคลินิค หรือการตรวจทางห้องปฏิบัติการที่เกี่ยวข้องกับโครงการวิจัยนี้ ผู้เข้าร่วมโครงการวิจัยทุกรายจะได้รับเงิน 300 บาท(ใน สถานที่วิจัยทุกแห่ง ยกเว้นสถานที่วิจัยในกรุงเทพฯ ที่จะได้รับค่าใช้จ่ายจำนวน 400 บาท) ในนัดหมายการวิจัยแต่ละครั้ง สำหรับค่าชดเชยในการเดินทาง(คณะผู้วิจัยที่สถานที่วิจัยจะจ่ายค่าชดเชยในการเดินทางให้เพิ่มขึ้นได้ ในกรณีที่มีเหตุผล) ทางโครงการจะจ่ายค่าอิมมิวโนโกลบูลิน (เอชบีไอจี) สำหรับทารกของผู้เข้าร่วมโครงการวิจัยทุกราย


0 9 3 10 1 0 8 ปีค. 2558 คณะกรรมการจริยธรรมดารวิจัยในมห การค้นพบข้อมูลและข่าวสารใหม่ๆ ที่เกี่ยวข้อง ทางโครงการจะแจ้งให้ท่านทราบเกี่ยวกับการค้นพบข้อมูลต่างๆ ที่เกิดขึ้น ใหม่ในระหว่างการวิจัยโดยเร็วที่สุดซึ่งอาจมีผลต่อท่าน และทารกของท่าน หรือความสมัครใจในการเข้าร่วมโครงการวิจัย ต่อไปของท่าน

การถอนตัวออกจากการวิจัย แพทย์ผู้ดูแลของท่านอาจแนะนำให้ท่านออกจากการวิจัยหากเกิดสภาวะหรือเหตุการณ์อันไม่ พึงประสงค์รุนแรงใดๆ และการเข้าร่วมการวิจัยต่อไปอาจก่อให้เกิดอันตรายต่อตัวท่านหรือทารกของท่าน ในกรณีนี้ท่านจะ ได้รับการดูแลรักษาตามมาตรฐานที่มีอยู่ อย่างไรก็ตามท่านไม่ควรจะหยุดการรักษาของท่านโดยปราศจากคำแนะนำทาง การแพทย์เพื่อหลีกเลี่ยงการเพิ่มขึ้นของเชื้อไวรัสตับอักเสบบีในตับของท่านอย่างรวดเร็วโดยไม่ได้รับการดูแลทางการแพทย์

ทางเลือกในการเข้าร่วมโครงการวิจัย ท่านมีอิสระอย่างเต็มที่ในการเลือกที่จะไม่เข้าร่วมหรือถอนตัวท่านหรือ/และทารก ของท่านออกจากโครงการวิจัยเมื่อใดก็ได้ ทางเลือกในการเข้าร่วมโครงการวิจัยนี้เป็นการดูแลรักษาตามปกติที่มีอยู่ให้แก่ หญิงตั้งครรภ์ที่ติดเชื้อไวรัสตับอักเสบบี ณ.โรงพยาบาลของท่าน

<u>การปกปิดความลับ</u>การเข้าร่วมโครงการวิจัยนี้ของท่านและทารกของท่านจะถูกปกปิดเป็นความลับและจะไม่แจ้งให้ใคร ทราบโดยไม่ได้รับความยินยอมซึ่งเป็นลายลักษณ์อักษรจากท่าน

การปกปิดความลับของข้อมูล ทางโครงการจะใช้ความพยายามเพื่อเก็บข้อมูลส่วนตัวของท่านและทารกของท่านไว้เป็น ความลับ ข้อมูลทางการแพทย์ของท่านจะถูกเก็บรักษาไว้เป็นความลับ และจะเปิดเผยข้อมูลให้ท่านทราบตลอดจนผู้ให้การ ดูแลรักษาท่านโดยตรงเพื่อการติดตามการวิจัยหรือเพื่อวัตถุประสงค์ในการตรวจสอบการวิจัย สมาชิกของคณะผู้วิจัย สำนักงานคณะกรรมการอาหารและยาประเทศไทย (เอฟดีเอ) คณะกรรมการจริยธรรมการวิจัยในมนุษย์ สถาบันพัฒนาการ คุ้มครองการวิจัยในมนุษย์คณะกรรมการพิจารณาด้านจริยธรรมการวิจัยในโรงพยาบาลของท่าน เจ้าหน้าที่วิจัย ผู้ติดตาม การวิจัย บริษัทยาที่สนับสนุนยาในการวิจัยนี้ (บริษัทกิลเลียด) และผู้ให้การสนับสนุนการวิจัย แบบบันทึกข้อมูลทั้งหมดของ โครงการวิจัยจะใช้หมายเลขรหัส และไม่มีการระบุชื่อของท่านในแบบบันทึกข้อมูลเหล่านี้ทางโครงการจะบันทึกเฉพาะรหัส ไว้ในฐานข้อมูลการวิจัยเพื่อใช้ในการวิเคราะห์เท่านั้น จะไม่ใช้ชื่อของทารกท่านหรือระบุตัวทารกของท่านเป็นการส่วนตัวใน การตีพิมพ์เอกสารใดๆ ของการวิจัยนี้ อย่างไรก็ตามทางโครงการไม่สามารถรับรองการรักษาความลับไว้ได้อย่างสิ้นเชิง และ ข้อมูลส่วนตัวของท่านอาจจะถูกเปิดเผยหากจำเป็นโดยข้อบังคับทางกฎหมาย

การจัดเก็บตัวอย่างเลือด ตัวอย่างเลือดที่นำมาเป็นส่วนหนึ่งของการวิจัยจะระบุโดยใช้หมายเลขรหัสและจะถูกเก็บรักษา เพื่อการตรวจยืนยันผลในกรณีที่จำเป็น โดยจะเก็บเป็นเวลา 10 ปีหลังจากสิ้นสุดการวิจัย ตัวอย่างเลือดจะเก็บรักษาใน ห้องปฏิบัติการของโครงการไอ อาร์ ดี-พี เอช พี ที ภายใต้คณะเทคนิคการแพทย์ มหาวิทยาลัยเชียงใหม่ ซึ่งจะมีเพียงผู้วิจัย และเจ้าหน้าที่ห้องปฏิบัติการที่ได้รับอนุญาตเท่านั้นที่สามารถเข้าถึงตัวอย่างเลือดนี้ได้ เจ้าหน้าที่ซึ่งทำงานที่โครงการจะ เข้าถึงตัวอย่างเลือดของท่านและทารกของท่านได้ด้วยเพื่อการติดตามตัวอย่างเลือด แต่เจ้าหน้าที่เหล่านี้จะไม่สามารถระบุ ได้ว่าเป็นตัวอย่างเลือดของทารกของท่านโดยตรง ตัวอย่างเลือดจะไม่ถูกขายหรือใช้โดยตรงเพื่อผลิตภัณฑ์ทางการค้า ท่าน สามารถร้องขอให้ถอนตัวอย่างเลือดของท่านและทารกออกจากศูนย์เก็บตัวอย่างเลือดเมื่อใดก็ได้และตัวอย่างเลือดจะถูก

0 4 3 โก. 2558 กละกรรมการจริยธรรมดารวิจัยในมนุษย์ ทำลายทันทีโดยเครื่องอบความร้อนสูงด้วยไอน้ำตามกระบวนการมาตรฐานของคณะเทคนิคการแพทย์ มหาวิทยาลัยเชียงใหม่ ตัวอย่างเลือดที่เหลืออาจจะถูกเก็บไว้เพื่อการตรวจยืนยันอื่นๆ หรือเพื่อการประเมินอื่นซึ่งอาจช่วยให้ เข้าใจกลไกของการถ่ายทอดเชื้อไวรัสตับอักเสบบีจากมารดาสู่ทารกและการทำลายตับ พร้อมทั้งการตรวจดูการสร้าง พันธุกรรมของแต่ละบุคคล (ดีเอ็นเอและอาร์เอ็นเอของท่าน) ว่าช่วยในการป้องกันหรือว่าทำให้มีความเสี่ยงในการถ่ายทอด เชื้อไวรัสตับอักเสบบีมากขึ้น การเพิ่มของปริมาณไวรัสหรือผลข้างเคียงของยา (พันธุศาสตร์ของบุคคลและเภสัชพันธุศาสตร์) ท่านอาจจะอนุญาตหรือปฏิเสธให้ใช้การตรวจดีเอ็นเอและอาร์เอ็นเอทั้งหมดโดยทำเครื่องหมายในช่องว่างด้านหน้าข้อความ ในแบบแสดงความยินยอมว่าท่านได้เลือกให้เก็บหรือไม่ให้เก็บตัวอย่างเลือดหากเห็นสมควรว่ามีความจำเป็นต้องมีการวิจัย อื่น ทางโครงการจะขอให้ท่านแสดงความยินยอมเพิ่มเติม และจะยื่นขออนุมัติโครงการวิจัยนี้กับคณะกรรมการจริยธรรม การวิจัยเนื่องจากเป็นการวิจัยจำเพาะ

<u>นโยบายเกี่ยวกับการได้รับอันตรายจากการวิจัย</u>ท่านจะได้รับการดูแลรักษาที่เหมาะสมที่มีทันทีหากท่านหรือทารกมี ปัญหาทางการแพทย์ที่เกี่ยวข้องกับการเข้าร่วมในโครงการวิจัยนี้โดยไม่ต้องเสียค่าใช้จ่าย อย่างไรก็ตามโครงการวิจัยจะไม่ รับผิดชอบสำหรับการรักษาที่ไม่เกี่ยวข้องกับการวิจัย และจะไม่มีการจ่ายค่าชดเชยแต่อย่างใด

## ความเสี่ยงของท่าน/ทารกของท่าน

แม้ว่าท่านถูกจัดให้รับประทานสารไร้ฤทธิ์ (แต่ท่านจะไม่ทราบว่าท่านรับประทานยาทีโนโฟเวียร์หรือสารไร้ฤทธิ์ใน ระหว่างการวิจัย) ก็จะไม่มีความแตกต่างในด้านมาตรฐานการดูแลประชากรบางรายที่ได้รับประทานยาประเภทเดียวกันกับ ยาทีโนโฟเวียร์ทำให้เกิดปัญหาด้านตับรุนแรงขึ้นเรียกว่า เกิดความเป็นพิษต่อตับ และตับโตขึ้น (ตับโต) และมีไขมันเกาะใน ตับ (ไขมันเกาะตับ)

หากท่านถูกจัดให้รับประทานยาทีโนโฟเวียร์ ผลข้างเคียงของยาอาจรวมถึง: ไตถูกทำลายหรือไตวาย กระดูกบางลง เกิดก๊าช เวียนศีรษะ รู้สึกเหนื่อย ฟอสเฟตในเลือดต่ำ และปฏิกิริยาภูมิแพ้ซึ่งอาจจะรวมถึงมีไข้ เกิดผื่น ท้องไส้ปั่นป่วน การ อาเจียน ถ่ายเหลวหรือถ่ายเป็นน้ำ ปวดท้อง เจ็บปวด หายใจขัด หรือมีความรู้สึกเจ็บป่วยทั่วไป

ความเสี่ยงที่สำคัญที่เป็นไปได้อย่างหนึ่งของการรับประทานยาทีโนโฟเวียร์คือการกระตุ้นให้เกิดตับอักเสบ (การ อักเสบหรือการระคายเคืองของตับ) ท่านควรจะทราบว่าจะมีการตรวจการทำงานของตับของท่านบ่อยขึ้น และอาการที่ เชื่อมโยงกับไวรัสตับอักเสบบีอาจจะทำให้ทรุดลงในบางช่วงในระหว่างการรักษาด้วยยาที่ใช้ในการวิจัยหรือหลังจากที่ท่าน หยุดรับประทานยาทีโนโฟเวียร์เป็นเวลาหลายสัปดาห์หรือหลายเดือนแล้ว ซึ่งก็คือเหตุผลว่าทำไมทางโครงการจะขอให้ท่าน มาตามนัดหมายการวิจัยทุกครั้งอย่างสม่ำเสมอและแจ้งให้แพทย์ผู้ดูแลท่านทราบหากท่านไม่สามารถมาตามนัดหมายได้เพื่อ ทำการจัดตารางนัดหมายอีกครั้ง

ความเสี่ยงที่สำคัญที่อาจเกิดขึ้นได้ที่เกี่ยวข้องกับการรับประทานยาทีโนโฟเวียร์ในช่วงตั้งครรภ์คือทารกแรกเกิดมี กระดูกบางลงและการเจริญเติบโตของทารกช้าลงเล็กน้อย

ความเสี่ยงและอาการไม่สบายจากการเจาะเลือดได้แก่ ความรู้สึกเจ็บ อาการบวม การฟกซ้ำ การอักเสบของเส้น เลือดดำ และเป็นลม หากจำเป็นท่านและทารกของท่านจะได้รับการดูแลรักษาที่เหมาะสมจากแพทย์ผู้ดูแลท่าน

<u>ผลประโยชน์ของท่าน/ทารกของท่าน</u> ระหว่างการวิจัย ท่านและทารกของท่านจะได้รับการติดตามทางการแพทย์อย่าง ใกล้ชิดเพื่อความปลอดภัย


0 8 ฟี.ค. 2558 คณะกรรมการจริยธรรมการวิจัยในมนุษย

สถาบันพัฒนาการกุ้นครองการวิจัยใน**บนุษย์ (สก**ม.

หากท่านถูกจัดให้อยู่ในกลุ่มที่รับประทานยาทีโนโฟเวียร์ ท่านอาจลดความเสี่ยงในการถ่ายทอดเชื้อไวรัสตับอักเสบ บีไปสู่ทารกของท่าน หากท่านถูกจัดให้รับประทานสารไร้ฤทธิ์ทารกของท่านอาจไม่ได้รับผลประโยชน์โดยตรงแต่ท่านและ ทารกของท่านจะได้รับประโยชน์จากการติดตามและได้รับการดูแลอย่างใกล้ชิดในโครงการวิจัย

<u>ปัญหาหรือข้อซักถามเพิ่มเติม</u> เมื่อใดก็ตามหากท่านมีคำถามเพิ่มเติมเกี่ยวกับการวิจัยนี้ หรือเกี่ยวกับสิทธิและผลประโยชน์ ของท่านในฐานะอาสาสมัครท่านสามารถติดต่อ:

| คณะกรรมการจริยธรรมการวิจัยในสถาบันพัฒนาการคุ้มครองการวิจัยในมนุษย์ |
|---|
| อาคาร 8 ชั้น 7 ห้อง 702 กรมวิทยาศาสตร์การแพทย์ |
| กระทรวงสาธารณสุข 11000 โทรศัพท์: 02-5913541, 02-5913517 โทรสาร: 02-5914125<br>หรือ |
| คณะกรรมการพิจารณาด้านจริยธรรมประจำโรงพยาบาลของท่าน |
| โทรศัพท์ |
| ตัวแทนคณะกรรมการพิจารณาด้านจริยธรรมประจำโรงพยาบาลของท่าน) |

สำหรับคำถามเกี่ยวกับโครงการวิจัย สิทธิของท่าน และอันตรายที่เกิดจากการวิจัย ท่านสามารถติดต่อแพทย์ผู้ซึ่งเป็นอิสระ จากโครงการวิจัยนี้:

ชื่อ นายแพทย์ สรกิจ ภาคีชีพ ที่อยู่ สำนักงานหลักประกันสุขภาพแห่งชาติ ศูนย์ราชการเฉลิมพระเกียรติ 80 พรรษ 5 ธันวาคม 2550 อาคาร บี 120 หมู่ 3 ถนน แจ้งวัฒนะ เขตหลักสี่ กรุงเทพฯ 10210 เบอร์โทรศัพท์: +66 2141 4000 โทรสาร: +66 2143 9730-1

แพทย์ผู้วิจัยที่ดูแลด้านความปลอดภัยและสิทธิของท่านและทารกของท่าน

| นพ./พญ | | (ชื่อผู้วิจัยหลักในสถานที่วิจัยแต่ละแห่ง) |
|---|---|---|
| ที่อยู่ | | |
| โทรศัพท์ที่ทำงาน: | โทรศัพท์ที่บ้าน: | โทรศัพท์มือถือ: |
| โทรสาร: | | |
| หรือ | | (ชื่อและตำแหน่งผู้อำนวยการโรงพยาบาล) |

## <u>การแสดงความยินยอมเข้าร่วมโครงการ</u>

เมื่อท่านเซ็นชื่อในแบบแสดงความยินยอมเข้าร่วมโครงการวิจัยนี้ ท่านยอมรับว่าได้มีการอธิบายวัตถุประสงค์ของการ ศึกษาวิจัย ขั้นตอนปฏิบัติตามแผนการวิจัย ความเสี่ยง และผลประโยชน์ต่างๆ ของการเข้าร่วมโครงการวิจัยนี้ให้ท่านฟังโดย ละเอียดแล้ว ท่านทราบว่า ท่านสามารถถอนตัวท่าน หรือทารกของท่านออกจากการเข้าร่วมการวิจัยได้ตลอดเวลา โดยไม่มี ผลกระทบใดๆ ต่อสิทธิของท่าน หฺรือทารกของท่านในการได้รับการรักษาทางการแพทย์ด้วยวิธีการอื่นๆ ที่ดีที่สุดเท่าที่มีอยู่

> **0 1 1 0** 0 8 **W**.A. 2558


คณะกรรมการจริยธรรมการวิจัยในมนุษย์

การปฏิเสธเข้าร่วมโครงการ หรือการถอนตัวออกจากการเข้าร่วมโครงการวิจัยจะไม่มีความผิดใดๆ และจะไม่ทำให้ท่าน สูญเสียผลประโยชน์อื่นๆ ที่ท่านควรได้รับตามสิทธิ์ที่ท่านพึงมี ข้าพเจ้ายินยอมเข้าร่วมโครงการวิจัยและยินยอมให้บุตรของข้าพเจ้าเข้าร่วมในโครงการวิจัยนี้ ข้าพเจ้ายินยอมให้บันทึกผลการตรวจทางห้องปฏิบัติการต่างๆ ของข้าพเจ้าที่เป็นการตรวจเพื่อการดูแลรักษาทางคลินิก ก่อนที่ข้าพเจ้าจะแสดงความยินยอมเข้าร่วมโครงการวิจัยนี้ลงในเอกสารของโครงการวิจัย ใช่ 🗆 ไข่ใช่ 🗆 ชื่อผู้เข้าร่วมโครงการวิจัย วันที่ ลายเซ็น (พิมพ์หรือเขียนตัวบรรจง) ชื่อตัวแทนผู้เข้าร่วมโครงการวิจัย วันที่ ลายเซ็น ที่ถูกต้องตามกฎหมาย/ผู้ปกครอง (ถ้ามี) "ข้าพเจ้ายินยอมให้บุตรของข้าพเจ้าเข้าร่วมในโครงการวิจัยนี้" ชื่อบิดาของเด็ก วันที่ ลายเซ็น (ถ้ามี และมารดาเด็กยินยอม พิมพ์หรือเขียนตัวบรรจง) ชื่อพยาน วันที่ ลายเซ็น (พิมพ์หรือเขียนตัวบรรจง) ชื่อพยาน วันที่ ลายเซ็น (พิมพ์หรือเขียนตัวบรรจง) ข้าพเจ้าได้อธิบายถึงวัตถุประสงค์ของโครงการวิจัยนี้ให้แก่อาสาสมัครรับทราบแล้ว ด้วยความรู้ที่ดีที่สุดของข้าพเจ้า และ อาสาสมัครเข้าใจถึงวัตถุประสงค์ ขั้นตอนปฏิบัติ ความเสี่ยง และประโยชน์ต่างๆ ต่อตนเองและทารกแล้ว วันที่ แพทย์ผู้วิจัย/ผู้ให้การปรึกษา ลายเซ็น (พิมพ์หรือเขียนตัวบรรจง)


**อาโมโก** 0 8 ปีเค. 2558 คณะกรรมการจริยธรรมการวิจัยในมนุษย์ สถาบันพัฒนาการคุ้มกรวมเการวิจัยในมนุษย์ (สคม

| | เร้กษาตัวอย่างเลือดและใช้เลือ | ทำเครื่องหมายในช่อง €ที่ข้าพเจ้าตั<br>ดที่เก็บรักษาไว้สำหรับการตรวจอื่เ | |
|---|---|---|---|
| | บรักษาตัวอย่างเลือดและใช้เลือ<br>กวามยินยอมนี้ <b>ยกเว้นการตรวจดี</b> | ดที่เก็บรักษาไว้สำหรับการตรวจอื่เ<br>เ <b>อ็นเอ</b> | มๆในอนาคตตามที่ได้ |
| <b>€</b> ข้าพเจ้าไม่อนุญาตให้เก็ | บรักษาเลือดของข้าพเจ้าสำหรับเ | าารตรวจอื่นๆในอนาคต | |
| ชื่อผู้เข้าร่วมโครงการ<br>(พิมพ์หรือเขียนตัวบรรจง) | ลายเช็น | วันที่ | |
| ชื่อพยาน<br>(พิมพ์หรือเขียนตัวบรรจง) | ลายเซ็น | <br>วันที่ | |
| | | มัครรับทราบแล้ว ด้วยความรู้ที่ดีที่<br>ประโยชน์ต่างๆ ต่ออาสาสมัครแล้ว | ์สุดของข้าพเจ้า และ |
| <br>แพทย์ผู้วิจัย/ผู้ให้การปรึกษา<br>(พิมพ์หรือเขียนตัวบรรจง) | <br>ลายเซ็น | วันที่ | |




# Appendix 1 (continued): Informed Consent Form to Participate in iTAP Study (English Language)

<u>Title of Study</u>: A phase III, placebo controlled, double blind, randomized clinical trial to assess the efficacy and safety of tenofovir disoproxil fumarate given from 28 weeks' gestation until 2 months postpartum to Hepatitis B (HB) virus chronically infected, HBsAg and HBeAg positive pregnant women to prevent perinatal transmission of HBV to their infants who receive HBV passive-active immunization(iTAP).

Short title: Maternal antiviral prophylaxis to prevent perinatal transmission of HBV in Thailand

#### **Purpose**

You, <u>as well as your baby</u>, are being invited to participate in a research study of tenofovir, which may help to prevent transmission of the hepatitis B virus (called HBV), from HBV-infected pregnant women to their babies. The purpose of this study is to determine if taking tenofovir, during the last trimester of pregnancy until two months after delivery can reduce the risk of HBV transmission to your baby.

This form, along with discussions with your physician, will provide you detailed information about the study so that you can decide if you want to participate.

Your participation in this research study would be entirely voluntary. You are free to decline to participate today or to withdraw from the study at any future date without jeopardizing your access to standard medical care or your possible participation in future research studies.

This research study is collaboration between researchers and doctors and is supported by the Ministry of Public Health in Thailand, the National Institutes of Health (NIH) and the Centers for Disease Control and Prevention (CDC) in the USA.

## Nature of the Study

People chronically infected with hepatitis B virus have small parts of the virus called hepatitis B **surface** antigens (HBsAg) in their blood that can be detected by a simple blood test, widely available in Thailand. An estimated 2 to 3 million adults in Thailand are chronically infected with the Hepatitis B virus (HBV). The inflammation caused by HBV can damage the liver cells and cause liver cirrhosis and cancer after a long time, usually in adulthood.

You are pregnant and infected with HBV, and you are not infected with HIV (HIV and HBV are two different viruses). Currently, all infants born to mothers infected with HBV must receive HBV vaccine at birth, 1, 2, 4 and 6 months of age to protect against this infection. In addition, the Pediatric Society of Thailand recommends that they also receive specific immunoglobulin (antibodies against HBV) within the first hours after birth.

However, pregnant women with high levels of HBV in the blood have a risk of about 10% to 12% of transmitting the virus to their baby, despite the use of the HBV vaccine and antibodies against HBV for prevention. Most adults with high levels of HBV in the blood also have another antigen that can be detected, called HB e antigen (HBeAg). In young people with HBsAg and HBeAg, the immune system has not reacted to HBV infection. If it does react, the level of a liver enzyme (called ALT, or most often SGPT in Thailand) in the blood is higher than normal. The amount of SGPT in the blood can be measured using a simple blood test, also widely available in Thailand. If the level of SGPT is normal, it means that the immune system is not reacting against HBV. In this study, only pregnant women with HBeAg detected in the blood and normal levels of SGPT (less than 30 U/L) will be asked to join the study.

Tenofovir is an anti-HBV drug approved by the Thai Food and Drug Administration for the treatment of HBV. It is unknown if taking tenofovir during the last trimester of pregnancy until two months after delivery will help reduce the risk of HBV transmission to the baby. More than 1370 pregnant women have received tenofovir and there is no evidence that tenofovir causes harm to the fetus. Tenofovir

9 4 9 167 ค. 8 พ.ศ. 2558 คณะกรรมการจรียธรรมการวิจัยในมนุษย์ สถาบันพัฒนาการจุ้นกรวงสามรูวิจัยในมนุษย์ (สคม.

interferes with bone metabolism. However, among infants of women receiving combination ARV regimens during pregnancy, in utero exposure to tenofovir does not appear to have an effect on infant birth weight or infant growth.

In this study, 328 HBV-infected pregnant women, at least 18 years old, will be enrolled over 2 years in 19 public hospitals throughout Thailand: provincial/regional hospitals in Phayao hospital, Chiang Rai Prachanukroh Hospital, Prapokklao Hospital, Chonburi Hospital, Bhumibol Adulyadej Royal Air Force hospital in Bangkok, Health Promotion Center Region 10, Chiang Mai, Lamphun Hospital, Chiang Kham Hospital, Mae Chan Hospital, Banglamung hospital, Nakornping Hospital, Nopparat Rajathanee Hospital, Khon Kaen Hospital, Samutsakhon Hospital, Nakhonpathom Hospital, Samutprakarn Hospital, Lampang Hospital, Maharaja Nakornratchasrima Hospital and Ranong Hospital.

Each mother will be assigned by chance to one of the following two equal groups:

- **Group 1 (tenofovir)**: Women will receive one tablet of tenofovir 300 mg to take once a day from 28 weeks' gestation until two months after delivery.
- **Group 2 (placebo)**: Women will receive one tablet of inactive substance to take once a day from 28 weeks' gestation until two months after delivery.

All babies will receive HBV immunoglobulin and vaccine, which is recommended by the Royal College of Thai Pediatricians for babies whose mothers have HBV infection. Neither you nor your doctor will be able to choose or to know which group you will be in.

### Study Procedures for You.

We will first propose to draw blood (5 cc or less than half a tablespoon) for a test to know if you have hepatitis B e antigen (HBeAg) in your blood and to measure the level of SGPT. These tests have to be done during pregnancy, early enough to know the results at the latest at 28 weeks of gestation.

We will ask for your authorization to record laboratory test results performed as part of your routine clinical care before your consent to participate in this study.

Only women with HBeAg, likely to have a high quantity of virus in their body and a high risk of transmission of HBV, will be asked to continue to participate in the study. However, if the level of SGPT is too high (more than 30 U/L), you will not be asked to participate further and we will recommend you to visit a specialist of HBV to advise you on further tests or treatment as necessary.

If you have hepatitis B e antigen (HBeAg) and a level of SGPT equal or below 30 U/L, it will be proposed that you continue in the study. At 26 weeks of pregnancy, your medical history will be reviewed and you will undergo a physical examination and blood will be drawn for some more blood tests (about 16 cc or approximately a tablespoon) to see if you qualify for the study.

If you qualify to continue in the study, you will be assigned by chance to one of the two groups at 28 weeks of gestation and you will receive one bottle of study drug. You will have to take one tablet once a day, at the same time every day until two months after delivery. You will not know if you are taking tenofovir or placebo tablets. After enrollment, you will receive routine medical check-ups provided at the antenatal clinic as for any pregnant woman, and we will evaluate your health for any apparent side effects of the therapy, with a blood draw (33 to 38 cc or approximately two and a half tablespoons) at each visit. Study visits will occur at 28, 32, 36 weeks' gestation during pregnancy. A special blood draws (30 cc or approximately two tablespoons) for peripheral blood mononuclear cells (PBMC) may be collected at different visits. The PBMC will be stored for future studies to analyze the of immune response against HBV before the occurrence of flares.

When you go into labor, you will go immediately to the maternity unit. When you arrive at the maternity unit, a blood draw will be performed for blood tests (about 10 cc or approximately a tablespoon). The blood tests are for: complete blood count (CBC), SGPT, creatinine level (to measure renal function), serum phosphorus (to measure bone metabolism), HBV DNA viral load, and tenofovir level to follow the effects of the treatment.


0 8 ฟิค. 2558 คณะกรรมการจริยธรรมสาราจัยในมนุษฮ สถาบันพัฒนาการคุ้มครองการวิดีสินมนุษฮ์ (สคม. After delivery, you will be asked to come for study visits at 1, 2, 3, 4, 6, and 12 months to follow the effects of the treatment. You will have a physical exam and a blood draw (about 38 to 43 cc or approximately three tablespoons) to follow the evolution of SGPT, serum phosphorus and creatinine, HBV DNA viral load, HBeAg and complete blood count.

During or after the period of treatment, you should call right away your doctor or the nurse in charge of the study (see contact numbers at the end of this form) if you suffer from another condition, in particular if you get the following signs or symptoms of liver problems:

- Your skin or the white part of your eyes turns yellow (jaundice).
- · Your urine turns dark.
- Your stools turn light in color.
- You don't feel like eating food for several days or longer.
- You feel sick to your stomach (nausea).
- You have lower stomach area (abdominal) pain.

If your level of SGPT increases to 60 IU/L or more, you will be contacted and asked to return to the clinic, as soon as possible within 3 days, for another blood draw to confirm the SGPT elevation. If you notice any of the signs or symptoms listed above, you should return immediately to the clinic. If the increase is confirmed on the second blood draw, you will be asked to come again two weeks later for a new blood draw. If, at any time, your level of SGPT is over 150 IU/L, your physician will consider reintroduction of the study treatment. You will then be followed in the study until one year after delivery. If you are started on treatment, after the end of your participation in the study, your treatment will be replaced with the commercial form of tenofovir or you will be told if you were receiving the inactive form of the study drug,, and followed by your internist according to the current guidelines. It is not known for how long you will have to continue this treatment.

## Study Procedures for Your Baby.

Your baby will receive HB immunoglobulin within 12 hours of birth, and HBV vaccine within 12 hours of birth and at 1, 2, 4 and 6 months of age. You will be asked to bring your baby 1, 2, 4, 6, 9 and 12 months after birth for clinical safety evaluation and determination of HBV status.

A blood sample from your baby (2 to 4 cc or no more than a teaspoon) will be taken at each visit to check for any side effects of the prophylaxis and to look for evidence of HBV infection.

<u>Breast-feeding:</u> You can breast-feed your baby because the risk to transmit HBV to your baby is not increased by breast-feeding.

<u>Safeguards for Your Health.</u> You and your baby will undergo careful check-ups throughout the study. It is very important that you keep all study appointments and take treatments as instructed. At each visit, you will be asked if you or your baby have suffered from any other condition, are taking any other medicines or have experienced any adverse events. If you need to, you may contact us or come to the clinic at any time, even if no visit is planned.

Costs to You for Participation. There is no cost to you or your baby for the medication, extra clinic visits or laboratory tests associated with this study. All study participants will receive 300 baht (in all sites except Bangkok site where the amount will be 400 Baht) at each visit to compensate for transportation costs (if justified, the research team at site will compensate for higher transportation costs). The study will pay for the cost of the immunoglobulin (HBIg) for all participants' babies.

Significant New Findings. Any significant new findings that develop during the study that could affect you, your baby, or your willingness to continue participation will be made available to you as soon as possible.

**อนุ่งเก็** 0.8 ปี.ค. 2558 คณะกรรมการจริยชรางเลารวิจัยในมนุษย สถาบันพัฒนาการคุ้มลสตาว เช่นอีถีนมนุษย์ (สคม

<u>Withdrawal from the Study</u>. Your physician could recommend that you withdraw from the study if any condition or severe adverse event developed that would make continued participation harmful to you or your baby. In such a case, you would be treated with the standard of care available. However, you should not interrupt your treatment without medical advice to avoid a sudden increase of the HBV virus in your liver without medical supervision.

<u>Alternatives to Participation</u>. You are completely free to choose not to participate in or to withdraw yourself or/and your baby from this study at any time. Your alternative to participation in this study is the usual care available to a pregnant woman with HBV infection at your health care facility.

<u>Confidentiality</u>. You and your baby's participation in this study will be kept confidential and will not be communicated to anyone without your written permission.

Confidentiality of Records. Efforts will be made to keep you and your child's personal information confidential. Your medical records will be kept confidential. They will be disclosed to you, to those heath care providers directly involved in your care and, for study monitoring or auditing purposes, to the members of the research team, the Thai Food and Drug Administration (FDA), the Ethics committee of Institute for the Development of Human Research Protections, local Ethics Committee in your hospital, study staff, study monitors, drug companies supporting this study (drug company names) and study sponsors. All study forms will be coded by number and your name will not be recorded on these forms. Only these code numbers will be kept in the study database that will be used for analysis. Any publication of this study will not use your child's name or identify you child personally. However, we cannot guarantee absolute confidentiality and your personal information may be disclosed if required by law.

Repository of Blood Specimens. Blood samples taken as part of the study, identified by code, will be kept for confirmation of results if needed until ten years after the end of the study. Blood samples will be stored at the IRD-PHPT Laboratory under Faculty of Associated Medical Sciences, Chiang Mai University, where only approved researchers and staff will have access to them. People who work at the facility will also have access to you and your baby's samples to keep track of them, but these people won't be able to directly identify your baby. Blood samples will not be sold or directly used to produce commercial products. You can withdraw you and your baby's blood samples from the sample repository at any time, and they will be immediately destroyed by autoclave following the standard procedure at the Faculty of Associated Medical Sciences, Chiang Mai University.

Remaining bloods samples may also be stored for confirmation of any test done, or other evaluations that may help understand the mechanism of HBV perinatal transmission and liver damage. Also, tests might look at how a person's genetic makeup (your DNA and RNA) either protects them or puts them at greater risk of HBV transmission, viral flare or drug side effects (host genetics and pharmacogenomics). You may approve or refuse the use of DNA and total RNA tests by ticking the right box in the informed consent form that selects your choice of sample storage. If other studies were deemed necessary, we would request additional consent and this would be submitted to the Ethics Committee as a specific study.

<u>Policy Regarding Research Related Injuries</u>. Immediate necessary care is available free of charge to you if you or your baby have a medical problem related to participation in this study. However, the study is not responsible for treatments unrelated to the study and no financial compensation will be provided.

## Risks to You / Your Child.

If you are assigned to take inactive substance (but you will not know during the study if you take tenofovir or placebo), there will be no difference from the standard of care.

Some people who have taken medicines like tenofovir have developed serious liver problems called hepatotoxicity, with liver enlargement (hepatomegaly) and fat in the liver (steatosis).

**0 1 1 10** 0 8 ปี ค. 2558 คณะกรรมการจริยธรรมลารวิจัยในม**นุษ**ย If you are assigned to take tenofovir, side effects can include: kidney damage or failure, bone thinning, gas, dizziness, feeling tired, low phosphate in the blood and allergic reaction, which may include fever, rash, upset stomach, vomiting, loose or watery stools, abdominal pain, achiness, shortness of breath or general feeling of illness.

One of the main possible risks of taking tenofovir is a reactivation of the hepatitis (inflammation or irritation of the liver). You should be aware that your liver function tests may increase, and symptoms associated with hepatitis may worsen at some point during the study treatment or in the weeks or months after you stop tenofovir. This is the reason why we will ask you to come regularly at all study visits and inform your physician if you cannot come so another appointment can be scheduled.

One of the potential risks associated with tenofovir during pregnancy is bone thinning in the newborn and slightly slower growth of infants.

The risks and discomforts of blood drawing include pain, swelling, bruising, inflammation of a vein and fainting. If necessary, you and your infant will receive appropriate care from your physician.

Benefits to You/Your Child. During the study, you and your baby will be provided with close medical follow-up for safety.

If you are assigned to take tenofovir you may have a decreased risk of HBV transmission to your baby. If you are assigned to receive placebo there is no direct benefit to your child but you and your child will benefit from the close follow-up and monitoring with the study.

<u>Further Questions</u>. At any time, if you have further questions about this study or your rights and benefits as a participant, you may contact:

## • The Ethic committee of research in Human

| Institute for th | ne Develo | opment of | Human | research | <b>Protections</b> |
|---|---|---|---|---|---|

Building 8, Floor 7, room 702 Medical Sciences Department

Ministry of Public Health 11000 Tel. 02-5913541, 02 -5913517 Fax. 02-5914125

| Or the your hospital's Ethics Committee | |
|-------------------------------------------|-------------|
| | Telephone # |
| (Representative of your hospital's Ethics | Committee) |

For questions about the research project, your rights, and research-related injuries, you may contact a doctor independent from the research team:

Name: Dr. Sorakij Bhakeecheep

Address: National Health Security Office (NHSO)

The Government Complex Commemorating His Majesty the King's 80th Birthday Anniversary

5th December, B.E. 2550 (2007) Building B

120 M. 3 Chaengwattana Road, Lak Si District, Bangkok 10210

Tel: +66 2141 4000Fax: +66 2143 9730-1

0 1 3 16 1 0 8 ปี.ค. 2558 คณะกรรมการจริยธรรมการวิจัยในมนุษย์ สถาบันพัฒนาการคุ้มกรองการวิจัยในมนุษย์ (สกม

| Maternal antiviral prophylaxis to prevent perinata | I transmission of HBV in T | hailand, version 3.0 dated 20 April 2015 | |
|---|---|---|---|
| The investigator responsible for safe | eguarding your wel | fare and the welfare of your baby, | |
| Dr. | (1 | Principal investigator name at each sit | æ) |
| Address: | | | , |
| Telephone # Office: | Home: | Mobile: | - |
| Fax: # | | | |
| or | | (name and title of Hospital Director) | ) |
| Consent to participate in this study | | | |
| the risks, and benefits of participal<br>completely free to withdraw your pa<br>your rights or those of your baby | ion have been full<br>articipation or your<br>to receive the bes | of this study, the procedures to be for<br>y explained to you. You know that y<br>baby's participation at any time without<br>the medical care otherwise available. For<br>loss of benefits to which you may o | you are still<br>out affecting<br>Refusing to |
| l agree for my participation and my | child's participation | in this study. | |
| I agree that my laboratory test resul<br>study can be recorded in the study o<br>Yes □ No □. | | nical care before my consent to partic | ipate in this |
| Woman's Name (typed or printed) | Signature | Date | |
| Woman's legal representative<br>/Guardian (if appropriate) | Signature | Date | |
| "I agree for my child's participation i | n this study." | | |
| Name of the Father of the child (If available and with the woman's c | Signature<br>onsent, typed or pr | Date inted) | |
| Witness Name (typed or printed) | Signature | Date | |
| Witness Name (typed or printed) | Signature | <br>Date | |




| Maternal antiviral prophylaxis to prevent perina | atal transmission of HBV in Thail | and, version 3.0 dated 20 April 2015 |
|---|---|---|
| I have explained the purpose of the purpose, procedures, risks an | | To the best of my knowledge, she understands r baby. |
| Investigator/Counselor Name (Typed or printed) | Signature | <br>Date |
| in this consent form. | rage and use of my stor | of my decision ed specimens for future test(s) as discussed red specimens for future test(s) as discussed |
| I do not permit to store my bloc | NA (pharmacogenomi | |
| Participant's Name (typed or print | ted) Signature | <br>Date |
| Witness Name (typed or printed) | Signature | <br>Date |
| I have explained the purpose of the patient understands the purpo | | t. To the best of my knowledge, the patient on benefits to the patient. |
| Physician/Counselor Name (Typed or printed) | Signature | <br>Date |




## Appendix 2: Exempted Congenital Anomaly/Birth Defect (Listed by Body Site)

#### Abdomen/Groin/Pelvis

Diastasis recti

Hernia, inguinal or umbilical without mention of

obstruction or gangrene

Hip click, with no follow-up or therapy

Umbilical artery, single

Umbilical cord atrophy

Urachus, patent

Chest/Thorax

Breast hypertrophy

Inverted nipples

Nipples, anomalies of

Rib, cervical

Face/Mouth

**Brushfield Spots** 

Duct, lacrimal, stenosis, stricture, or obstruction

of

Epicanthal folds

Epstein's Pearls

Esotropia

Exotropia

Gum cysts - includes epulis, ranula, mucocele

Macrocheilia (large lips)

Microcheilia (small lips)

Nose, congenital deviation of septum of

Nose, flat bridge of

Nystagmus

Palate, high-arched

Palsy, facial

Protruding tongue

Sclera, blue

Teeth, natal

Tongue tie


Foot/Toe

Foot, rocker-bottom

Tibia, torsion of

Toes, long

Toes, overlapping

Toes, webbing

Hand/Finger

Clinodactyly of fifth finger

Fingers, long

Metatarsus varus or adductus

Polydactyly, postaxial

Simian crease

Head/Neck

Dolichocephaly

Ear, malformations of external ear

Ear, preauricular sinus, cyst, or pit of

Fontanelle, large or small

Occiput, flat or prominent

Scaphocephaly, no mention of craniosynostosis

Neck, webbing or redundant skin folds of

Neck, short

Skin

**Albinism** 

Birthmark, NOS

Dimple, sacral, pilonidal

Lanugo, persistent or excessive

Mongolian spots

Neonatal acne

Neoplasm, benign

Nevus, flammaeus

Skin tags on hands or feet

**Urogenital Rectal** 

Anal fissure

Anus, skin tags of

Clitoromegaly, enlarged clitoris, hypertrophy

Hydrocele

Hymen, imperforate

**Phimosis** 

Redundant foreskin

Scrotum, hypoplastic due to cryptorchidism


Testes, torsion of, or torsion of spermatic cord

Testes, retractile

Testicle, undescended (unilateral, bilateral or

NOS)

Vagina, embryonal cyst of

Vagina, tag of


# Exempted Congenital Anomaly/Birth Defect (Listed Alphabetically)

Albinism

Anal fissure

Anus, skin tags of

Birthmark, NOS

Breast hypertrophy

**Brushfield Spots** 

Clinodactyly of fifth finger

Clitoromegaly, enlarged clitoris, hypertrophy

Diastasis recti

Dimple, sacral, pilonidal

Dolichocephaly

Duct, lacrimal, stenosis, stricture, or obstruction

of

Ear, malformations of external ear

Ear, preauricular sinus, cyst, or pit of

Epicanthal folds

Epstein's Pearls

Esotropia

Exotropia

Fingers, long

Fontanelle, large or small

Foot, rocker-bottom

Gum cysts - includes epulis, ranula, mucocele

Hernia, inguinal or umbilical without mention of

obstruction or gangrene

Hip click, with no follow-up or therapy

Hydrocele

Hymen, imperforate

Inverted nipples

Lanugo, persistent or excessive

Macrocheilia (large lips)

Metatarsus varus or adductus

Microcheilia (small lips)

Mongolian spots

Neck, short

Neck, webbing or redundant skin folds of

Neonatal acne

Neoplasm, benign

Nevus, flammaeus

Nipples, anomalies of

Nose, congenital deviation of septum of

Nose, flat bridge of

Nystagmus

Occiput, flat or prominent

Palate, high-arched


Palsy, facial

**Phimosis** 

Polydactyly, postaxial

Protruding tongue

Redundant foreskin

Rib, cervical

Scaphocephaly, no mention of craniosynostosis

Sclera, blue

Scrotum, hypoplastic due to cryptorchidism

Simian crease

Skin tags on hands or feet

Teeth, natal

Testes, retractile

Testes, torsion of, or torsion of spermatic cord

Testicle, undescended (unilateral, bilateral or

NOS)

Tibia, torsion of

Toes, long

Toes, overlapping

Toes, webbing

Tongue tie

Umbilical artery, single

Umbilical cord atrophy

Urachus, patent

Vagina, embryonal cyst of

Vagina, tag of



อลาบันพัฒนาการคุ้มครองการวิจักใน**มนุษย์ (สกม** 

# Appendix 3: Screening program for symptoms possibly associated with mitochondrial dysfunction in the EPF cohort (68)

List of symptoms leading to the initial selection of the file (at least 1 major sign or 2 different minor signs at two different follow-up consultations)\*

#### **NEUROLOGICAL SIGNS**

## Major signs

Non-febrile seizures, including neonatal seizures

Febrile seizures, either repeated (≥ 2 episodes) or in children aged < 6 months

Peripheral neuropathy

Acquired microcephaly

Cranial nerves paresis

Impaired cognitive development (for children older than 1 year)

Cerebellar dysfunction and ataxia

Motor disabilities, paraparesis, spasticity

Abnormalities on MRI or CT scan

## Minor signs

Febrile seizures

Isolated changes in muscular tone, hyper-and hypotonia

Behavorial disturbances and hyperactivity disorder

Hypotonia, hypertonia

Moderate cognitive delay

## **OTHER ORGANS**

## Major signs

Pancreatitis (including biological signs)

Cardiomyopathy

Myopathy

Decrease in visual acuity, retinopathy

Abnormal ocular motor function

Nystagmus

Deafness

Unexplained death

#### Minor signs

Increase in transaminase levels\*

Persistent anemia, neutropenia or thrombopenia

Tubular defect

01116 0 8 ปีเค. 2558 กณะการมการจริยธรรมการวิจัยในมนุษย์

<sup>\*</sup> The abnormalities selected for this screening correspond to factors systematically tested as part of the French perinatal survey (EPF). The determinations of lactates, creatine phosphor kinase and lipase plasma level introduced during 1999 were not taken into account in this screening.

## Appendix 4: Cockcroft-Gault formula for women

# (140-age [in years]) x weight [in kg] x0.85 (72 x creatinine [in mg/dL])

Calculation on line at: http://nephron.com/cgi-bin/CGSI.cgi



## Appendix 5: How to Measure Head Circumference, Length and Weight

Growth is assessed at each visit by measuring the weight, height, and head circumference. (from PACTG 219)

## a) How to Measure Head Circumference

The measuring tape is placed across the forehead with the lower border of the tape just above the eyebrows, around the head, above the ears and over the occipital prominence at the back of the head. Pull tape firmly to compress the hair and underlying soft tissues. Positioning of the tape over the forehead and occiput should be done to yield the maximum head circumference. Record head circumference in centimeters to the nearest 0.1 cm.

## b) How to Measure Length

For children up to 24 months, measure supine on a standard measuring board. Keep child's legs straight and toes up, bringing movable footboard to rest firmly against child's heels. Measure height in centimeters to the nearest 0.1 cm.

## c) How to Measure Weight

All weights should be obtained without shoes, diapers and clothing; whenever possible, the same scales should be used for these measurements. The scale should be set to zero each time. Measure weight to the nearest gram.



# Appendix 6: Additional Informed Consent Form to Participate in Tenofovir Plasma Level Measurements (Thai Language)

## แบบแสดงความยินยอมเข้าร่วมโครงการวิจัยเพิ่มเติมสำหรับการตรวจวัดระดับยาทีโนโฟเวียร์ในพลาสมา

## <u>วัตถุประสงค์</u>

ท่านและบุตรของท่านอยู่ระหว่างการเข้าร่วมการศึกษาวิจัย "ยาต้านไวรัสสำหรับมารดาเพื่อป้องกันการถ่ายทอด เชื้อไวรัสตับอักเสบบีจากมารดาสู่ทารกในประเทศไทย" ความเสี่ยงที่สำคัญที่อาจเกิดขึ้นได้อย่างหนึ่งที่เกี่ยวกับการ รับประทานยาทีโนโฟเวียร์ในช่วงตั้งครรภ์คือทารกแรกเกิดมีภาวะกระดูกบางและการเจริญเติบโตของทารกช้าลงเล็กน้อย ได้มีการวิจัยประเด็นนี้ในทารกที่คลอดจากมารดาที่ติด เชื้อไวรัสชนิดอื่นๆ แต่ไม่มีการวิจัยในทารกที่คลอดจากมารดาที่ติด เชื้อไวรัสชนิดอื่นๆ แต่ไม่มีการวิจัยในทารกที่คลอดจากมารดาที่ติด เชื้อไวรัสตับอักเสบบีเรื้อรัง

ระดับของยาที่โนโฟเวียร์ในเลือดของแต่ละคนนั้นมีความแตกต่างกัน และเป็นไปได้ว่าความหนาแน่นของมวล กระดูกที่ลดลงมีความสัมพันธ์กับระดับยาที่โนโฟเวียร์ในกระแสเลือดที่สูงในระหว่างที่รับการรักษา

เพื่อช่วยอธิบาย 2 คำถามนี้ ทางโครงการขอเสนอให้ท่านเข้าร่วมในการประเมินระดับยาทีโนโฟเวียร์ในพลาสมาใน ระหว่างตั้งครรภ์

แบบแสดงความยินยอมเข้าร่วมการวิจัยนี้ มีรายละเอียดข้อมูลเกี่ยวกับการประเมินเพิ่มเติมเหล่านี้ ซึ่งแพทย์หรือ พยาบาลที่ดูแลท่านจะอธิบายข้อมูลให้ท่านทราบเพื่อให้ท่านสามารถตัดสินใจได้ว่าท่านต้องการเข้าร่วมในการวิจัยนี้หรือไม่ การเข้าร่วมในการประเมินการวิจัยเพิ่มเติมนี้ของท่านจะเป็นไปโดยสมัครใจอย่างเต็มที่ ท่านมีอิสระที่จะปฏิเสธการเข้าร่วม การวิจัยในวันนี้หรือเปลี่ยนแปลงการตัดสินใจในอนาคตได้ทุกเมื่อโดยไม่สูญเสียโอกาสในการเข้าร่วมโครงการวิจัยนี้หรือการ ได้รับบริการทางการแพทย์ที่ได้มาตรฐานของท่าน หรือโอกาสในการเข้าร่วมการศึกษาวิจัยอื่นๆ ในอนาคตของท่าน

## ลักษณะของการวิจัย

ทางโครงการจะศึกษาความสัมพันธ์ระหว่างระดับของยาทีโนโฟเวียร์ในกระแสเลือดในระหว่างตั้งครรภ์และความหนาแน่น ของมวลกระดูกในมารดาและบุตร จะประเมินค่าเฉลี่ยความเข้มข้นของยาทีโนโฟเวียร์ในกระแสเลือดโดยยึดตามค่าความ เข้มข้นที่สังเกตได้ในช่วงเวลาแตกต่างกันหลังจากได้รับประทานยาที่ใช้ในการวิจัย

## ขั้นตอนการวิจัยสำหรับท่าน

ทางโครงการจะขอให้ท่านรับประทานยาที่ใช้ในการวิจัยทุกเช้าก่อนนัดหมายการวิจัยในสัปดาห์ที่ 32 และ 36 ของการ ตั้งครรภ์ สำหรับนัดหมายการวิจัย 2 ครั้งนี้ จะขอให้ท่านมาโรงพยาบาลในช่วงเช้าก่อนที่ท่านจะรับประทานยาที่ใช้ในการ วิจัยของท่านตามปกติ จะมีการเจาะเลือดท่าน (ปริมาณ 2 ซีซีหรือครึ่งช้อนชา) ก่อนที่ท่านจะรับประทานยาที่ใช้ในการวิจัย หลังจากการเจาะเลือดเรียบร้อยแล้ว ท่านจะต้องรับประทานยาที่ใช้ในการวิจัยของท่านตามปกติ ซึ่งจะเป็นช่วงเวลาเดิมที่ ท่านเคยรับประทานยาที่ใช้ในการวิจัยในทุกเช้า หลังจากนั้นจะมีการเจาะเลือดตามตารางเวลาที่กำหนดในช่วงระหว่างครึ่ง ชั่วโมงถึง 3 ชั่วโมงหลังจากท่านรับประทานยาที่ใช้ในการวิจัยแล้ว และจากนั้นจะมีการเจาะเลือดท่านอีก 2 ซีซีหลังจาก 1 ชั่วโมงไปแล้ว

## ระยะเวลาของการเข้าร่วมโครงการวิจัยของอาสาสมัคร

จะทำการเจาะเลือดเพิ่มเติมนี้ 2 ครั้งในนัดหมายที่มาฝากครรภ์เมื่ออายุครรภ์ 32 สัปดาห์และเมื่อ 36 สัปดาห์

0 % ปี ค.ศ. 2558 กณะกรรมการจริยธรรมดารวิจัยในมนุษย


สถาบันพัฒนาการคุ้มกรองการวิจัยในมนุษย์ (สคม.

## ค่าใช้จ่ายในการเข้าร่วมโครงการวิจัยของท่าน

ท่านไม่ต้องเสียค่าใช้จ่ายเพิ่มเติมสำหรับการเข้าร่วมโครงการวิจัยนี้ จะมีค่าชดเชยสำหรับการเสียเวลาของท่านเนื่องจาก ท่านจำเป็นต้องอยู่ในโรงพยาบาลเพื่อการเจาะเลือด นอกจากนี้จะมีค่าใช้จ่ายในการเดินทางให้แก่ท่านที่เข้าร่วมในนัดหมาย การวิจัยเหล่านี้ด้วย

การค้นพบข้อมูลและข่าวสารใหม่ๆ ที่เกี่ยวข้อง

ทางโครงการจะแจ้งให้ท่านทราบเกี่ยวกับการค้นพบข้อมูลต่างๆ ที่เกิดขึ้นใหม่ในระหว่างการวิจัยโดยเร็วที่สุดซึ่งอาจมีผลต่อ ความสมัครใจในการเข้าร่วมโครงการวิจัยต่อไปของท่าน

## การถอนตัวออกจากการวิจัย

ท่านมีอิสระที่จะตัดสินใจไม่เข้าร่วมในการประเมินนี้เมื่อใดก็ได้โดยไม่สูญเสียโอกาสการได้รับบริการทางการแพทย์ที่ได้ มาตรฐานของท่าน หรือโอกาสในการเข้าร่วมการศึกษาวิจัยอื่นๆ ในอนาคตของท่าน

## การปกปิดความลับ

การเข้าร่วมโครงการวิจัยนี้ของท่านจะถูกปกปิดเป็นความลับและจะไม่แจ้งให้ใครทราบโดยไม่ได้รับความยินยอมซึ่งเป็นลาย ลักษณ์อักษรจากท่าน

## การปกปิดความลับของข้อมูล

ทางโครงการจะใช้ความพยายามเพื่อเก็บข้อมูลส่วนตัวของท่านไว้เป็นความลับ ข้อมูลทางการแพทย์ของท่านจะถูกเก็บ รักษาไว้เป็นความลับ และจะเปิดเผยข้อมูลให้ท่านทราบตลอดจนผู้ให้การดูแลรักษาท่านโดยตรงเพื่อการติดตามการวิจัย หรือเพื่อวัตถุประสงค์ในการตรวจสอบการวิจัย สมาชิกของคณะผู้วิจัยสำนักงานคณะกรรมการอาหารและยาประเทศไทย (เอฟดีเอ) คณะกรรมการจริยธรรมการวิจัยในมนุษย์ สถาบันพัฒนาการคุ้มครองการวิจัยในมนุษย์คณะกรรมการพิจารณา ด้านจริยธรรมการวิจัยในโรงพยาบาลของท่าน เจ้าหน้าที่วิจัย ผู้ติดตามการวิจัย บริษัทยาที่สนับสนุนยาในการวิจัยนี้ (บริษัท กิลเลียด) และผู้ให้การสนับสนุนการวิจัย แบบบันทึกข้อมูลทั้งหมดของโครงการวิจัยจะใช้หมายเลขรหัส และไม่มีการระบุชื่อ ของท่านในแบบบันทึกข้อมูลเหล่านี้ ทางโครงการจะบันทึกเฉพาะรหัสไว้ในฐานข้อมูลการวิจัยเพื่อใช้ในการวิเคราะห์เท่านั้น จะไม่ใช้ชื่อของท่านหรือระบุตัวท่านเป็นการส่วนตัวในการตีพิมพ์เอกสารใดๆ ของการวิจัยนี้ อย่างไรก็ตามทางโครงการไม่ สามารถรับรองการรักษาความลับไว้ได้อย่างสิ้นเชิง และข้อมูลส่วนตัวของท่านอาจจะถูกเปิดเผยหากจำเป็นโดยข้อบังคับ ทางกฎหมาย

## <u>นโยบายที่เกี่ยวข้องกับการได้รับอันตรายจากการวิจัย</u>

ท่านจะได้รับการดูแลรักษาที่เหมาะสมที่มีทันทีหากท่านมีปัญหาทางการแพทย์ที่เกี่ยวข้องกับการเข้าร่วมในโครงการวิจัยนี้ โดยไม่ต้องเสียค่าใช้จ่าย อย่างไรก็ตามโครงการวิจัยจะไม่รับผิดชอบสำหรับการรักษาที่ไม่เกี่ยวข้องกับการวิจัย และจะไม่มี การจ่ายค่าชดเชยแต่อย่างใด

## ความเสี่ยงของท่าน

ความเสี่ยงอันเนื่องมาจากการเจาะเลือดเพิ่มเติม 2 ครั้งนั้นคือความเสี่ยงที่เกี่ยวข้องกับการเจาะเลือดโดยทั่วไป ความเสี่ยง และอาการไม่สบายจากการเจาะเลือดได้แก่ ความรู้สึกเจ็บ อาการบวม การฟกซ้ำ การอักเสบของเส้นเลือดดำ และเป็นลม หากจำเป็นท่านจะได้รับการดูแลรักษาที่เหมาะสมจากแพทย์ผู้ดูแลท่าน

0 8 ปี ค.ศ. 2558 คณะกรรมการจริยธรรมดารวิจัยในมนุษย ผลประโยชน์ของท่าน

วัตถุประสงค์ของการวิจัยนี้คือเพื่อทำการประเมินและให้เข้าใจความสัมพันธ์ที่เป็นไปได้ระหว่างยาทีโนโฟเวียร์และความ หนาแน่นของมวลกระดูกได้มากขึ้น อย่างไรก็ตามท่านจะไม่ได้รับประโยชน์โดยตรงจากผลของการวิจัยนี้เนื่องจาก ผลการวิจัยจะสรุปเมื่อสิ้นสุดการวิจัยแล้ว

<u>ปัญหาหรือข้อซักถามเพิ่มเติม</u> เมื่อใดก็ตามหากท่านมีคำถามเพิ่มเติมเกี่ยวกับการวิจัยนี้ หรือเกี่ยวกับสิทธิและผลประโยชน์ ของท่านในฐานะอาสาสมัครท่านสามารถติดต่อ:

| 02-5913517 โทรสาร: 02-5914125<br>ลของท่าน |
|-------------------------------------------------------|
| ลของท่าน |
| งพยาบาลของท่าน) |
| เกิดจากการวิจัย ท่านสามารถติดต่อแพทย์ผู้ซึ่งเป็นอิสระ |
| 50 อาคาร บี |
| 0 |
| 9730-1 |
| 9730-1 |
| ของท่าน |
| (ชื่อผู้วิจัยหลักในสถานที่วิจัยแต่ละแห่ง) |
| · |
| <br>โทรศัพท์มือถือ: |
| (ชื่อและตำแหน่งผู้อำนวยการโรงพยาบาล) |

การแสดงความยินยอมเข้าร่วมโครงการ

เมื่อท่านเซ็นชื่อในแบบแสดงความยินยอมเข้าร่วมโครงการวิจัยนี้ ท่านยอมรับว่าได้มีการอธิบายวัตถุประสงค์ของการ ้ศึกษาวิจัย ขั้นตอนปฏิบัติตามแผนการวิจัย ความเสี่ยง และผลประโยชน์ต่างๆ ของการเข้าร่วมโครงการวิจัยนี้ให้ท่านฟังโดย ละเอียดแล้ว ท่านทราบว่าท่านมีอิสระที่จะถอนตัวท่านออกจากการเข้าร่วมการวิจัยได้ตลอดเวลา โดยไม่มีผลกระทบใดๆ ต่อสิทธิของท่านในการได้รับการรักษาทางการแพทย์ด้วยวิธีการอื่นๆ ที่ดีที่สุดเท่าที่มีอยู่ การปฏิเสธเข้าร่วมโครงการ หรือ การถอนตัวออกจากการเข้าร่วมโครงการวิจัยจะไม่มีความผิดใดๆ และจะไม่ทำให้ท่านสูญเสียผลปุระโยชน์อื่นๆ ที่ท่านควร ได้รับตามสิทธิ์ที่ท่านพึงมี

0 94 31 67 nwensenn 8 30 57 57 57 58 50 1 4 4 4 0

# Appendix 6 (continued): Additional Informed Consent Form to Participate in Tenofovir Plasma Level Measurements (English Language)

## **Purpose**

You and your infant are participating in the study "Maternal antiviral prophylaxis to prevent perinatal transmission of HBV in Thailand". One of the potential risks associated with tenofovir during pregnancy is bone thinning in the newborn and slightly slower growth of infants. This has been studied in infants born to mothers with other viral infections but not in infants born to mothers with hepatitis B chronic infection.

The levels of tenofovir in the blood can vary from one person to another. It is possible that high tenofovir blood levels during the treatment are associated with lower bone mineral density.

To help answer these two questions, we propose that you participate in an evaluation of tenofovir plasma levels during pregnancy.

This form, along with discussions with your physician or nurse, will provide you detailed information about these additional assessments so that you can decide if you want to participate in this part of the research study. Your participation in this additional research assessment is entirely voluntary. You are free to decline participation today, or to change your decision at any future date without jeopardizing your participation in the study, your standard medical care or your possible participation in future research studies.

## Nature of the Study

We will look for a relationship between the levels of tenofovir in the blood during pregnancy and bone mineral density in mothers and infants. The average concentration of tenofovir in the blood will be estimated based on the concentrations observed at different time points after taking the study treatment.

## Study Procedures for You

You will be asked to take your study treatment every morning before the study visits at Week 32 and 36 of your pregnancy. At these two visits, you will be asked to come to the hospital in the morning before you normally take your treatment. A blood sample (2 cc or half a teaspoon) will be taken <u>before</u> you take your study treatment. After the blood draw you will take your study treatment as normal. This will be approximately at the same time you take the treatment every morning. You will then have the regular blood draw between half an hour and three hours after you have taken the study treatment, and then another 2 cc blood draw taken at least 1 hour later.

#### Duration of the subject's participation

These two additional blood draws will be performed at the 32 weeks and 36 weeks' pregnancy visits.

#### Costs to You for Participation

There is no additional cost for your participation. There will be a compensation for your time that you need to stay in the hospital for the blood draws, in addition to the reimbursement of transportation costs planned for your participation in these study visits.

## Significant New Findings

Any significant new findings that are developed during the study which could affect your willingness to continue participation will be made available to you as soon as possible.

## Withdrawal from the Study

You are free to decide not to participate in this evaluation at any time without jeopardizing your standard medical care or your possible participation in future research studies.

### Confidentiality

Your participation in this study will be kept confidential and will not be communicated to anyone without your written permission.

### Confidentiality of Records

Efforts will be made to keep your personal information confidential. Your medical records will be kept confidential. They will be disclosed to you, to those heath care providers directly involved in your care and, for study monitoring or auditing purposes, to the members of the research team, the Thai Food and Drug Administration (FDA), the Ethics committee of Institute for the Development of Human Research Protections, local Ethics Committee in your hospital, study staff, study monitors, drug companies supporting this study (drug company names) and study sponsors. All study forms will be coded by number and your name will not be recorded on these forms. Only these code numbers will be kept in the study database that will be used for analysis. Any publication of this study will not use your name or identify your personally. However, we cannot guarantee absolute confidentiality and your personal information may be disclosed if required by law.

## Policy Regarding Research Related Injuries

Immediate necessary care is available free of charge to you if you have a medical problem related to participation in this study. However, the study is not responsible for treatments unrelated to the study and no financial compensation will be provided.

## Risks to You

The risks associated with the two additional blood draws are those associated with any blood draw. The risks and discomforts of blood drawing include pain, swelling, bruising, inflammation of a vein and fainting. If necessary, you will receive appropriate care from your physician.

### Benefits to You

The objective of the study is to better assess and understand a possible relationship between tenofovir and bone mineral density but you will not directly benefit from the results of the study because the results will be known only at the end of the study.

<u>Further Questions</u> At any time, if you have further questions about this study or your rights and benefits as a participant, you may contact:

| | of Human research Protections Medical Sciences Department |
|---|---|
| | 00 Tel. 02-5913541, 02 -5913517 Fax. 02-5914125 |
| Or the your hospital's Ethics | Committee |
| | Telephone # |
| (Representative of your hosp | ital's Ethics Committee) |

For questions about the research project, your rights, and research-related injuries, you may contact a doctor independent from the research team:

Name: Dr. Sorakij Bhakeecheep

Address: National Health Security Office (NHSO)

The Government Complex Commemorating His Majesty the King's 80th Birthday Anniversary

5th December, B.E. 2550 (2007) Building B

The Ethic committee of research in Human

120 M. 3 Chaengwattana Road, Lak Si District, Bangkok 10210

Tel: +66 2141 4000 Fax: +66 2143 9730-1



| Maternal antiviral prophylaxis to prevent perinata | l transmission of HBV in Th | ailand, version 3.0 dated 20 April 20 | 15<br> |
|---|---|---|---|
| The investigator responsible for saf | eguarding your welfa | are and the welfare of your<br>ncipal investigator name at | –<br>baby,<br>t each site] |
| Address: | | | |
| Address: Telephone # Office: | Home: | Mobile: | |
| Fax: # | | | |
| or | | (name and title of Hospital | l Director) |
| Consent to participate in this study | | | |
| By signing this form, you are statin<br>the risks, and benefits of participa<br>completely free to withdraw your p<br>best medical care otherwise avai<br>penalty or loss of benefits to which | tion have been fully<br>participation at any t<br>lable. Refusing to p | explained to you. You k<br>ime without affecting your<br>participate or withdrawing | now that you are still rights to receive the |
| I agree for my participation in this s | tudy. | | |
| Woman's Name (typed or printed) | Signature | Date | |
| Woman's legal representative /Guardian (if appropriate) | Signature | Date | |
| Witness Name (typed or printed) | Signature | Date | |
| Witness Name (typed or printed) | Signature | Date | |
| I have explained the purpose of this understands the purpose, procedur | | | wledge, she |
| Investigator/Counselor Name (Typed or printed) | Signature | Date | |

# Appendix 7: Additional Informed Consent Form to Participate in DXA Scan Assessments (Thai Language)

## แบบแสดงความยินยอมเข้าร่วมโครงการวิจัยเพิ่มเติมสำหรับการตรวจประเมินความหนาแน่นของมวลกระดูกโดยการ ตรวจด้วยเครื่องดีเอ็กซ์เอ สแกน

## <u>วัตถูประสงศ์</u>

ท่านและบุตรของท่านอยู่ระหว่างการเข้าร่วมการศึกษาวิจัย "ยาต้านไวรัสสำหรับมารดาเพื่อป้องกันการถ่ายทอด เชื้อไวรัสตับอักเสบบีจากมารดาสู่ทารกในประเทศไทย" ความเสี่ยงที่สำคัญที่อาจเกิดขึ้นได้อย่างหนึ่งที่เกี่ยวกับการ รับประทานยาทีโนโฟเวียร์ในช่วงตั้งครรภ์คือทารกแรกเกิดมีภาวะกระดูกบางและการเจริญเติบโตของทารกช้าลงเล็กน้อย ได้มีการวิจัยประเด็นนี้ในทารกที่คลอดจากมารดาที่ติด เชื้อไวรัสชนิดอื่นๆ แต่ไม่มีการวิจัยในทารกที่คลอดจากมารดาที่ติด เชื้อไวรัสชนิดอื่นๆ แต่ไม่มีการวิจัยในทารกที่คลอดจากมารดาที่ติด เชื้อไวรัสตับอักเสบบีเรื้อรัง

ระดับของยาที่โนโฟเวียร์ในเลือดของแต่ละคนนั้นมีความแตกต่างกัน นอกจากนี้ยังไม่ทราบชัดเจนว่าความหนาแน่น ของมวลกระดูกที่ลดลงมีความสัมพันธ์กับระดับยาที่โนโฟเวียร์ในกระแสเลือดที่สูงในระหว่างที่รับการรักษาหรือไม่

เพื่อช่วยอธิบายเกี่ยวกับ 2 คำถามนี้ ทางโครงการขอเสนอให้ท่านและบุตรของท่านเข้าร่วมในการประเมินความ หนาแน่นของมวลกระดูกหลังคลอดบุตรแล้ว 1 ปี และเมื่อบุตรของท่านมีอายุ 1 ปี

แบบแสดงความยินยอมเข้าร่วมการวิจัยนี้ มีรายละเอียดข้อมูลเกี่ยวกับการประเมินเพิ่มเติมนี้ ซึ่งแพทย์หรือ พยาบาลผู้ดูแลท่านจะอธิบายข้อมูลให้ท่านทราบ เพื่อให้ท่านสามารถตัดสินใจได้ว่าท่านต้องการเข้าร่วมในการวิจัยนี้หรือไม่

การเข้าร่วมในการประเมินการวิจัยเพิ่มเติมนี้ของท่านจะเป็นไปโดยสมัครใจอย่างเต็มที่ ท่านมีอิสระที่จะปฏิเสธการ เข้าร่วมการวิจัยในวันนี้หรือเปลี่ยนแปลงการตัดสินใจในอนาคตได้ทุกเมื่อโดยไม่สูญเสียโอกาสในการเข้าร่วมโครงการวิจัยนี้ หรือการได้รับบริการทางการแพทย์ที่ได้มาตรฐานของท่าน หรือโอกาสในการเข้าร่วมการศึกษาวิจัยอื่นๆ ในอนาคตของท่าน

## ลักษณะของการวิจัยโดยการตรวจด้วยเครื่องดีเอ็กซ์เอ สแกน

ทางโครงการจะตรวจวัดปริมาณแคลเซียมและแร่ธาตุอื่นๆ ในมวลกระดูกของท่านและบุตรของท่าน การตรวจชนิดนี้ เรียกว่าการตรวจความหนาแน่นของมวลกระดูก โดยใช้เครื่องมือตรวจที่เรียกว่า "เครื่องตรวจโดยใช้รังสีเอ็กซ์ 2 พลังงาน" หรือเรียกว่า "ดีเอ็กซ์เอ" สแกน ซึ่งจะทำการตรวจในมารดาหลังคลอดแล้ว 1 ปีและในบุตรที่มีอายุ 1 ปี ทางโครงการจะ เปรียบเทียบการตรวจเหล่านี้ระหว่างกลุ่มการวิจัย 2 กลุ่ม (คือกลุ่มอาสาสมัครที่ได้รับยาทีโนโฟเวียร์และกลุ่มอาสาสมัครที่ ได้รับสารไร้ฤทธิ์ที่แทนยาทีโนโฟเวียร์) นอกจากนี้ทางโครงการจะศึกษาความสัมพันธ์ระหว่างระดับยาทีโนโฟเวียร์ในช่วง ตั้งครรภ์และความหนาแน่นของมวลกระดูกในมารดาและบุตรด้วย

## ขั้นตอนการวิจัยสำหรับท่าน

หลังจากที่ท่านได้คลอดบุตรแล้วก่อนครบเวลา 1 ปีหลังคลอด คณะผู้วิจัยจะติดต่อท่านเพื่อทำการนัดหมายกับท่านเพื่อ เตรียมการนำท่านและบุตรของท่านไปยังสถานที่ที่สามารถตรวจความหนาแน่นของมวลกระดูกด้วยเครื่องดีเอ็กซ์เอ สแกน ทั้งนี้ขึ้นอยู่กับว่าท่านพักอาศัยอยู่ที่ใด ซึ่งท่านต้องใช้เวลาเพื่อเดินทางไปสถานที่ตรวจนั้น โดยมีผู่ช่วยนักวิจัยหรือพยาบาล วิจัยซึ่งท่านได้รู้จักแล้วจะเดินทางไปยังสถานที่ตรวจนี้พร้อมกับท่าน ในกรณีที่ท่านทราบว่าท่านไม่สามารถไปตามนัดหมาย ได้ ท่านสามารถติดต่อคณะผู้วิจัยเพื่อนัดหมายเป็นวันอื่นได้

เครื่องดีเอ็กซ์เอใช้รังสีเอ็กซ์ในการตรวจวัดปริมาณแคลเซียมและแร่ธาตุต่างๆ ในมวลกระดูกในส่วนที่เป็นกระดูก (ได้แก่ บริเวณสะโพก กระดูกสันหลัง ข้อมือ ส้นเท้า หรือนิ้วมือ) สำหรับการประเมินนี้ ไม่มีการเจาะเลือดเพิ่มเติม ไม่มีการรักษา และไม่มีการฉีดยา โดยเป็นวิธีการตรวจที่ไม่มีอันตรายต่อร่างกาย ไม่เกิดความเจ็บปวด และใช้เวลุาไม่มาน การสัมผัสกับ

> 04857 08 โป๊ค. 2558 คณะกรรมการวริยธรรมการวิจัยโนมนุษย

รังสีมีน้อย (น้อยกว่า 5 มิลลิเร็ม) นั่นคือน้อยกว่าการถ่ายภาพรังสีธรรมดาของทรวงอก ท่านจะต้องอยู่นิ่งๆ ในระหว่างการ ตรวจ ดังนั้นอาจมีความรู้สึกไม่สบายเล็กน้อยจากการนอนในท่าเดิมเป็นเวลา 5-10 นาที

## ระยะเวลาของการเข้าร่วมโครงการวิจัยของอาสาสมัคร

ท่านและบุตรของท่านจะมีนัดหมายการวิจัยพร้อมกันเพียงครั้งเดียวเพื่อทำการตรวจวัดโดยเครื่องดีเอ็กซ์เอ สแกน

## ค่าใช้จ่ายในการเข้าร่วมโครงการวิจัยของท่าน

ท่านไม่ต้องเสียค่าใช้จ่ายเพิ่มเติมสำหรับการเข้าร่วมโครงการวิจัยนี้ จะมีค่าชดเชยสำหรับการเสียเวลาของท่านและค่าใช้จ่าย ในการเดินทางให้แก่ท่าน

## การค้นพบข้อมูลและข่าวสารใหม่ๆ ที่เกี่ยวข้อง

ทางโครงการจะแจ้งให้ท่านทราบเกี่ยวกับการค้นพบข้อมูลต่างๆ ที่เกิดขึ้นใหม่ในระหว่างการวิจัยโดยเร็วที่สุดซึ่งอาจมีผลต่อ ความสมัครใจในการเข้าร่วมโครงการวิจัยต่อไปของท่าน

## การถอนตัวออกจากการวิจัย

ท่านมีอิสระที่จะตัดสินใจไม่เข้าร่วมในการประเมินนี้เมื่อใดก็ได้โดยไม่สูญเสียโอกาสการได้รับบริการทางการแพทย์ที่ได้ มาตรฐานของท่าน หรือโอกาสในการเข้าร่วมการศึกษาวิจัยอื่นๆ ในอนาคตของท่าน

## การปกปิดความลับ

การเข้าร่วมโครงการวิจัยนี้ของท่านและบุตรของท่านจะถูกปกปิดเป็นความลับและจะไม่แจ้งให้ใครทราบโดยไม่ได้รับความ ยินยอมซึ่งเป็นลายลักษณ์อักษรจากท่าน

## การปกปิดความลับของข้อมูล

ทางโครงการจะใช้ความพยายามเพื่อเก็บข้อมูลส่วนตัวของท่านและบุตรของท่านไว้เป็นความลับ ข้อมูลทางการแพทย์ของ ท่านจะถูกเก็บรักษาไว้เป็นความลับ และจะเปิดเผยข้อมูลให้ท่านทราบตลอดจนผู้ให้การดูแลรักษาท่านโดยตรงเพื่อการ ติดตามการวิจัยหรือเพื่อวัตถุประสงค์ในการตรวจสอบการวิจัย สมาชิกของคณะผู้วิจัยสำนักงานคณะกรรมการอาหารและ ยาประเทศไทย (เอฟดีเอ) คณะกรรมการจริยธรรมการวิจัยในมนุษย์ สถาบันพัฒนาการคุ้มครองการวิจัยในมนุษย์ คณะกรรมการพิจารณาด้านจริยธรรมการวิจัยในโรงพยาบาลของท่าน เจ้าหน้าที่วิจัย ผู้ติดตามการวิจัย บริษัทยาที่สนับสนุน ยาในการวิจัยนี้ (บริษัทกิลเลียด) และผู้ให้การสนับสนุนการวิจัย แบบบันทึกข้อมูลทั้งหมดของโครงการวิจัยจะใช้หมายเลข รหัส และไม่มีการระบุชื่อของท่านในแบบบันทึกข้อมูลเหล่านี้ทางโครงการจะบันทึกเฉพาะรหัสไว้ในฐานข้อมูลการวิจัยเพื่อ ใช้ในการวิเคราะห์เท่านั้น จะไม่ใช้ชื่อของบุตรท่านหรือระบุตัวบุตรของท่านเป็นการส่วนตัวในการตีพิมพ์เอกสารใดๆ ของ การวิจัยนี้ อย่างไรก็ตามทางโครงการไม่สามารถรับรองการรักษาความลับไว้ได้อย่างสิ้นเชิง และข้อมูลส่วนตัวของท่าน อาจจะถูกเปิดเผยหากจำเป็นโดยข้อบังคับทางกฎหมาย

## นโยบายที่เกี่ยวข้องกับการได้รับอันตรายจากการวิจัย

ท่านจะได้รับการดูแลรักษาตามแนวทางปฏิบัติของประเทศและแนวทางปฏิบัติสากล



| | a | | | |
|-----|-----|-----|------|---|
| ควา | มเส | ยงข | องทำ | u |

ความเสี่ยงที่เกี่ยวข้องกับการตรวจวัดโดยเครื่องดีเอ็กซ์เอ สแกน จะเหมือนกันกับการตรวจรังสีทรวงอก รังสีที่ได้รับจาก เครื่องดีเอ็กซ์เอ สแกนจะต่ำกว่าการตรวจรังสีทรวงอก

## ผลประโยชน์ของท่าน

ท่านจะไม่ได้รับประโยชน์โดยตรงจากผลของการวิจัยเนื่องจากท่านได้รับประทานยาที่ใช้ในการวิจัยแล้วในขณะที่ทำการ ตรวจความหนาแน่นของมวลกระดูกของท่านและบุตรของท่าน

<u>ปัญหาหรือข้อซักถามเพิ่มเติม</u> เมื่อใดก็ตามหากท่านมีคำถามเพิ่มเติมเกี่ยวกับการวิจัยนี้ หรือเกี่ยวกับสิทธิและผลประโยชน์ ของท่านในฐานะอาสาสมัครท่านสามารถติดต่อ:

# คณะกรรมการจริยธรรมการวิจัยในสถาบันพัฒนาการคุ้มครองการวิจัยในมนุษย์ อาคาร 8 ชั้น 7 ห้อง 702 กรมวิทยาศาสตร์การแพทย์ กระทรวงสาธารณสุข 11000 โทรศัพท์: 02-5913541, 02-5913517 โทรสาร: 02-5914125 หรือ คณะกรรมการพิจารณาด้านจริยธรรมประจำโรงพยาบาลของท่าน \_\_\_\_\_\_\_\_ โทรศัพท์

สำหรับคำถามเกี่ยวกับโครงการวิจัย สิทธิของท่าน และอันตรายที่เกิดจากการวิจัย ท่านสามารถติดต่อแพทย์ผู้ซึ่งเป็นอิสระ จากโครงการวิจัยนี้:

ชื่อ นายแพทย์ สรกิจ ภาคีชีพ ที่อยู่ สำนักงานหลักประกันสุขภาพแห่งชาติ ศูนย์ราชการเฉลิมพระเกียรติ อาคาร บี 2550 ธันวาคม 5 พรรษา 80 10210 ถนนแจ้งวัฒนะ เขตหลักสี่ กรุงเทพฯ 3 หมู่ 120 เบอร์โทรศัพท์: +66 2141 4000 โทรสาร: +66 2143 9730-1

(ตัวแทนคณะกรรมการพิจารณาด้านจริยธรรมประจำโรงพยาบาลของท่าน)

แพทย์ผู้วิจัยที่ดูแลด้านความปลอดภัยและสิทธิของท่านและทารกของท่าน

| นพ .พญ/ | | (ชื่อผู้วิจัยหลักในสถานที่วิจัยแต่ละแห่ง) |
|---|---|---|
| ที่อยู่ | | · |
| โทรศัพท์ที่ทำงาน: | โทรศัพท์ที่บ้าน: | โทรศัพท์มือถือ: |
| โทรสาร: | | |
| หรือ | | (ชื่อและตำแหน่งผู้อำนวยการโรงพยาบาล) |
| | | 01116 |
| | | 0 8 W.A. 2558 |


คณะกรรมการจริยธรรมลารวิจัยในบนุษย

## การแสดงความยินยอมเข้าร่วมโครงการ

เมื่อท่านเซ็นชื่อในแบบแสดงความยินยอมเข้าร่วมโครงการวิจัยนี้ ท่านยอมรับว่าได้มีการอธิบายวัตถุประสงค์ของการ ศึกษาวิจัย ขั้นตอนปฏิบัติตามแผนการวิจัย ความเสี่ยง และผลประโยชน์ต่างๆ ของการเข้าร่วมโครงการวิจัยนี้ให้ท่านฟังโดย ละเอียดแล้ว ท่านทราบว่าท่านมีอิสระที่จะถอนตัวท่าน หรือบุตรของท่านออกจากการเข้าร่วมการวิจัยได้ตลอดเวลา โดยไม่ มีผลกระทบใดๆ ต่อสิทธิของท่าน หรือบุตรของท่านในการได้รับการรักษาทางการแพทย์ด้วยวิธีการอื่นๆ ที่ดีที่สุดเท่าที่มีอยู่ การปฏิเสธเข้าร่วมโครงการ หรือการถอนตัวออกจากการเข้าร่วมโครงการวิจัยจะไม่มีความผิดใดๆ และจะไม่ทำให้ท่าน สูญเสียผลประโยชน์อื่นๆ ที่ท่านควรได้รับตามสิทธิ์ที่ท่านพึงมี

| ข้าพเจ้ายินยอมเข้าร่วมโครงการวิจัย | , | | |
|---|---|---|---|
| ชื่อผู้เข้าร่วมโครงการวิจัย<br>(พิมพ์หรือเขียนตัวบรรจง) | ลายเช็น | วันที่ | |
| ชื่อตัวแทนผู้เข้าร่วมโครงการวิจัย<br>ที่ถูกต้องตามกฎหมาย / ผู้ปกครอง | ลายเซ็น<br>(ถ้ามี) | <br>วันที่ | |
| "ข้าพเจ้ายินยอมให้บุตรของข้าพเจ้า | เข้าร่วมในโครงการวิจัยนี้" | | |
| ชื่อบิดาของเด็ก<br>(ถ้ามี และมารดาเด็กยินยอม<br>พิมพ์หรือเขียนตัวบรรจง) | ลายเซ็น | <br>วันที่ | |
| ชื่อพยาน<br>(พิมพ์หรือเขียนตัวบรรจง) | ลายเซ็น | วันที่ | |
| | ลายเซ็น | <br>วันที่ | |
| | | สมัครรับทราบแล้ว ด้วยความรู้ที่ดีที่สุดขอ<br> ระโยชน์ต่างๆ ต่อตนเองและบุตรแล้ว | งข้าพเจ้า และ |
| | ลายเซ็น | วันที่ | ต<br>รีวิจัยในมนุษย |

# Appendix 7 (continued): Additional Informed Consent Form to Participate in DXA Scan Assessments (English Language)

#### Purpose

You and your infant are participating in the study "Maternal antiviral prophylaxis to prevent perinatal transmission of HBV in Thailand". One of the potential risks associated with tenofovir during pregnancy is bone thinning in the newborn and slightly slower growth of infants. This has been studied in infants born to mothers with other viral infections but not in infants born to mothers with hepatitis B chronic infection.

The levels of tenofovir in the blood can vary from one person to another. It is also unclear whether a lower bone mineral density could be related to high tenofovir levels in the blood during treatment.

To help clarify these two questions, we propose that you and your infant participate in an evaluation of bone mineral density one year after delivery, when your infant will be one year of age.

This form, along with discussions with your physician or nurse, will provide you detailed information about this additional assessment so that you can decide if you want to participate in this research.

Your participation in this additional research assessment is entirely voluntary. You are free to decline participation today or to change your decision at any future date without jeopardizing your participation in the study, your standard medical care or your possible participation in future research studies.

#### Nature of the DXA scan study

We will measure calcium and other minerals in your and your infant's bone. This measure is called bone mineral density. It is done using a machine called a "Dual-energy X-ray absorptiometry" or "DXA" scan. The measures will be performed in the mothers one year after delivery and infants at one year of age. We will compare these measures between the two study groups (i.e. those subjects receiving tenofovir and those subjects receiving tenofovir-placebo). We will also look for a relationship between the level of tenofovir during pregnancy and the bone mineral density in mothers and infants.

## Study Procedures for You

Sometime before one year after delivery, the study team will contact you to organize with you an appointment to go with you and your infant to a facility where DXA scan can be performed). Depending on where you stay, you will have to spend some time to go there. A research assistant or a study nurse that you already know will accompany you to this facility. In case you learn that you cannot be available for the appointment, you can contact the study team to find another date.

DXA uses X-rays to measure calcium and other bone minerals in a given area of bone (hip, spine, wrist, heel, or finger). For this assessment, there are no additional blood draws, no treatment and no injection. The technique is non-invasive, painless, and takes a few minutes. Radiation exposure is low (< 5 mrem), i.e. less than that of a plain radiograph of the chest. You will need to remain still during the test so there may be some minor discomfort from lying in the same position for 5 to 10 minutes.

## Duration of the subject's participation

For the DXA scan measurements, there will be only one visit for you and your infant at the same time.

## Costs to You for Participation

There are no additional costs for your participation. There will be a compensation for your time and reimbursement of your transportation costs.

## Significant New Findings

Any significant new findings that are developed during the study which could affect your willingness to continue participation will be made available to you as soon as possible.


#### Withdrawal from the Study

You are free to decide not to participate in this evaluation at any time without jeopardizing your standard medical care or your possible participation in future research studies.

## Confidentiality

You and your baby's participation in this study will be kept confidential and will not be communicated to anyone without your written permission.

## Confidentiality of Records

Efforts will be made to keep you and your child's personal information confidential. Your medical records will be kept confidential. They will be disclosed to you, to those heath care providers directly involved in your care and, for study monitoring or auditing purposes, to the members of the research team, the Thai Food and Drug Administration (FDA), the Ethics committee of Institute for the Development of Human Research Protections, local Ethics Committee in your hospital, study staff, study monitors, drug companies supporting this study (drug company names) and study sponsors. All study forms will be coded by number and your name will not be recorded on these forms. Only these code numbers will be kept in the study database that will be used for analysis. Any publication of this study will not use your child's name or identify your child personally. However, we cannot guarantee absolute confidentiality and your personal information may be disclosed if required by law.

## Policy Regarding Research Related Injuries

You will be receiving care according to national and international guidelines.

## Risks to You

The risks associated to a DXA scan measurement are similar to those of a chest X-Ray. The radiations received from a DXA scan are lower than for a chest X-Ray.

#### Benefits to You

You will not benefit directly from the results of the study because you will have already taken the study treatment when bone mineral density will be measured in you and your child.

<u>Further Questions:</u> At any time, if you have further questions about this study or your rights and benefits as a participant, you may contact:

| The Ethic committee of research in Human |
|------------------------------------------------------------------------------|
| Institute for the Development of Human research Protections |
| Building 8, Floor 7, room 702 Medical Sciences Department |
| Ministry of Public Health 11000 Tel. 02-5913541, 02 -5913517 Fax. 02-5914125 |
| Or the your hospital's Ethics Committee |
| Telephone # |
| (Representative of your hospital's Ethics Committee) |

For questions about the research project, your rights, and research-related injuries, you may contact a doctor independent from the research team:

Name: Dr. Sorakij Bhakeecheep

Address: National Health Security Office (NHSO)

The Government Complex Commemorating His Majesty the King's 80th Birthday Anniversary

5th December, B.E. 2550 (2007) Building B

120 M. 3 Chaengwattana Road, Lak Si District, Bangkok 10210

Tel: +66 2141 4000 Fax: +66 2143 9730-1



คณะกรรมการจรียธรรมดารวิจัยในหนุษฮ

| Maternal antiviral prophylaxis to prevent perinata | i transmission of tiby ii | in manand, version 5.0 dated 20 April 2015 |
|---|---|---|
| The investigator responsible for safe Dr. | | Principal investigator name at each site] |
| Address: | | |
| Telephone # Office: | Home: | Mobile: |
| Fax: # | | |
| or | | (name and title of Hospital Director) |
| Consent to participate in this study | | |
| the risks, and benefits of participal<br>completely free to withdraw your payour rights or those of your baby | tion have been for<br>articipation or you<br>to receive the b | te of this study, the procedures to be followed, and ully explained to you. You know that you are still ur baby's participation at any time without affecting est medical care otherwise available. Refusing to yor loss of benefits to which you may otherwise be |
| I agree for my participation and my | child's participation | on in this study. |
| Woman's Name (typed or printed) | Signature | Date |
| Woman's legal representative<br>/Guardian (if appropriate) | Signature | Date |
| "I agree for my child's participation | in this study." | |
| Name of the Father of the child<br>(If available and with the woman's<br>consent, typed or printed) | Signature | Date |
| Witness Name (typed or printed) | Signature | <br>Date |
| Witness Name (typed or printed) | Signature | <br>Date |
| I have explained the purpose of this the purpose, procedures, risks and | | ent. To the best of my knowledge, she understand nd her baby. |
| Investigator/Counselor Name (Typed or printed) | Signature | Date |



คณะกรรมการจริยธรรมการวิจัยในมนุษฮ